### STATISTICAL ANALYSIS PLAN

## A Phase 1b/2 Study of FT-2102 in Patients with Advanced Solid Tumors and Gliomas with an IDH1 Mutation

Protocol 2102-ONC-102 (NCT03684811)

**Protocol Number:** 2102-ONC-102

**Protocol Version and Date:** Amendment 3: 10 May 2019

Amendment 2: 01 November 2018 Amendment 1: 26 July 2018 Original: 19 June 2018

Name of Test Drug: FT-2102

Phase: Phase 1b/2

Methodology: Open-label basket study

**Sponsor:** FORMA Therapeutics

500 Arsenal St., Suite 100, Watertown MA 02472

Tel: (617) 679-1970

**Analysis Plan Date:** 28 June 2019

**Analysis Plan Version:** Version 2.0

The information contained in this document is confidential and the property of FORMA Therapeutics. Any unauthorized use or disclosure of such information without the prior written authorization of FORMA is expressly prohibited.

# **TABLE OF CONTENTS**

| Sect | ion | | | Page |
|---|---|---|---|---|
| 1. | Intro | Introduction and Objectives | | 8 |
| | 1.1. | Introduction | | 8 |
| | 1.2. | Study Objectives | | 8 |
| | 1.3. | Study Endpoints | | 10 |
| | 1.4. | Study 1 | Design | 11 |
| | | 1.4.1. | Synopsis of Study Design | 11 |
| | | 1.4.2. | Randomization Methodology | 12 |
| | | 1.4.3. | Stopping Rules and Unblinding | 12 |
| | | 1.4.4. | Study Procedures | 12 |
| | | 1.4.5. | Efficacy, Pharmacokinetic, Pharmacodynamic and Safety Parameters | 12 |
| 2. | Patier | Patient Population | | 15 |
| | 2.1. | Analys | sis Sets | 15 |
| | 2.2. | Protoc | ol Violations | 16 |
| 3. | Gener | General Statistical Methods | | |
| | 3.1. | Sample Size Justification | | 17 |
| | 3.2. | General Methods | | 18 |
| | 3.3. | Computing Environment | | 19 |
| | 3.4. | Baseline Definitions | | 20 |
| | 3.5. | Methods of Pooling Data | | 20 |
| | 3.6. | Adjustments for Covariates | | 20 |
| | 3.7. | Multiple Comparisons/Multiplicity | | 20 |
| | 3.8. | Subpopulations | | 20 |
| | 3.9. | Withdrawals, Dropouts, Loss to Follow-up | | 22 |
| | 3.10. | Missing, Unused, and Spurious Data | | 22 |
| | 3.11. | Visit Windows | | 23 |
| | 3.12. | Interim Analyses | | 23 |
| 4 | Study | Analyse | es. | 25 |

| Secti | on | | | Page |
|---|---|---|---|---|
| | 4.1. | Patient | t Disposition | 25 |
| | 4.2. | Demog | graphics and Baseline Disease Characteristics | 25 |
| | 4.3. | Efficac | ey Evaluations | 28 |
| | | 4.3.1. | Disease Response and Survival Analyses | 28 |
| | | 4.3.2. | Quality of Life Assessment Analysis | 32 |
| | 4.4. | Pharm | acokinetic and Pharmacodynamic Evaluations | 33 |
| | 4.5. | Safety | Analyses | 38 |
| | | 4.5.1. | Study Drug Exposure | 38 |
| | | 4.5.2. | Adverse Events | 39 |
| | | 4.5.3. | Laboratory Data | 42 |
| | | 4.5.4. | Vital Signs and Physical Examination | 46 |
| | | 4.5.5. | Electrocardiogram | 46 |
| | | 4.5.6. | Concomitant Medications and Procedures | 47 |
| | | 4.5.7. | Performance Status | 48 |
| 5. | Expl | oratory A | Analyses | 49 |
| 6. | Char | iges to Pl | anned Analyses | 50 |
| 7. | Refe | rences | | 51 |
| 8. | Clinical Study Report Appendices | | 52 | |
| | 8.1. | Statistical Tables and Figures to be Generated | | 53 |
| | 8.2. | Data L | istings to be Generated | 65 |
| 9. | Tabl | e and Fig | gure Shells | 67 |
| 10. | Data | Listing S | Shells | 152 |
| 11. | Revis | sion Histo | ory | 199 |
| 12. | Stud | y Schema | ntic | 201 |

# TABLES INCLUDED IN THE TEXT

| | | Page |
|---------|-----------------------------------------|------|
| Table 1 | Pharmacokinetic Parameters for Analysis | 34 |

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation | Definition |
|---|---|
| 2-HG | (R)-2-hydroxyglutarate |
| AE | Adverse event |
| AFP | Alpha-fetoprotein |
| α-KG | $\alpha$ -ketoglutarate |
| ALP | Alkaline phosphatase |
| ALT (SGPT) | Alanine aminotransferase (serum glutamic pyruvic transaminase) |
| ANC | Absolute neutrophil count |
| AST (SGOT) | Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) |
| ATC | Anatomic therapeutic class |
| AUC | Area under the concentration versus time curve |
| $\mathrm{AUC}_{0\text{-}24}$ | Area under the concentration versus time curve from time 0 to the end of the dosing interval 24 hours later, calculated using linear trapezoid rule |
| β-HCG | Beta human chorionic gonadotropin |
| BOR | Best overall response |
| BQL | Below quantifiable limit |
| $C_{\text{max}}$ | Maximum plasma concentration |
| $C_{\min}$ | Trough plasma concentration, taken 24 hours after dose and prior to subsequent dose |
| CBC | Complete blood count |
| CEA | Carcinoembryonic antigen |
| CI | Confidence interval |
| cm | Centimeter |
| CNS | Central nervous system |
| CR | Complete response |
| CRF | Case report form |
| CSF | Cerebrospinal fluid |
| CSR | Clinical study report |
| CT | Computed tomography |
| ctDNA | Circulating tumor DNA |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CV | Coefficient of variation |
| DLT | Dose-limiting toxicity |
| DNA | Deoxyribonucleic acid |
| DOR | Duration of response |

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| ECOG | Eastern Cooperative Oncology Group |
| ECG | Electrocardiogram |
| FDA | Food and Drug Administration |
| g | Gram |
| HBC | hepatobiliary cancer |
| ICH | International Conference on Harmonisation |
| IDH1 | Isocitrate dehydrogenase 1 |
| IDH2 | Isocitrate dehydrogenase 2 |
| IHCC | intrahepatic cholangiocarcinoma |
| IRB | Institutional Review Board |
| IWG | International Working Group |
| IV | Intravenous |
| kg | Kilogram |
| KM | Kaplan Meier |
| L | Liter |
| LDH | Lactic dehydrogenase |
| $m^2$ | Square meter |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mEq | Milliequivalence |
| mg | Milligram |
| mL | Milliliter |
| mm | Millimeter |
| $mm^3$ | Cubic millimeter |
| MR | Minor response |
| MRI | Magnetic resonance imaging |
| MRS | Magnetic resonance spectroscopy |
| MTD | Maximum tolerated dose |
| N | Number |
| NOS | Not otherwise specified |
| ORR | Overall response rate |
| OS | Overall survival |
| PD | Progressive disease |
| % | Percent |
| PFS | Progression-free survival |
| рН | Hydrogen ion concentration |

| Abbreviation | Definition |
|------------------|---------------------------------------------|
| PK | Pharmacokinetic |
| PR | Partial response |
| PT | Preferred term |
| PTT | Partial thromboplastin time |
| QD | quaque die/ once daily |
| QOL | Quality of life |
| QT | Interval between Q and T waves |
| QTc | Corrected interval between Q and T waves |
| RBC | Red blood cell (count) |
| Rel Day | Relative study day |
| RP2D | Recommended phase 2 dose |
| RTF | Rich text format |
| SAE | Serious adverse events |
| SAP | Statistical analysis plan |
| SC | Subcutaneous |
| SD | Stable disease <i>or</i> Standard deviation |
| SI | International System of Units |
| SOC | System organ class |
| $T_{1/2}$ | Half-life |
| $T_{\text{max}}$ | Time to maximum plasma concentration |
| TT | Treatment termination |
| TTP | Time to progression |
| TTR | Time to response |
| ULN | Upper limit of normal |
| $V_{ m dss}$ | Volume of distribution at steady state |
| WBC | White blood cell (count) |
| WHO | World Health Organization |

### 1. INTRODUCTION AND OBJECTIVES

#### 1.1. Introduction

Isocitrate dehydrogenase 1 (IDH1) and isocitrate dehydrogenase 2 (IDH2) mutations in cancer result in abnormal hypermethylation of histones and DNA and suppression of normal cellular differentiation. The metabolic enzyme IDH1 catalyzes the oxidative decarboxylation of isocitrate to  $\alpha$ -ketoglutarate ( $\alpha$ -KG). In both hematologic and solid tumor malignancies, IDH1 mutations lead to aberrant accumulation of (R)-2-hydroxyglutarate (2-HG). 2-HG has been proposed to act as an "oncometabolite" that has pleotropic effects on tumorigenesis. Excess production of 2-HG has been shown to inhibit  $\alpha$ -KG-dependent enzymes involved in epigenetic regulation, collagen synthesis, and cell signaling, thereby leading to a block in normal differentiation of progenitor cells and the subsequent development of cancer (Gross et al, 2010; Cairns et al, 2019; Losman et al, 2013). Therefore, inhibition of mutated IDH1 in tumor cells and the concomitant decrease in 2-HG production is expected to restore normal cellular differentiation and provide therapeutic benefit in IDH1-mutated cancers.

The identification of frequent mutations in the IDH1 and IDH2 genes in human cancers including glioma, hepatocellular carcinomas, chondrosarcomas and intrahepatic cholangiocarcinoma (IHCC) has provided novel therapeutic targets in these diseases (Yan et al, 2009; Amary et al, 2011; Wang et al, 2013; Lee et al, 2017). IDH mutation specific inhibitors have been shown to reduce aberrantly elevated levels of the oncometabolite 2-HG, resulting in antitumor efficacy in preclinical models (Rohle et al, 2013; Saha et al, 2014). Clinical investigation in patients with IHCC, gliomas and chondrosarcomas are ongoing with several other IDH1 inhibitors. A comparable IDH1 inhibitor, ivosidenib has published preliminary data regarding clinical activity in gliomas, chondrosarcomas and IHCC (Tap et al, 2016; Ishii et al, 2017; Mellinghoff et al, 2017).

# 1.2. Study Objectives

This statistical analysis plan (SAP) is designed to outline the methods to be used in the analysis of study data in order to answer the study objectives. Populations for analysis, data handling rules, statistical methods, and formats for data presentation are provided. The statistical analyses and summary tabulations described in this SAP will provide the basis for the results sections of the clinical study report (CSR) for this trial.

This SAP will also outline any differences in the currently planned analytical objectives relative to those planned in the study protocol.

## **Primary Objectives**

Phase 1b: Evaluate the safety and tolerability of FT-2102 as monotherapy and confirm the dose to be further examined in expansion cohorts as monotherapy and combination therapy.

Phase 2: Evaluate the clinical activity of FT-2102 as monotherapy or in combination in patients with glioma, HBC, chondrosarcoma, and IHCC harboring an IDH1 mutation.

#### **Secondary Objectives**

#### Phase 1b:

- Evaluate the PK of FT-2102 as monotherapy and in combination with other anticancer agents
- Evaluate the clinical activity of FT-2102 as a single agent or in combination in patients with glioma, HBC, chondrosarcoma, and IHCC harboring an IDH1 mutation

#### Phase 2:

- Evaluate the safety of FT-2102 administered as monotherapy and in combination with other anti-cancer agents in patients with glioma, HBC, chondrosarcoma, and IHCC harboring an IDH1 mutation
- Evaluate the PK of FT-2102 as monotherapy and in combination with other anticancer agents
- Evaluate additional measures of antitumor activity of FT-2102 as monotherapy or in combination with other anti-cancer agents

#### **Exploratory Objectives**

- Evaluate potential biomarkers of response, resistance, and/or safety
- Evaluate pharmacodynamic and PK/pharmacodynamic relationship of FT-2102 as monotherapy and in combination with other anti-cancer agents
- Evaluate the biological effects of FT-2102 on tumor tissue, including tumor cells, CSF, immune cells, and vasculature
- Evaluate the biological effects of FT-2102 on tumor tissue, including tumor cells, CSF, immune cells, and vasculature
- Assess IDH1 mutations in ctDNA and correlate with mutations in tumor tissues

• Evaluate the health-related quality of life (QOL)

## 1.3. Study Endpoints

### **Primary Endpoint**

Phase 1b: DLTs (Safety Lead-in Periods), adverse event (AEs), and safety laboratory values

Phase 2: Objective response rate (ORR), as determined by applicable disease criteria, for disease-specific cohorts

## **Secondary Endpoints**

- AEs, and safety laboratory values (Phase 2)
- ORR (Phase 1b only)
- PFS, defined as the time from the first dose to disease progression as determined by applicable disease criteria or death due to any cause, whichever is sooner
- Time to progression (TTP), defined as the time from start of treatment until disease specified progression
- Duration of response (DOR), defined as the time from the first response to documented disease progression as determined by applicable disease criteria
- OS, defined as the time from the first dose to death due to any cause
- Time to Response (TTR), defined as the time from first dose to first response
- AEs and abnormal laboratory findings
- PK parameters derived from plasma/cerebrospinal fluid (CSF) FT-2102 concentrations

### **Exploratory Endpoints**

• Pharacodynamic and PK/pharmacodynamic in relationship with clinical safety and clinical activity

- Changes in 2-hyroxygluterate (2-HG levels) (pharmacodynamic, biomarker) in plasma and tumor tissue (1H magnetic resonance spectroscopy (MRS) and CSF in intracranial gliomas and tumor biopsies for other tumors)
- Characterization of biological effects of FT-2102 on tumor biopsies
- Cancer-associated mutations and/or genetic alterations
- IDH1 mutation in ctDNA
- Health-related QOL patient-reported questionnaire (EQ5D)

## 1.4. Study Design

### 1.4.1. Synopsis of Study Design

This is a multicenter, Phase 1b/2, open-label, multiple-cohort study examining the efficacy and safety of FT-2102 as a single agent or in combination for the treatment of patients with advanced solid tumors and gliomas with IDH1 R132X mutations.

The study is comprised of 5 cohorts, where four cohorts represent different types of solid tumors and one represents gliomas. Within three of the solid tumor and the glioma cohorts, initially FT-2102 will be administered in a single agent regimen. Each cohort is designed as an independent Simon 2-stage study. If, within a cohort, the Simon 2-stage stops either at the interim analysis for futility or if the final analysis fails to accept the alternative hypothesis, dosing with FT-2102 in combination with other therapies (specific to the disease under study) may commence in a new Simon 2-Stage assessment. Cohort 5 is comprised of "other non-central nervous system (CNS) solid tumors" for patients harboring an IDH-R132X mutation (i.e. other solid tumors that do not fit into the first 4 cohorts). This cohort is purely exploratory, and thus is not designed as a Simon 2-stage. There are no plans to administer any combination therapy for patients enrolled into cohort 5; it is designed as a single agent therapy cohort only.

The Phase 1b part of the study is a safety-lead in, 3+3 study design in which the dose of 150 mg BID, which has been selected as the Phase 2 dose in a concurrent study in AML (2102-HEM-101) will be evaluated for safety. Once the Phase 1b portion is complete and the recommended Phase 2 dose (RP2D) has been selected for a cohort, the Phase 2 portion of the study may commence. The RP2D may differ for each cohort. Patients in the Phase 1b portion who were dosed at the RP2D dose level may contribute to the Phase 2 Simon 2-Stage evaluation.

An overview of the study is depicted in Section 12 of the SAP.

## 1.4.2. Randomization Methodology

N/A; study is open-label.

#### 1.4.3. Stopping Rules and Unblinding

Unblinding is not applicable as study is open label. Several stopping rules apply, as there are Simon 2-Stage study designs within each cohort.

#### 1.4.4. Study Procedures

The schedule of assessments is outlined in the study protocol, Tables 2-8. Refer to the study protocol for these details.

- 1.4.5. Efficacy, Pharmacokinetic, Pharmacodynamic and Safety Parameters
- 1.4.5.1. Efficacy Parameters

Objective Response Rate is defined as follows:

- Glioma: the proportion of patients with a best response of CR, PR or MR (LGG)
- HBC: the proportion of patients with a best response of CR or PR
- Chondrosarcoma: the proportion of patients with a best response of CR or PR
- Cholangiocarcinoma: the proportion of patients with a best response of CR or PR

Best overall response (BOR): BOR is the best response achieved by the patient at any time while on study.

Progression Free Survival (PFS): defined as the time from the date of the first dose to the date of disease progression as determined by applicable disease criteria or death due to any cause, whichever is sooner. If a patient withdraws from the study prior to an event occurring, the patient will be censored at the date of the last response evaluation.

Time to Progression (TTP): defined as the time from the date of the first dose to the date of disease progression as determined by applicable disease criteria. If progression does not occur while on study, the patient will be censored at the date of the last response evaluation.

Duration of Response (DOR): defined as the time from the date of the first response to the date of the documented disease progression as determined by applicable disease criteria. If progression does not occur while on study, the patient will be censored at the date of the last response evaluation. This will only be calculated for those patients who have a best response of MR or better.

Overall Survival (OS): defined as the time from the date of the first dose to the date of death due to any cause. If death is not recorded, the patient will be censored at the date of the last known alive.

Time to Response (TTR): defined as the time from the date of first dose to the date of first CR, PR or MR response. This will only be calculated for those patients who have a best response of MR or better.

Best percent change in tumor burden while on study: Maximum percentage reduction or minimum percentage increase at a single time point of the patient's tumor burden post first dose of study drug.

Time on treatment: Time from the date of first FT-2102 dose to the date of the last FT-2102 dose.

Health-related QOL patient-reported questionnaire (EQ5D): Change from baseline for each dimension and overall, number of patients reporting each score for each dimension and overall, and number of patients reporting some problems on each dimension.

#### 1.4.5.2. Pharmacokinetic Parameters

Blood samples for determination of FT-2102 pharmacokinetics are to be collected as outlined in the protocol. Pharmacokinetic parameters to be derived from FT-2102 plasma concentrations collected in Phase 1b (Stage 1) include minimum plasma concentration ( $C_{min}$ ), maximum plasma concentration ( $C_{max}$ ), time to maximum plasma concentration ( $T_{max}$ ), and area under the concentration versus time curve (AUC).

#### 1.4.5.3. Pharmacodynamic Parameters

Pharacodynamic assessments being performed in this study include:

- Changes in 2-hyroxygluterate (2-HG) levels (PD, biomarker) in plasma, urine and tumor tissue (1H magnetic resonance spectroscopy (MRS)) and CSF (if available) in intracranial gliomas and tumor biopsies for other tumors)
- Characterization of biological effects of FT-2102 on tumor biopsies
- Cancer-associated mutations and/or genetic alterations
- IDH1 mutation in ctDNA

### 1.4.5.4. Safety Parameters

DLTs will be assessed for each dose evaluated in the Phase 1b phase.

The maximum tolerated dose (MTD) will be evaluated.

The RP2D will be determined for each cohort based on both safety and efficacy.

Safety evaluations performed during the study included physical examinations, measurement of vital signs, 12-lead electrocardiograms, clinical laboratory evaluations including hematology, serum chemistry, and urinalysis, and monitoring of adverse events and concomitant medications.

### 2. PATIENT POPULATION

## 2.1. Analysis Sets

## **Dose-Limiting Toxicity-Evaluable Analysis Set**

The DLT-Evaluable Analysis Set is defined as all patients in the Safety Lead-in Periods (single- agent FT-2102, combination FT-2102 + 5-azacitidine, combination FT-2102 + GemCis and combination FT-2102 + PD-1 inhibitor) who either experienced a DLT during Cycle 1 or completed at least 75% of the prescribed Cycle 1 dose. This analysis set will be used to assess the tolerability of FT-2102.

#### Safety Analysis Set

The Safety Analysis Set is defined as all patients who received any amount of study drug(s) (FT-2102 and combination agents, if appropriate).

This analysis set will be the primary analysis set for all safety endpoints, excluding DLT evaluation. Safety analysis will be by cohort and by treatment within cohort if more than 1 dose or dosing combination are initiated for a particular indication cohort.

### Response-Evaluable Analysis Set

The Response-Evaluable Analysis Set is defined as all patients with measurable disease at baseline are included in the Safety Analysis Set and had at least 1 post-baseline response assessment or discontinued the treatment phase due to disease progression (including death caused by disease progression) within 8 weeks (+2-week window) of the first dose of study treatment. This analysis set will be the primary analysis set for efficacy endpoints. All response evaluations will be by cohort, and by treatment within cohort if more than 1 doses or dosing combinations are initiated for a particular indication cohort.

### **Pharmacokinetics Analysis Set**

The PK analysis set is defined as patients from Stage 1 who have received at least one dose of FT-2102 and for whom it is possible to calculate at least one primary PK parameter (e.g.  $C_{max}$ ,  $AUC_{last}$ ).

#### **Pharmacodynamics Analysis Set**

The Pharmacodynamic analysis set is defined as all patients who received at least one dose of FT-2102 and have completed at least one pharmacodynamic assessment.

## 2.2. Protocol Violations

Major protocol violations, as determined by a de-identified review of the data, may result in the removal of a patient's data from the Response Evaluable population. The Sponsor will be responsible for producing the final protocol violation file (formatted as a Microsoft Excel file), this file will include a description of the protocol violation and clearly identify whether this violation warrants exclusion from the Response Evaluable population. This file will be finalized prior to database lock.

All protocol violations will be presented in a data listing.

### 3. GENERAL STATISTICAL METHODS

## 3.1. Sample Size Justification

This study will enroll up to approximately 200 patients.

A single-agent Safety Lead-in Period will be implemented that may enroll approximately 12 patients, which includes approximately 6 patients with glioma and 6 patients with solid tumors. Following successful completion of the Safety Lead-in Period, the study will then enroll 4 disease-specific cohorts examining FT-2102 as either a single agent or in combination. These cohorts include Cohort 1 (glioma) with 16-46 patients; Cohort 2 (HBC) with 21-78 patients; Cohort 3 (chondrosarcoma) with 16-46 patients; and Cohort 4 (IHCC) with 21-78 patients. There will be a fifth cohort of R132X IDH1 mutant solid tumors, non-CNS with up to 6 patients, single-agent only.

### Cohort 1a, Cohort 2a, Cohort 3a (single-agent FT-2102)

Cohorts, 1a, 2a and 3a will employ an optimal Simon's 2-Stage design with a 1-sided alpha of 0.025, power of 80%, null hypothesis of 5% and alternative hypothesis of 25%. Stage 1 of these cohorts will evaluate 8 patients for efficacy over 4 treatment cycles; if there are 1 or more responses, Stage 2 will initiate with additional 15 patients. If there are 4 or more responses out of the total 23 patients, the null hypothesis of 5% will be rejected. If there is no response in Stage 1 with single-agent FT-2102, or if the null hypothesis is not rejected at the end of Stage 2, combination therapy may be evaluated.

#### Cohort 4a (single-agent FT-2102)

Cohort 4a employs an optimal Simon's 2-Stage design with a 1-sided alpha of 0.025, power of 80%, null hypothesis of 8% and alternative hypothesis of 35%. Stage 1 will evaluate 8 patients and if there are 2 or more responses Stage 2 will initiate with additional 14 patients. If there are 5 or more responses out of the total 22 patients, the null hypothesis of 8% will be rejected. If there is 0 or 1 response in Stage 1 with single-agent FT-2102, or if the null hypothesis is not rejected at the end of Stage 2, combination may be evaluated.

#### Combination Cohorts (1b, 2b, 3b, 4b)

If there is no response in Stage 1 with single-agent FT-2102, combination cohorts may be examined.

#### Cohort 1b and Cohort 3b

For Cohorts 1b and 3b (combination therapy), an optimal Simon's 2-Stage design will be implemented with a 1-sided alpha of 0.025, 80% power, with a null hypothesis of 5% and alternative hypothesis of 25%. Stage 1 of each cohort will evaluate 8 patients for efficacy over 4 treatment cycles; if there are 1 or more responses, Stage 2 will initiate with

additional 15 patients. If there are 4 or more responses out of the total 23 patients, the null hypothesis of 5% will be rejected.

### Cohort 2b

Cohort 2b employs an optimal Simon's 2-Stage design with a 1-sided alpha of 0.025, power of 80%, null hypothesis of 20% and alternative hypothesis of 40%. Stage 1 will evaluate 13 patients for efficacy; if there are 4 or more responses Stage 2 will initiate with an additional 42 patients. If there are 17 or more responses out of the total 55 patients, the null hypothesis of 20% will be rejected.

#### Cohort 4b

Cohort 4b employs an optimal Simon's 2-Stage design with a 1-sided alpha of 0.025, power of 80%, null hypothesis of 20% and alternative hypothesis of 40%. Stage 1 will evaluate 13 patients and if there are 4 or more responses Stage 2 will initiate with additional 42 patients. If there are 17 or more responses out of the total 55 patients, the null hypothesis of 20% will be rejected.

#### Cohort 5

Cohort 5, due to the diverse population, this is an exploratory cohort without pre-defined efficacy/futility determinations (n=6).

#### 3.2. General Methods

Data will be summarized in the following groupings:

| Group Description | Table Column Header |
|-------------------------------------------------|---------------------|
| Cohort 1A: Glioma FT-2102 | C1A Glioma SA |
| Cohort 1B: Glioma FT-2102 + Azacitidine | C1B Glioma Combo |
| Cohort 1: Glioma | C1 Glioma Overall |
| Cohort 2A: HBC FT-2102 | C2A HBC SA |
| Cohort 2B: HBC FT-2102 + Nivolumab | C2B HBC Combo |
| Cohort 2: HBC | C2 HBC Overall |
| Cohort 3A: Chondrosarcoma FT-2102 | C3A Chondro SA |
| Cohort 3B: Chondrosarcoma FT-2102 + Azacitidine | C3B Chondro Combo |

| Cohort 3: Chondrosarcoma | C3 Chondro Overall |
|---|---|
| Cohort 4A: Cholangiocarcinoma FT-2102 | C4A Cholangio SA |
| Cohort 4B: Cholangiocarcinoma FT-2102<br>+ Gemcitibine + Cisplatin | C4B Cholangio Combo |
| Cohort 4: Cholangiocarcinoma | C4 Cholangio Overall |
| Cohort 5: Other Solid Tumors FT-2102 | C5 Other Tumors SA |

All data listings that contain an evaluation date will contain a relative study day (Rel Day). Pre-treatment and on-treatment study days are numbered relative to the day of the first dose of study medication which is designated as Day 1. The preceding day is Day -1, the day before that is Day -2, etc.

All output will be incorporated into Microsoft Word files, sorted and labeled according to the International Conference on Harmonisation (ICH) recommendations, and formatted to the appropriate page size(s).

Tabulations will be produced for appropriate demographic, baseline, efficacy, pharmacokinetic, and safety parameters. For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) of the parameter will be presented. For continuous variables, the number of patients, mean, median, standard deviation (SD), minimum, and maximum values will be presented. Time-to-event data will be summarized using Kaplan-Meier methodology using 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles with associated 2-sided 95% confidence intervals, as well as percentage of censored observations. Minimum and maximum values will be presented to the same decimal precision as the raw values, mean and median values to one more, and the standard deviation to two more decimal places that the raw values. And for categorical: all percentages will be presented to one decimal place.

Formal statistical hypothesis testing will be performed on overall response rate with all tests conducted at the 1-sided, 0.025 level of significance. Summary statistics will be presented, as well as confidence intervals on selected parameters, as described in the sections below.

Aside from the primary endpoint of overall response rate, other data analyses are descriptive and will be summarized using descriptive statistics noted above.

#### Relevant Output

Listing 16.2.0.1 Treatment Codes Applicable to Tables and Listings

# 3.3. Computing Environment

All descriptive statistical analyses will be performed using SAS statistical software Version 9.3 or higher, unless otherwise noted. Medical history and adverse events will

be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 21.0. Concomitant medications and prior therapies will be coded using the World Health Organization (WHO) Drug Dictionary Version Global B3 format March 2018.

#### 3.4. Baseline Definitions

For all analyses, baseline will be defined as the most recent measurement prior to the first administration of study drug.

## 3.5. Methods of Pooling Data

Data will be pooled for the Phase 1b and Phase 2 patients who are in the EE Population who are dosed at the same level for purposes of the test of the primary endpoint and other efficacy analyses.

Data for each cohort will be pooled for patients within treatment regimen. Data from all study sites and countries will be pooled together.

# 3.6. Adjustments for Covariates

No formal statistical analyses that adjust for possible covariate effects are planned. Ad hoc analyses examining covariate effects may be performed.

# 3.7. Multiple Comparisons/Multiplicity

No adjustments to the overall alpha of this study have been made. Each cohort is independent and will be tested with a single primary endpoint at the 1-sided 0.025 level, so the control of false positives is maintained within each cohort.

# 3.8. Subpopulations

Selected analyses will be performed by subgroup. Some subgroups only apply to selected cohorts. The following subgroups will be examined:

- Gender
- Caucasian vs. other races
- Asian vs. other races (Cohorts 2 and 4 only)
- Baseline ECOG 0/1 vs 2
- Baseline Child-Pugh Score (Cohorts 2 and 4 only)
- Age  $(18-40, 41-59, \ge 60)$
- Prior surgery only vs. prior surgery and other anti-cancer therapies

- Number of prior regimens (1, 2, 3, >3)
- Prior IDH1 therapy (yes, no) (combination therapy patients only- Cohort 1b, 2b, 3b, 4b)
- Prior temozolomide (yes, no) (Cohort 1 only)
- Prior procarbazine/CCNU/vincristine (yes, no) (Cohort 1 only)
- Prior radiation therapy (yes, no) (Cohort 1 only)
- Baseline steroids (yes, no) (Cohort 1 only)
- Baseline tumor grade (I or II, III, IV)
- Baseline tumor grade (Stage I, II, or III vs. Stage IV)
- Hepatitis B positive (yes, no) (Cohort 2 only)
- Hepatitis C positive (yes, no) (Cohort 2 only)
- Hepatitis B or C positive (yes, no) (Cohort 2 only)
- Prior gemcitabine-based therapy (yes, no) (Cohorts 2 and 4 only)
- Prior nivolumab or pembrolizumab therapy (yes, no) (Cohort 2)
- Cancer diagnosis (hepatocellular carcinoma, gallbladder carcinoma, IHCC, extrahepatic cholangiocarcinoma, biliary tumor NOS) (Cohort 2 only)
- Glioma diagnosis (Cohort 1 only). Diagnosis subgroupings to be determined based on the data from enrolled patients.
- Chondrosarcoma diagnosis (differentiated, mesenchymal, clear cell, unknown/ other) (Cohort 3 only)
- IDH1 mutation subtype (R132H, R132C, other R132 subtypes)
- Co-mutations. Subgroupings to be determined based on the data from enrolled patients.
- Responder status (best overall response of MR or better vs. non-responder)
- Tumor imaging method (enhancing, non-enhancing). Enhancing = yes if: Screening imaging assessment was performed via T1 MRI post contrast. Otherwise enhancing = no.

## 3.9. Withdrawals, Dropouts, Loss to Follow-up

Patients who drop out from Phase 1b who are not able to be included in the DLT evaluable population will be replaced to fill the required numbers of patients to evaluate each dose level per the study protocol.

As the sample size for Phase 2 is based on the Response Evaluable Population, if patients drop out before they become evaluable for Response they will be replaced.

## 3.10. Missing, Unused, and Spurious Data

In general, there will be no substitutions made to accommodate missing data points. All data recorded on the case report form will be included in data listings that will accompany the clinical study report.

Handling of values listed as BLQ for PK and PD data is described in Section 4.4.

Missing partial date of adverse events or concomitant medications will be imputed for purposes of classification as treatment emergent or concomitant, but in data listings the reported date, not the imputed date, will be presented. In cases where a date part is missing, a relday will not be calculated and presented in the listing; the relday will be missing.

#### Adverse events

When tabulating adverse event data, partial dates will be handled as follows. If the day of the month is missing, the onset day will be set to the first day of the month unless it is the same month and year as study treatment. In this case, in order to conservatively report the event as treatment-emergent, the onset date will be assumed to be the date of treatment. If the onset day and month are both missing, the day and month will be assumed to be January 1, unless the event occurred in the same year as the study treatment. In this case, the event onset will be coded to the day of treatment in order to conservatively report the event as treatment-emergent. A missing onset date will be coded as the day of treatment.

#### Concomitant medications

For records with a missing medication start and/or stop date, the following procedure will be employed for use in determining whether the medication is prior or concomitant:

- Medication start dates with a missing day and non-missing month will be assumed to occur on the first day of the non-missing month, except for medications occurring in the first month of dosing, in which case the date will be the first day of dosing.
- Medication start dates with missing month will be assumed to occur on the first day of the non-missing year (i.e., January 1), except for medications

occurring in the first year of dosing, in which case the date will be the first day of dosing.

- Medication start year is unknown, the date will not be imputed.
- Medications that are not ongoing and have a medication stop date with a
  missing day and non-missing month will be assumed to occur on the last day
  of the non-missing month.
- Medications that are not ongoing and have a medication stop date with a missing month will be assumed to occur on the last day of the non-missing year (ie, December 31).
- Medications that are not ongoing and have a medication stop date with a missing year will be assumed to occur on the first day of dosing.

#### 3.11. Visit Windows

It is expected that all visits should occur according to the protocol schedule. All data will be tabulated per the evaluation visit as recorded on the CRF even if the assessment is outside of the visit window. In data listings, the relative day of all dates will be presented.

## 3.12. Interim Analyses

Within each cohort, Optimal Simon's 2-Stage designs are employed for both the single agent treatment and also for combination treatment. There are different hypotheses being tested for each cohort, and thus there are different stopping rules for the cohorts, which are described below. All of the following interim analyses are to be conducted on the Response Evaluable Set.

Combination therapy in cohorts 1-4 may also be examined in the event that the single agent cohort passes the futility analysis and the enrollment in the single agent cohort is completed following review by the SRC (below).

#### Cohort 1a, Cohort 2a, Cohort 3a (single-agent FT-2102)

Cohorts 1a, 2a, and 3a will employ an optimal Simon's 2-Stage design testing a null hypothesis of 5% response versus alternative hypothesis of 25% response. Stage 1 will evaluate 8 patients for efficacy over 4 treatment cycles; if there are 1 or more responses, Stage 2 will initiate with additional 15 patients. If there is no response in Stage 1 with single-agent FT-2102, combination therapy will be evaluated (Cohorts 1b, 2b, 3b).

#### Cohort 4a (single-agent FT-2102)

Cohort 4a employs an optimal Simon's 2-Stage design testing a null hypothesis of 8% response versus the alternative hypothesis of 35% response. Stage 1 will evaluate 8 patients and if there are 2 or more responses Stage 2 will initiate with additional 14 patients. If there is 0 or 1 response in Stage 1 with single-agent FT-2102, combination therapy will be evaluated (Cohort 4b).

#### Cohort 1b and Cohort 3b

For Cohorts 1b and 3b (combination therapy), an optimal Simon's 2-Stage design will be implemented to test a null hypothesis of 5% response versus the alternative hypothesis of 25% response. Stage 1 of each cohort will evaluate 8 patients for efficacy over 4 treatment cycles; if there are 1 or more responses, Stage 2 will initiate with additional 15 patients. If there is no response in Stage 1, enrollment will cease, and the null hypothesis will fail to be rejected.

#### Cohorts 2b and 4b

Cohorts 2b and 4b employ an optimal Simon's 2-Stage design to test a null hypothesis of 20% response versus alternative hypothesis of 40% response. Stage 1 will evaluate 13 patients for efficacy; if there are 4 or more responses Stage 2 will initiate with an additional 42 patients. If there are 3 or fewer responses, enrollment will cease, and the null hypothesis will fail to be rejected.

### 4. STUDY ANALYSES

## 4.1. Patient Disposition

Patient disposition will be tabulated and include the number screened, the number treated in total, the number dosed with FT-2102, the number dosed with azacitidine, nivolumab, or gemcitabine/cisplatin, the number in each patient population for analysis, the number of patients who are ongoing in treatment FT-2102 or, if they have ceased treatment with FT-2102, the reason for stopping. The number of patients who are ongoing in the study (whether on treatment or off treatment still in follow up), or if they have ceased study participation the reason for stopping participation in the study. Separate tables will be run for each cohort and within each cohort, tables will be tabulated by single agent therapy and combination therapy.

A by-patient data listing of study disposition information will be presented by cohort and dose level.

#### Relevant Output

| Table 14.1.1 Table 14.1.1 Table 14.1.1 Table 14.1.1 Table 14.1.1 | Patient Enrollment and Disposition (Cohort 1) Patient Enrollment and Disposition (Cohort 2) Patient Enrollment and Disposition (Cohort 3) Patient Enrollment and Disposition (Cohort 4) Patient Enrollment and Disposition (Cohort 5) |
|---|---|
| Listing 16.2.1.1<br>Listing 16.2.1.2<br>Listing 16.2.1.3<br>Listing 16.2.2.1<br>Listing 16.2.2.2<br>Listing 16.2.3.1 | Study Completion Status Pre-Screening Consent Enrollment Inclusion and Exclusion Criteria Protocol Violations Analysis Sets |

# 4.2. Demographics and Baseline Disease Characteristics

Demographics, baseline characteristics, prior anti-cancer therapies, and IDH1 and other mutation data, will be summarized for each cohort by treatment regimen for the Safety and Response Evaluable Populations using descriptive statistics.

BMI will be calculated as: weight  $(kg) / (height (m))^2$ 

Medical history information will be summarized for the Safety Population. Baseline Child-Pugh score and category (A, B, C) will be summarized within the baseline disease characteristics table for Cohorts 2 and 4. Hepatitis B and C status (positive or negative) will also be summarized within the baseline disease characteristics table. No formal statistical comparisons will be performed.

Medical history data will be coded via MedDRA. Prior anti-cancer therapies data will be coded via WHODrug.

In summarization of time since initial cancer diagnosis and months since recurrence, if a partial date is given in the data, month and day will be imputed as January and 01, respectively. Time since cancer diagnosis and months since recurrence will be derived as: informed consent date- date (diagnosis or recurrence) +1.

All demographic and baseline data for each patient will be provided in data listings. Prior radiotherapy and major surgical tumor resections will only be listed; they will not be summarized.

| Relevant Output | |
|---|---|
| Table 14.1.2.1a | Demographics and Baseline Characteristics (Cohort 1, Response Evaluable Population) |
| Table 14.1.2.1b | Demographics and Baseline Characteristics (Cohort 2, Response Evaluable Population) |
| Table 14.1.2.1c | Demographics and Baseline Characteristics (Cohort 3, Response Evaluable Population) |
| Table 14.1.2.1d | Demographics and Baseline Characteristics (Cohort 4, Response Evaluable Population) |
| Table 14.1.2.1e | Demographics and Baseline Characteristics (Cohort 5, Response Evaluable Population) |
| Table 14.1.2.2a | Demographics and Baseline Characteristics (Cohort 1, Safety Population) |
| Table 14.1.2.2b | Demographics and Baseline Characteristics (Cohort 2, Safety Population) |
| Table 14.1.2.2c | Demographics and Baseline Characteristics (Cohort 3, Safety Population) |
| Table 14.1.2.2d | Demographics and Baseline Characteristics (Cohort 4, Safety Population) |
| Table 14.1.2.2e | Demographics and Baseline Characteristics (Cohort 5, Safety Population) |
| Table 14.1.3.1a | Baseline Disease Characteristics (Cohort 1, Response Evaluable Population) |
| Table 14.1.3.1b | Baseline Disease Characteristics (Cohort 2, Response Evaluable Population) |
| Table 14.1.3.1c | Baseline Disease Characteristics (Cohort 3, Response Evaluable Population) |
| Table 14.1.3.1d | Baseline Disease Characteristics (Cohort 4, Response Evaluable Population) |

| Table 14.1.3.1e | Baseline Disease Characteristics (Cohort 5, Response Evaluable Population) |
|---|---|
| Table 14.1.3.2a Table 14.1.3.2b Table 14.1.3.2c Table 14.1.3.2d Table 14.1.3.2e | Baseline Disease Characteristics (Cohort 1, Safety Population) Baseline Disease Characteristics (Cohort 2, Safety Population) Baseline Disease Characteristics (Cohort 3, Safety Population) Baseline Disease Characteristics (Cohort 4, Safety Population) Baseline Disease Characteristics (Cohort 5, Safety Population) |
| Table 14.1.4.1a | IDH1 and Other Mutations (Cohort 1, Response Evaluable Population) |
| Table 14.1.4.1b | IDH1 and Other Mutations (Cohort 2, Response Evaluable Population) |
| Table 14.1.4.1c | IDH1 and Other Mutations (Cohort 3, Response Evaluable Population) |
| Table 14.1.4.1d | IDH1 and Other Mutations (Cohort 4, Response Evaluable Population) |
| Table 14.1.4.1e | IDH1 and Other Mutations (Cohort 5, Response Evaluable Population) |
| Table 14.1.4.2a Table 14.1.4.2b Table 14.1.4.2c Table 14.1.4.2d Table 14.1.4.2e | IDH1 and Other Mutations (Cohort 1, Safety Population) IDH1 and Other Mutations (Cohort 2, Safety Population) IDH1 and Other Mutations (Cohort 3, Safety Population) IDH1 and Other Mutations (Cohort 4, Safety Population) IDH1 and Other Mutations (Cohort 5, Safety Population) |
| Table 14.1.5.1a Table 14.1.5.1b Table 14.1.5.1c Table 14.1.5.1d Table 14.1.5.1e | Prior Therapies (Cohort 1, Response Evaluable Population) Prior Therapies (Cohort 2, Response Evaluable Population) Prior Therapies (Cohort 3, Response Evaluable Population) Prior Therapies (Cohort 4, Response Evaluable Population) Prior Therapies (Cohort 5, Response Evaluable Population) |
| Table 14.1.5.2a Table 14.1.5.2b Table 14.1.5.2c Table 14.1.5.2d Table 14.1.5.2e | Prior Therapies (Cohort 1, Safety Population) Prior Therapies (Cohort 2, Safety Population) Prior Therapies (Cohort 3, Safety Population) Prior Therapies (Cohort 4, Safety Population) Prior Therapies (Cohort 5, Safety Population) |
| Table 14.1.6a<br>Table 14.1.6b<br>Table 14.1.6c | Medical History (Cohort 1, Safety Population)<br>Medical History (Cohort 2, Safety Population)<br>Medical History (Cohort 3, Safety Population) |

| Table 14.1.6d | Medical History (Cohort 4, Safety Population) |
|-------------------|-----------------------------------------------|
| Table 14.1.6e | Medical History (Cohort 5, Safety Population) |
| Listing 16.2.4.1 | Demographics and Baseline Information |
| Listing 16.2.4.2 | Baseline Disease Data and Cancer Diagnosis |
| Listing 16.2.4.3 | IDH1 Mutation and Other Mutations |
| Listing 16.2.4.4 | Medical History |
| Listing 16.2.4.5 | Prior Anti-Cancer Therapies |
| Listing 16.2.4.6 | Prior Radiotherapy |
| Listing 16.2.4.7 | Major Surgical Tumor Resections |
| Listing 16.2.4.8 | Child-Pugh Score |
| Listing 16.2.4.9 | Hepatitis B and C |
| Listing 16.2.4.10 | Archival Tumor Tissue |

## 4.3. Efficacy Evaluations

### 4.3.1. Disease Response and Survival Analyses

In general, efficacy analyses will be conducted using the Response Evaluable population, with the exception of overall survival and the figure of time on treatment, which will be conducted on both the Response Evaluable and the Safety Population.

Best overall response and overall response rate will be summarized by cohort and treatment regimen (single agent or combination therapy) in the disease response assessment table. Disease response assessment will be further examined by subgroups, as described in Section 3.8. PFS, TTP, DOR, and TTR will be summarized by cohort and treatment regimen in another table. OS will be summarized for both the Response Evaluable and the Safety populations.

Time to event endpoints (OS, PFS, DOR) will be expressed as the number of weeks from first dose to the event and will be analyzed using Kaplan-Meier (KM) methods for each cohort. Censoring for each time to event endpoint is defined in Section 1.4.5. The median time to event will be presented along with the 95% confidence intervals, 1st and 3rd quartiles, and minimum and maximum values. The estimated probability of OS and PFS over time will be plotted as KM curves for each cohort and treatment regimen. The probability of survival for each cohort at 3, 6, 9, and 12 months will also be estimated using KM methods.

A plot of time on treatment (aka "swim plot") will be created for patients in the Safety Population to visualize the time on treatment. The plot will be color coded by best overall response. Time of first response (earliest response assessment where overall response was MR or better) will be annotated on the plot. Patients who are still receiving treatment with FT-2102 will be indicated with arrows at the end of the bar. Patients who are no longer receiving treatment with FT-2102 will have the reason for stopping FT-

2102 treatment annotated at the end of the bar. One plot will be created for each cohort and treatment regimen.

A waterfall plot will be produced for the Response Evaluable population to depict the best percentage change in the total tumor burden while on treatment. One bar will represent each patient, and they will be sorted by maximum percentage to least percentage. Each bar will be color coded by best overall response. One plot will be created for each cohort and treatment regimen. Total tumor burden is calculated as the sum of the longest diameter of each target lesion for RECIST assessments. Total tumor burden is calculated as the sum of the product of the diameters (longest diameter x perpendicular measurement) for all measurable lesions for RANO assessments. If a patient in Cohort 5 is evaluated by Cheson criteria, total tumor burden is calculated as the sum of the product diameters (longest diameter x perpendicular measurement) for all target lesions. Percent change for each follow up assessment is then calculated as the percent increase or decrease in total tumor burden from the screening imaging assessment.

Serum AFP, CA19-9, CEA are biomarkers indicative of response in Cohorts 2 and 4. They are not assessed in other cohorts. These markers will be summarized descriptively for the Response Evaluable population by cohort and visit. Additionally, box and whisker plots will be created for each parameter by cohort, visit, and responder status to compare change in responders vs non-responders over time.

### Relevant Output

| • | |
|---|---|
| Table 14.2.1a | Disease Response Assessment Overall and by Subgroup (Cohort 1, |
| | Response Evaluable Population) |
| Table 14.2.1b | Disease Response Assessment Overall and by Subgroup (Cohort 2, |
| | Response Evaluable Population) |
| Table 14.2.1c | Disease Response Assessment Overall and by Subgroup (Cohort 3, |
| | Response Evaluable Population) |
| Table 14.2.1d | Disease Response Assessment Overall and by Subgroup (Cohort 4, |
| | Response Evaluable Population) |
| Table 14.2.1e | Disease Response Assessment Overall and by Subgroup (Cohort 5, |
| | Response Evaluable Population) |
| Figure 14.2.2.1a | Best Percent Change from Baseline in Tumor Burden (Cohort 1 |
| | Single Agent, Response Evaluable Population) |
| Figure 14.2.2.2a | Best Percent Change from Baseline in Tumor Burden (Cohort 1 |
| | Combination Therapy, Response Evaluable Population) |
| Figure 14.2.2.1b | Best Percent Change from Baseline in Tumor Burden (Cohort 2 |
| | Single Agent, Response Evaluable Population) |
| Figure 14.2.2.2b | Best Percent Change from Baseline in Tumor Burden (Cohort 2 |
| | Combination Therapy, Response Evaluable Population) |

| Figure 14.2.2.1c | Best Percent Change from Baseline in Tumor Burden (Cohort 3<br>Single Agent, Response Evaluable Population) |
|---|---|
| Figure 14.2.2.2c | Best Percent Change from Baseline in Tumor Burden (Cohort 3 Combination Therapy, Response Evaluable Population) |
| Figure 14.2.2.1d | Best Percent Change from Baseline in Tumor Burden (Cohort 4<br>Single Agent, Response Evaluable Population) |
| Figure 14.2.2.2d | Best Percent Change from Baseline in Tumor Burden (Cohort 4<br>Combination Therapy, Response Evaluable Population) |
| Figure 14.2.2.1e | Best Percent Change from Baseline in Tumor Burden (Cohort 5, Response Evaluable Population) |
| Figure 14.2.3.1a | Time on Treatment (Cohort 1 Single Agent, Safety Population) |
| Figure 14.2.3.2a | Time on Treatment (Cohort 1 Combination Therapy, Safety Population) |
| Figure 14.2.3.1b | Time on Treatment (Cohort 2 Single Agent, Safety Population) |
| Figure 14.2.3.2b | Time on Treatment (Cohort 2 Combination Therapy, Safety Population) |
| Figure 14.2.3.1c | Time on Treatment (Cohort 3 Single Agent, Safety Population) |
| Figure 14.2.3.2c | Time on Treatment (Cohort 3 Combination Therapy, Safety Population) |
| Figure 14.2.3.1d | Time on Treatment (Cohort 4 Single Agent, Safety Population) |
| Figure 14.2.3.2d | Time on Treatment (Cohort 4 Combination Therapy, Safety Population) |
| Figure 14.2.3.1e | Time on Treatment (Cohort 5, Safety Population) |
| Table 14.2.4a | Progression-Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 1, Response Evaluable Population) |
| Table 14.2.4b | Progression-Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 2, Response Evaluable Population) |
| Table 14.2.4c | Progression-Free Survival, Time to Progression, Duration of |
| 12.10 | Response, and Time to Response (Cohort 3, Response Evaluable Population) |
| Table 14.2.4d | Progression-Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 4, Response Evaluable Population) |
| Table 14.2.4e | Progression-Free Survival, Time to Progression, Duration of<br>Response, and Time to Response (Cohort 5, Response Evaluable<br>Population) |

| Table 14.2.5.1<br>Table14.2.5.2 | Overall Survival (Response Evaluable Population)<br>Overall Survival (Safety Population) |
|---|---|
| Figure 14.2.5.3a | Kaplan-Meier Plot of Overall Survival (Cohort 1, Response Evaluable Population) |
| Figure 14.2.5.3b | Kaplan-Meier Plot of Overall Survival (Cohort 2, Response Evaluable Population) |
| Figure 14.2.5.3c | Kaplan-Meier Plot of Overall Survival (Cohort 3, Response Evaluable Population) |
| Figure 14.2.5.3d | Kaplan-Meier Plot of Overall Survival (Cohort 4, Response Evaluable Population) |
| Figure 14.2.5.3e | Kaplan-Meier Plot of Overall Survival (Cohort 5, Response Evaluable Population) |
| Figure 14.2.5.4a | Kaplan-Meier Plot of Overall Survival (Cohort 1, Safety Population) |
| Figure 14.2.5.4b | Kaplan-Meier Plot of Overall Survival (Cohort 2, Safety Population) |
| Figure 14.2.5.4c | Kaplan-Meier Plot of Overall Survival (Cohort 3, Safety Population) |
| Figure 14.2.5.4d | Kaplan-Meier Plot of Overall Survival (Cohort 4, Safety Population) |
| Figure 14.2.5.4e | Kaplan-Meier Plot of Overall Survival (Cohort 5, Safety Population) |
| Figure 14.2.5.5a | Kaplan-Meier Plot of Progression Free Survival (Cohort 1, Response Evaluable Population) |
| Figure 14.2.5.5b | Kaplan-Meier Plot of Progression Free Survival (Cohort 2, Response Evaluable Population) |
| Figure 14.2.5.5c | Kaplan-Meier Plot of Progression Free Survival (Cohort 3, Response Evaluable Population) |
| Figure 14.2.5.5d | Kaplan-Meier Plot of Progression Free Survival (Cohort 4, Response Evaluable Population) |
| Figure 14.2.5.5e | Kaplan-Meier Plot of Progression Free Survival (Cohort 5, Response Evaluable Population) |
| Figure 14.2.5.6a | Kaplan-Meier Plot of Progression Free Survival (Cohort 1, Safety Population) |
| Figure 14.2.5.6b | Kaplan-Meier Plot of Progression Free Survival (Cohort 2, Safety Population) |

| Figure 14.2.5.6c | Kaplan-Meier Plot of Progression Free Survival (Cohort 3, Safety Population) |
|---|---|
| Figure 14.2.5.6d | Kaplan-Meier Plot of Progression Free Survival (Cohort 4, Safety Population) |
| Figure 14.2.5.6e | Kaplan-Meier Plot of Progression Free Survival (Cohort 5, Safety Population) |
| Table 14.2.6a | Serum AFP, CA19-9, CEA (Cohort 2, Response Evaluable Population) |
| Table 14.2.6b | Serum AFP, CA19-9, CEA (Cohort 4, Response Evaluable Population) |
| Figure 14.2.7a | Serum AFP, CA19-9, CEA (Cohort 2, Response Evaluable Population) |
| Figure 14.2.7b | Serum AFP, CA19-9, CEA (Cohort 4, Response Evaluable Population) |
| Listing 16.2.6.1 | Target Lesions (RECIST) |
| Listing 16.2.6.2 | Non-Target and New Lesions (RECIST) |
| Listing 16.2.6.3 | Measurable Lesions (RANO) |
| Listing 16.2.6.4 | Non-Measurable and New Lesions (RANO) |
| Listing 16.2.6.5 | Response Assessment (RECIST) |
| Listing 16.2.6.6 | Response Assessment (RANO and LGG RANO) |
| Listing 16.2.6.7 | Response Assessment (Cheson) |
| Listing 16.2.6.8 | Survival Status |
| Listing 16.2.6.9 | Serum AFP, CA19-9, CEA |

### 4.3.2. Quality of Life Assessment Analysis

The EQ-5D-5L is a validated assessment of the quality of life which consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of one's health state: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient indicates his/her health state by selecting the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

EQ-5D-5L data will be summarized by nominal visit for the Response Evaluable Population. The number and percentage of patients reporting each score per dimension will be summarized, as well as the number reporting some problems on that dimension (score >1). The change from baseline in the number reporting some problems in each dimension will also be reported (raw and percent change). Furthermore, a stacked bar

chart will be produced to illustrate the EQ-5D-5L values. In the chart, the x axis will represent nominal visit (screening, cycle 3, and end of treatment) and the y axis will represent percentage. Each bar will add to 100% and be color coded to represent the percent of patients reporting each level (1-5) of problems within the dimension for that visit. A table below the figure will show the number of patients contributing data to each visit. A separate chart will be created for each of the dimensions. This figure will be created for each cohort and treatment regimen.

#### All EO-5D-5L data will be listed.

| EQ-5D-5L Summary (Cohort 1, Response Evaluable Population) |
|------------------------------------------------------------|
| EQ-5D-5L Summary (Cohort 2, Response Evaluable Population) |
| EQ-5D-5L Summary (Cohort 3, Response Evaluable Population) |
| EQ-5D-5L Summary (Cohort 4, Response Evaluable Population) |
| EQ-5D-5L Summary (Cohort 5, Response Evaluable Population) |
| EQ-5D-5L Quality of Life Assessment (Cohort 1, Response |
| Evaluable Population) |
| EQ-5D-5L Quality of Life Assessment (Cohort 2, Response |
| Evaluable Population) |
| EQ-5D-5L Quality of Life Assessment (Cohort 3, Response |
| Evaluable Population) |
| EQ-5D-5L Quality of Life Assessment (Cohort 4, Response |
| Evaluable Population) |
| EQ-5D-5L Quality of Life Assessment (Cohort 5, Response |
| Evaluable Population) |
| EQ5D-5L Quality of Life Assessment |

# 4.4. Pharmacokinetic and Pharmacodynamic Evaluations

Pharmacokinetic analyses will be conducted using the PK population. Pharmacodynamic analyses will be conducted on the 2-HG biomarker using the Pharmacodynamic population.

Evaluation of 2-HG has been done in a number of types of biological samples for this study: plasma, urine, and for glioma patients magnetic resonance spectroscopy (MRS) evaluation of 2-HG in tumor tissue, and cerebral spinal fluid. Each of these types of 2-HG evaluations will be summarized separately; they will not be combined. 2-HG will be summarized for each disease cohort and treatment regimen by actual value, change from baseline, and percent change by nominal visit. In such tables, unscheduled visit results will not be included. Furthermore, 2-HG will also be summarized by subgroup. Percent change from baseline will be plotted in a box plot where the x-axis will represent nominal visit and the y-axis will represent percent change from baseline, and separate boxes will be plotted for sample type (plasma, tumor tissue, CSF, urine). Separate figures will be produced for each cohort.

Pharmacokinetic variables will be calculated from the plasma concentration data using standard non-compartmental methods. The pharmacokinetic variables to be determined are summarized below:

Table 1 Pharmacokinetic Parameters for Analysis

| Parameter | Description |
|---|---|
| AUC <sub>all</sub> | Area under the concentration versus time curve from Time 0 (pre-dose) to the last quantifiable concentration; calculated using the linear-log trapezoidal method. |
| AUC <sub>tau</sub> | Area under the concentration versus time curve over the dosing interval at steady-state; calculated using the linear-log trapezoidal method. |
| $C_{min}$ | The trough plasma concentration taken prior to a subsequent dose. |
| $C_{max}$ | Maximum plasma concentration; the highest concentration observed during a dosage interval. |
| $T_{\text{max}}$ | The time $C_{max}$ was observed. |

FT-2102 concentrations below the lower limit of quantitation (LLOQ) will be indicated by BLQ in the listings and will be treated as follows:

• For pre-dose samples prior to the FT-2102 administration: Concentrations that are BLQ or missing will be assigned a numerical value of zero for the calculation of AUC. Any anomalous concentration values observed at pre-dose will be included in the computation of AUC. If the pre-dose concentration is greater than 5% of C<sub>max</sub>, the data will be evaluated on a case-by-case basis to determine if exclusion of the affected profile is warranted.

For all other BLQ concentrations: Any other BLQ concentrations will be assigned a value of zero if they precede quantifiable samples in the initial portion of the concentration-time profile. A BLQ value that occurs between quantifiable data points, especially prior to  $C_{max}$ , will be evaluated to determine if an assigned concentration of zero makes sense, or if exclusion of the data is warranted. Following  $C_{max}$ , BLQ values embedded between 2 quantifiable data points will be treated as missing when calculating AUC. If BLQ values occur at the end of the collection interval (after the last quantifiable concentration), these will be set to zero. If consecutive BLQ concentrations are followed by quantifiable concentrations in the terminal portion of the concentration curve, these quantified values will be excluded from the PK analysis by setting them to missing, unless otherwise warranted by the concentration-time profile.

Pharmacokinetic concentration data will be listed by patient including actual sampling times relative to dosing. Plasma concentrations will be summarized by disease cohort, treatment regimen, and nominal visit. The following descriptive statistics will be presented at each nominal time point: n, arithmetic mean, standard deviation, coefficient of variation (CV%), geometric mean, geometric standard deviation, geometric CV%, median, minimum and maximum values.

For each cohort, the individual plasma concentration versus actual time profiles for each patient, as well as the geometric mean plasma concentration versus nominal time profiles will be presented graphically on a linear-linear and log-linear scale.

The following PK parameters will be listed by patient and summarized by disease cohort, and treatment regimen. Descriptive statistics for calculated PK parameters will include: n, arithmetic mean, standard deviation, CV%, geometric mean, median, minimum and maximum values. No descriptive statistics will be presented for an individual PK parameter when fewer than three patients have values for that parameter.

All plasma and CSF (if any) concentration and pharmacodynamic data and the per-patient pharmacokinetic parameters will be displayed in data listings.

| Table 14.2.10.1a | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 1, PD Population) |
|---|---|
| Table 14.2.10.1b | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 2, PD Population) |
| Table 14.2.10.1c | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 3, PD Population) |
| Table 14.2.10.1d | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 4, PD Population) |
| Table 14.2.10.1e | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 5, PD Population) |
| Table 14.2.10.2a | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 1, PD Population) |
| Table 14.2.10.2b | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 2, PD Population) |
| Table 14.2.10.2c | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 3, PD Population) |
| Table 14.2.10.2d | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 4, PD Population) |
| Table 14.2.10.2e | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 5, PD Population) |
| Figure 14.2.11.1a | Boxplot of Plasma 2-HG by Time Point (Cohort 1, PD Population) |
| Figure 14.2.11.1b<br>Figure 14.2.11.1c | Boxplot of Plasma 2-HG by Time Point (Cohort 2, PD Population)<br>Boxplot of Plasma 2-HG by Time Point (Cohort 3, PD Population) |
| Figure 14.2.11.1d | Boxplot of Plasma 2-HG by Time Point (Cohort 4, PD Population) |
| Figure 14.2.11.1e | Boxplot of Plasma 2-HG by Time Point (Cohort 5, PD Population) |
| Figure 14.2.11.2a | Boxplot of Urine 2-HG by Time Point (Cohort 1, PD Population) |
| Figure 14.2.11.2b<br>Figure 14.2.11.2c | Boxplot of Urine 2-HG by Time Point (Cohort 2, PD Population) Boxplot of Urine 2-HG by Time Point (Cohort 3, PD Population) |
| Figure 14.2.11.2d | Boxplot of Urine 2-HG by Time Point (Cohort 4, PD Population) |
| Figure 14.2.11.2e | Boxplot of Urine 2-HG by Time Point (Cohort 5, PD Population) |

| Figure 14.2.11.3 | Boxplot of Tumor 2-HG Assessed by MRS by Time Point (Cohort 1, PD Population) |
|---|---|
| Figure 14.2.11.4 | Boxplot of CSF 2-HG by Time Point (Cohort 1, PD Population) |
| Table 14.2.12a | FT-2102 Plasma Concentration over Time (Cohort 1, PK Population) |
| Table 14.2.12b | FT-2102 Plasma Concentration over Time (Cohort 2, PK Population) |
| Table 14.2.12c | FT-2102 Plasma Concentration over Time (Cohort 3, PK Population) |
| Table 14.2.12d | FT-2102 Plasma Concentration over Time (Cohort 4, PK Population) |
| Table 14.2.12e | FT-2102 Plasma Concentration over Time (Cohort 5, PK Population) |
| Table 14.2.13a | Summary of Pharmacokinetic Parameters (All Patients on Single Agent Therapy, PK Population) |
| Table 14.2.13b | Summary of Pharmacokinetic Parameters (Cohort 1, PK Population) |
| Table 14.2.13c | Summary of Pharmacokinetic Parameters (Cohort 2, PK Population) |
| Table 14.2.13d | Summary of Pharmacokinetic Parameters (Cohort 3, PK Population) |
| Table 14.2.13e | Summary of Pharmacokinetic Parameters (Cohort 4, PK Population) |
| Table 14.2.13f | Summary of Pharmacokinetic Parameters (Cohort 5, PK Population) |
| Figure 14.2.14.1a | Geometric Mean FT-2102 Plasma Concentration over Time (Cohort 1, PK Population) |
| Figure 14.2.14.1b | Geometric Mean FT-2102 Plasma Concentration over Time (Cohort 2, PK Population) |
| Figure 14.2.14.1c | Geometric Mean FT-2102 Plasma Concentration over Time (Cohort 3, PK Population) |
| Figure 14.2.14.1d | Geometric Mean FT-2102 Plasma Concentration over Time (Cohort 4, PK Population) |
| Figure 14.2.14.1e | Geometric Mean FT-2102 Plasma Concentration over Time (Cohort 5, PK Population) |
| Figure 14.2.14.2a | Geometric Mean FT-2102 Plasma Concentration over Log-Time (Cohort 1, PK Population) |
|---|---|
| Figure 14.2.14.2b | Geometric Mean FT-2102 Plasma Concentration over Log-Time (Cohort 2, PK Population) |
| Figure 14.2.14.2c | Geometric Mean FT-2102 Plasma Concentration over Log-Time (Cohort 3, PK Population) |
| Figure 14.2.14.2d | Geometric Mean FT-2102 Plasma Concentration over Log-Time (Cohort 4, PK Population) |
| Figure 14.2.14.2e | Geometric Mean FT-2102 Plasma Concentration over Log-Time (Cohort 5, PK Population) |
| Figure 14.2.15a | FT-2102 Geometric Mean Plasma Concentration over Nominal Time (All Patients on Single Agent Therapy, PK Population) |
| Figure 14.2.15b | FT-2102 Geometric Mean Plasma Concentration over Nominal Time (Cohort 1, PK Population) |
| Figure 14.2.15c | FT-2102 Geometric Mean Plasma Concentration over Nominal Time (Cohort 2, PK Population) |
| Figure 14.2.15d | FT-2102 Geometric Mean Plasma Concentration over Nominal Time (Cohort 3, PK Population) |
| Figure 14.2.15e | FT-2102 Geometric Mean Plasma Concentration over Nominal Time (Cohort 4, PK Population) |
| Figure 14.2.15f | FT-2102 Geometric Mean Plasma Concentration over Nominal Time (Cohort 5, PK Population) |
| Listing 16.2.5.4<br>Listing 16.2.5.5<br>Listing 16.2.6.11<br>Listing 16.2.6.12<br>Listing 16.2.6.13 | Pharmacokinetic Concentrations Pharmacokinetic Parameters 2-HG MRS Assessments Archival Tumor Tissue and Tumor Biopsy Pharmacogenomics Samples |

### 4.5. Safety Analyses

Safety analyses will be conducted using the Safety population. In tables summarizing data by cycle, only cycles with 3 or more patients having data for the cycle will be summarized.

#### 4.5.1. Study Drug Exposure

Study drug exposure will be characterized by duration of exposure, amount of exposure, and percent compliance. Additionally, in the summary table containing duration of exposure, the number of patients and events of the following types will be summarized: dose reduced, dose increased, dose held, drug withdrawn, and non-compliance. These parameters will be calculated over all for the study and summarized by cohort. Amount of exposure and percent compliance will also be calculated by cycle and tabulated. Additionally, these parameters will be listed, along with raw data from the exposure and drug accountability logs.

<u>Duration of FT-2102 Exposure:</u> Duration of study drug exposure to FT-2102 will be calculated as the number of days that patients were administered study drug, as determined below, and will be summarized by treatment group using descriptive statistics.

 $Duration \ of \ Study \ Drug \ Exposure = (Date \ of \ lastdose - Date of firstdose) + 1$ 

Total assigned dose (mg): For each cycle, the total assigned dose will be calculated for each log line in the FT-2102 administration form as: total assigned dose= (assigned dose\*1 (if frequency=QD) or assigned dose\*2 if frequency=BID)\*number of days comprising the log line (eg. End date-start date+1). To get the total assigned dose for the cycle, the sum of the log lines within the cycle will be calculated. To get the total assigned dose for the study, the sum of the total assigned dose for all cycles will be calculated.

<u>Total dose not taken and not returned (mg)</u>: This will be calculated from the drug accountability log. This will be calculated by taking the number of pills dispensed (last cycle)-number of pills returned (this cycle)-doses taken per patient diary (this cycle). That yields the number of pills taken and not returned, to get the dose taken and not returned, multiply the number of pills taken and not returned by the pill strength.

Total dose taken (mg): for each cycle the total dose taken will be calculated based on the drug accountability log. The number of tablets dispensed times the tablet strength (50 or 150 mg) will yield the total dose dispensed and the number of tablets returned times the tablet strength will yield the total dose returned. Total dose taken equals total dose dispensed minus total dose returned minus total dose not taken and not returned. This will be calculated by cycle, and then the sum of all cycles will yield the total dose taken for the study.

<u>Percent compliance</u>: percent compliance will be calculated by cycle and overall for the study. It is calculated as the total assigned dose-total dose taken, divided by total assign

Percent compliance= (total assigned dose - (total assigned dose-total dose taken)) \*100 total assigned dose

For patients receiving combination therapy, the combination drugs are administered via IV or SC. Duration of treatment with combination agents and duration of total treatment including IV therapy and oral therapy (in days) will be presented by treatment group for the Safety and Response Evaluable populations, where duration of treatment is calculated as the end date minus the start date plus 1. Descriptive statistics (both continuous and categorical) will also be presented for the number of doses received for IV therapy. The number of patients who experienced dose interruptions will be tabulated, as well as the reason for the interruption (e.g., adverse event, other reason).

Dosing information for each patient will be presented in a data listing.

### Relevant Output

| Table 14.2.16.1a | Study Drug Exposure (Cohort 1, Response Evaluable Population) |
|---|---|
| Table 14.2.16.1b | Study Drug Exposure (Cohort 2, Response Evaluable Population) |
| Table 14.2.16.1c | Study Drug Exposure (Cohort 3, Response Evaluable Population) |
| Table 14.2.16.1d | Study Drug Exposure (Cohort 4, Response Evaluable Population) |
| Table 14.2.16.1e | Study Drug Exposure (Cohort 5, Response Evaluable Population) |
| Table 14.2.16.2a | Study Drug Exposure (Cohort 1, Safety Population) |
| Table 14.2.16.2b | Study Drug Exposure (Cohort 2, Safety Population) |
| Table 14.2.16.2c | Study Drug Exposure (Cohort 3, Safety Population) |
| Table 14.2.16.2d | Study Drug Exposure (Cohort 4, Safety Population) |
| Table 14.2.16.2e | Study Drug Exposure (Cohort 5, Safety Population) |
| Table 14.2.17a | Study Drug Exposure to Azacitidine (Cohort 1, Safety Population) |
| Table 14.2.17b | Study Drug Exposure to Nivolumab (Cohort 2, Safety Population) |
| Table 14.2.17c | Study Drug Exposure to Azacitidine (Cohort 3, Safety Population) |
| Table 14.2.17d | Study Drug Exposure to Gemcitabine and Cisplatin (Cohort 4, |
| | Safety Population) |
| Listing 16.2.5.1 | FT-2102 Administration |
| Listing 16.2.5.2 | Drug Accountability |
| Listing 16.2.5.3 | Azacitidine, Nivolumab, Cisplatin, and Gemcitibine |
| | Administration |

#### 4.5.2. Adverse Events

All AEs will be coded using the MedDRA coding system and displayed in tables and data listings using system organ class (SOC) and preferred term.

Analyses of adverse events will be performed for those events that are considered treatment-emergent. A treatment-emergent adverse event (TEAE) is an AE that begins or worsens in the period from the first dose of study treatment to 28 days after the last dose of study drug. Study drug is defined as FT-2102 or, for patients assigned to receive combination therapy, azacitidine, nivolumab, gemcitabine, or cisplatin.

Adverse events are summarized by patient incidence rates; therefore, in any tabulation, a patient contributes only once to the count for a given adverse event, SOC, or preferred term.

The number and percentage of patients with any treatment-emergent adverse event, with any treatment-emergent adverse event assessed by the Investigator as related to treatment (definite, probable, or possible relationship), and with any serious adverse event will be summarized by treatment group and overall. In these tabulations, each patient will contribute only once (i.e., the most related occurrence or the most intense occurrence) to each of the incidence rates in the descriptive analysis, regardless of the number of episodes.

An additional summary of TEAEs will be produced in which MedDRA PTs are presented, sorted from most frequent to least.

No formal hypothesis-testing analysis of adverse event incidence rates will be performed.

All adverse events gathered in the clinical database, whether treatment emergent or not, will be listed in patient data listings.

By-patient listings also will be provided for the following: patient deaths, serious adverse events, adverse events leading to withdrawal, and dose-limiting toxicities.

### Relevant Output

| 11010 01110 0 010 010 | |
|---|---|
| Table 14.3.1.1a | Summary of Treatment-Emergent Adverse Events, Overall and by |
| | Dose Group (Cohort 1, Safety Population) |
| Table 14.3.1.1b | Summary of Treatment-Emergent Adverse Events, Overall and by |
| | Dose Group (Cohort 2, Safety Population) |
| Table 14.3.1.1c | Summary of Treatment-Emergent Adverse Events, Overall and by |
| | Dose Group (Cohort 3, Safety Population) |
| Table 14.3.1.1d | Summary of Treatment-Emergent Adverse Events, Overall and by |
| | Dose Group (Cohort 4, Safety Population) |
| Table 14.3.1.1e | Summary of Treatment-Emergent Adverse Events, Overall and by |
| | Dose Group (Cohort 5, Safety Population) |
| Table 14.3.1.a | Treatment-Emergent Adverse Events by MedDRA System Organ |
| | Class and Preferred Term (All Patients Receiving Single Agent |
| | Therapy, Safety Population) |
| | /r J, ~ J - ~ r/ |

| Table 14.3.1.b | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (All Patients Receiving Combination<br>Therapy, Safety Population) |
|---|---|
| Table 14.3.1.c | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (All Patients, Safety Population) |
| Table 14.3.1.d | Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Cohort 1, Safety Population) |
| Table 14.3.1.e | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 2, Safety Population) |
| Table 14.3.1.2f | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 3, Safety Population) |
| Table 14.3.1.g | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 4, Safety Population) |
| Table 14.3.1.h | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 5, Safety Population) |
| Table 14.3.1.3a | Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 1, Safety Population) |
| Table 14.3.1.3b | Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 2, Safety Population) |
| Table 14.3.1.3c | Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 3, Safety Population) |
| Table 14.3.1.3d | Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 4, Safety Population) |
| Table 14.3.1.3e | Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 5, Safety Population) |
| Table 14.3.1.4a | Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Cohort 1, Safety Population) |
| Table 14.3.1.4b | Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Cohort 2, Safety Population) |
| Table 14.3.1.4c | Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Cohort 3, Safety Population) |
| Table 14.3.1.4d | Severe Treatment-Emergent Adverse Events by MedDRA System<br>Organ Class and Preferred Term (Cohort 4, Safety Population) |

| Table 14.3.1.4e | Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Cohort 5, Safety Population) |
|---|---|
| Table 14.3.1.5a | Severe Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 1, Safety Population) |
| Table 14.3.1.5b | Severe Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 2, Safety Population) |
| Table 14.3.1.5c | Severe Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 3, Safety Population) |
| Table 14.3.1.5d | Severe Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 4, Safety Population) |
| Table 14.3.1.5e | Severe Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 5, Safety Population) |
| Table 14.3.1.6a | TEAEs by MedDRA Preferred Term (Cohort 1, Safety Population) |
| Table 14.3.1.6b | TEAEs by MedDRA Preferred Term (Cohort 2, Safety Population) |
| Table 14.3.1.6c | TEAEs by MedDRA Preferred Term (Cohort 3, Safety Population) |
| Table 14.3.1.6d | TEAEs by MedDRA Preferred Term (Cohort 4, Safety Population) |
| Table 14.3.1.6e | TEAEs by MedDRA Preferred Term (Cohort 5, Safety Population) |
| Table 14.3.2.1 | Listing of Deaths |
| Table 14.3.2.2 | Listing of Serious Adverse Events |
| Table 14.3.2.3 | Listing of Adverse Events Resulting in Drug Interruptions or Withdrawals |
| Table 14.3.2.4 | Listing of Dose-Limiting Toxicities |
| Listing 16.2.7.1 | Adverse Events by Patient and Verbatim Term |
| Listing 16.2.7.2 | Adverse Events by Patient and MedDRA System Organ Class and Preferred Term |
| Listing 16.2.7.3 | Adverse Events by MedDRA System Organ Class, Preferred Term, Cohort, and Patient |

### 4.5.3. Laboratory Data

Clinical laboratory values (including hematology, coagulation, chemistry, and urinalysis) will be expressed in SI units. CTCAE v 4.03 grading will be applied to laboratory values (for laboratory tests that are graded by CTCAE). In cases where a laboratory reports only hematology differentials in percentage, the absolute values may be derived

programmatically for reporting. The derivation of the absolute value would be calculated by taking the percent of the absolute WBC value.

The actual value and change from baseline to each on-study evaluation will be summarized for each clinical laboratory parameter, including hematology and clinical chemistry. In the event of repeat values, the last non-missing value per study day/time will be used. Unscheduled laboratory draws will not be included in these summaries. Coagulation labs are only drawn pre-treatment, and so will be combined with the hematology table for applicable visits.

Shifts from baseline to worst CTCAE grade experienced on study will be presented. In cases where CTCAE grades may be bi-directional (i.e., sodium, potassium), shifts to highest value and lowest value will be presented. Unscheduled laboratory draws will be included in the consideration of worst value on study.

A separate summary of liver function test abnormalities will be produced, based on the FDA's guidance for industry on drug induced liver injury (June 2009), in addition to the summaries described above. The number and percentage of patients experiencing the following abnormalities will be summarized for the Safety analysis set. A supportive listing of this data will also be produced illustrating which values have received flags applied to this table.

| Clinical Laboratory Parameter | Category |
|---|---|
| ALT | >3 × ULN; >5 × ULN; >10 × ULN; >20 × ULN |
| AST | >3 × ULN; >5 × ULN; >10 × ULN; >20 × ULN |
| AST or ALT | >3 × ULN; >5 × ULN; >10 × ULN; >20 × ULN |
| Total Bilirubin (TBL) | >1.5 × ULN; ≥2 × ULN |
| ALP | >2.5 × ULN; >5 x ULN |
| Concurrent AST, ALT and Total Bilirubin | (ALT or AST >3 x ULN) and (TBL >1.5 x ULN); |
| | (ALT or AST >3 x ULN) and (TBL >2 x ULN) |
| Concurrent AST, ALT and Total Bilirubin | (ALT or AST >3 x ULN) and (TBL >1.5 x ULN); |
| without ALP abnormality | (ALT or AST >3 x ULN) and (TBL >2 x ULN) |
| ALT>3 x ULN or AST>3 x ULN with<br>Concurrent report of selected TEAEs during<br>study | (ALT > 3 x ULN) or (AST >3 x ULN and with TEAEs* |

<sup>\*</sup>Selected TEAEs include nausea, vomiting, anorexia, abdominal pain, abdominal discomfort, fatigue, jaundice, pruritus, chromaturia, and feces discolored.

Concurrent test values are defined as post-baseline values measured within +/- 7 days of test dates for the related parameters.

All laboratory data will be provided in data listings, and will be flagged with CTCAE grade if applicable, and H or L if above or below the normal limit.

Subset listings will be presented for all abnormal laboratory values and laboratory values with CTCAE severity grade 3 or 4.

| Relevant Output | |
|---|---|
| Table 14.3.4.1 | Listing of Abnormal Laboratory Values |
| Table 14.3.4.2 | Listing of Laboratory Values with CTCAE Severity ≥Grade 3 |
| Table 14.3.4.3 | Listing of Liver Function Tests of Potential Concern |
| Table 14.3.5.1a | Summary and Change from Baseline for Hematology and Coagulation Parameters by Time Point, Overall and by Dose Group (Cohort 1, Safety Population) |
| Table 14.3.5.1b | Summary and Change from Baseline for Hematology and<br>Coagulation Parameters by Time Point, Overall and by Dose<br>Group (Cohort 2, Safety Population) |
| Table 14.3.5.1c | Summary and Change from Baseline for Hematology and<br>Coagulation Parameters by Time Point, Overall and by Dose<br>Group (Cohort 3, Safety Population) |
| Table 14.3.5.1d | Summary and Change from Baseline for Hematology and Coagulation Parameters by Time Point, Overall and by Dose Group (Cohort 4, Safety Population) |
| Table 14.3.5.1e | Summary and Change from Baseline for Hematology and<br>Coagulation Parameters by Time Point, Overall and by Dose<br>Group (Cohort 5, Safety Population) |
| Table 14.3.5.2a | Summary and Change from Baseline for Chemistry Parameters by Time Point, Overall and by Dose Group (Cohort 1, Safety Population) |
| Table 14.3.5.2b | Summary and Change from Baseline for Chemistry Parameters by Time Point, Overall and by Dose Group (Cohort 2, Safety Population) |
| Table 14.3.5.2c | Summary and Change from Baseline for Chemistry Parameters by Time Point, Overall and by Dose Group (Cohort 3, Safety Population) |
| Table 14.3.5.2d | Summary and Change from Baseline for Chemistry Parameters by<br>Time Point, Overall and by Dose Group (Cohort 4, Safety<br>Population) |
| Table 14.3.5.2e | Summary and Change from Baseline for Chemistry Parameters by<br>Time Point, Overall and by Dose Group (Cohort 5, Safety<br>Population) |
| Table 14.3.6.1a | Shifts from Baseline to Worst Value on Study in Hematology and Coagulation, Overall and by Dose Group (Cohort 1, Safety Population) |

| Shifts from Baseline to Worst Value on Study in Hematology and Coagulation, Overall and by Dose Group (Cohort 2, Safety |
|---|
| Population) |
| Shifts from Baseline to Worst Value on Study in Hematology and Coagulation, Overall and by Dose Group (Cohort 3, Safety Population) |
| Shifts from Baseline to Worst Value on Study in Hematology and Coagulation, Overall and by Dose Group (Cohort 4, Safety Population) |
| Shifts from Baseline to Worst Value on Study in Hematology and Coagulation, Overall and by Dose Group (Cohort 5, Safety Population) |
| Shifts from Baseline to Worst Value on Study in Chemistry,<br>Overall and by Dose Group (Cohort 1, Safety Population) |
| Shifts from Baseline to Worst Value on Study in Chemistry,<br>Overall and by Dose Group (Cohort 2, Safety Population) |
| Shifts from Baseline to Worst Value on Study in Chemistry,<br>Overall and by Dose Group (Cohort 3, Safety Population) |
| Shifts from Baseline to Worst Value on Study in Chemistry,<br>Overall and by Dose Group (Cohort 4, Safety Population) |
| Shifts from Baseline to Worst Value on Study in Chemistry,<br>Overall and by Dose Group (Cohort 5, Safety Population) |
| Summary of Liver Function Test Results (All Patients Receiving Single Agent Therapy, Safety Population) |
| Summary of Liver Function Test Results (Cohort 1, Safety Population) |
| Summary of Liver Function Test Results (Cohort 2, Safety Population) |
| Summary of Liver Function Test Results (Cohort 3, Safety Population) |
| Summary of Liver Function Test Results (Cohort 4, Safety Population) |
| Summary of Liver Function Test Results (Cohort 5, Safety Population) |
| Laboratory Results: Hematology |
| Laboratory Results: Chemistry |
| Laboratory Results: Urinalysis |
| Laboratory Results: Coagulation |
| Laboratory Normal Ranges |
| Laboratory Results: Other Screening Tests and Pregnancy Tests |

#### 4.5.4. Vital Signs and Physical Examination

The actual value and change from baseline to each on-study evaluation will be summarized for vital signs.

Vital sign measurements will be presented for each patient in a data listing.

All physical examinations will be presented in a data listing.

#### Relevant Output

| Table 14.3.8a | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 1, Safety Population) |
|---|---|
| Table 14.3.8b | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 2, Safety Population) |
| Table 14.3.8c | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 3, Safety Population) |
| Table 14.3.8d | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 4, Safety Population) |
| Table 14.3.8e | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 5, Safety Population) |
| Listing 16.2.9.1<br>Listing 16.2.9.2 | Vital Signs Physical Examinations |

#### 4.5.5. Electrocardiogram

Electrocardiogram results will be summarized descriptively, including the number and percentage of patients with normal, abnormal, and clinically significant abnormal results at baseline and each study visit.

In addition, the number and percentage of patient experiencing the following events will be tabulated and summarized by baseline QTcF ( $<450, \ge 450$  to  $\le 480, \ge 481$  to  $\le 500, \ge 501$ ):

Absolute change from baseline in QTcF at any time during study

- >30 to <60 msec
- >60 msec

Reaching a value in QTcF at any time during study

- $\geq$ 450 to  $\leq$ 480 msec
- $\geq$ 481 to  $\leq$ 500 msec
- $\geq$ 501 msec

A scatter plot will also be produced which plots a single dot for each patient in the Safety set. It will plot the patient's baseline QTcF on the x axis and the maximum post baseline QTcF on the Y axis. Reference lines will be shown at 450 on both axes. Electrocardiogram data for each patient will be provided in a data listing.

### Relevant Output

| Electrocardiogram Results (Cohort 1, Safety Population) |
|---------------------------------------------------------------------|
| Electrocardiogram Results (Cohort 2, Safety Population) |
| Electrocardiogram Results (Cohort 3, Safety Population) |
| Electrocardiogram Results (Cohort 4, Safety Population) |
| Electrocardiogram Results (Cohort 5, Safety Population) |
| QTcF Shifts from Baseline (Single Agent Therapy, Safety Population) |
| QTcF Shifts from Baseline (Combination Therapy, Safety |
| Population) |
| Maximum Post Baseline QTcF vs Baseline QTcF (Single Agent |
| Therapy, Safety Population) |
| Maximum Post Baseline QTcF vs Baseline QTcF (Combination |
| Therapy, Safety Population) |
| Electrocardiogram Results |

#### 4.5.6. Concomitant Medications and Procedures

Concomitant medication is a medication taken during the treatment period. It will be operationally defined as any medication with a start date prior to the date of the first dose of study treatment and continuing after the first dose of study treatment or with a start date between the dates of the first and last dose of study treatment. Any medication with a start date after the date of the last dose of study treatment will not be considered a concomitant medication. Any medication with a start and end date before the first dose of study treatment will be considered a prior medication. Concomitant medications will be coded using the WHO Drug Dictionary. Results will be tabulated by anatomic therapeutic class (ATC) and preferred term.

If there are parts of the start date or stop date of the medication, to determine whether the medication is prior or concomitant, rules described in Section 3.10 will be used.

The concomitant medications will be summarized by ATC classification and PT. For each medication term, the numbers and percentages of patients experiencing a medication with that term. If a patient reports the occurrence of a medication more than once, the medication is only counted once. These will be summarized for the Safety Population.

The use of prior and concomitant medications will be included in a by-patient data listing.

Concomitant procedures experienced while on study will not be summarized; they will be listed.

Systemic steroid use is gathered only for glioma patients as it is part of what is considered for RANO response assessment. This data will not be summarized; it will be listed.

#### Relevant Output

| Table 14.3.11a Table 14.3.11b Table 14.3.11c Table 14.3.11d Table 14.3.11e | Concomitant Medications (Cohort 1, Safety Population)<br>Concomitant Medications (Cohort 2, Safety Population)<br>Concomitant Medications (Cohort 3, Safety Population)<br>Concomitant Medications (Cohort 4, Safety Population)<br>Concomitant Medications (Cohort 5, Safety Population) |
|---|---|
| Listing 16.2.9.4<br>Listing 16.2.9.5<br>Listing 16.2.9.6 | Prior and Concomitant Medications Concomitant Procedures Systemic Steroid Dosing |

#### 4.5.7. Performance Status

The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). All ECOG performance status data will be listed.

Listing 16.2.9.7 ECOG Performance Status

## 5. EXPLORATORY ANALYSES

Quantification of ctDNA over time will be analyzed in an exploratory fashion. Phamacogenomics will also be analyzed in an exploratory manner. The results of these analyses may be presented in a separate report.

### 6. CHANGES TO PLANNED ANALYSES

All changes from procedures outlined in the protocol and procedures outlined in this SAP will be summarized in the study report. Decisions to deviate from planned analyses will be documented at the time they are made.

If any modifications in the experimental design, dosages, parameters, patient selection, or any other sections of the protocol are indicated or required, the Investigator will consult with the Sponsor before such changes are instituted. Modifications will be accomplished through formal amendments to this protocol by the Sponsor and approval from the appropriate Institutional Review Board (IRB) or Independent Ethics Committee (IEC).

#### 7. REFERENCES

Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA. (2014) Recommendations for initial evaluation, staging, and response assessment of Hodgkin and Non-Hodgkin lymphoma: the Lugano classification. J Clin Onc. 32(27): 3059-3067.

Eisenhauer EA, Therasse P, Bogaerts J, et al. (2009) New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 45(2):228-47.

Food and Drug Administration. (2009). Guidance for Industry Drug Induced Liver Injury: Premarketing Clinical Evaluation.

Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X (2011). Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. Dec; 20(10):1727-1736

International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use. (1995). ICH harmonized tripartite guideline structure and content of clinical study reports E3.

Oken M, Creech R, Tormey D, et al. (1982). Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 5: 649-655.

van den Bent MJ, Wefel JS, Schiff D, et al. (2011) Response assessment in neuro-oncology (a report of the RANO group): assessment of outcome in trials of diffuse low-grade gliomas. Lancet Oncol. 12(6): 583-93.

Wen PY, Macdonald DR, Reardon DA, et al. (2010) Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 28(11): 1963-72.

## 8. CLINICAL STUDY REPORT APPENDICES

## 8.1. Statistical Tables and Figures to be Generated

Disposition/Demographics/Baseline (CSR Table Section 14.1)

| Table 14.1.1a | Patient Enrollment and Disposition (Cohort 1) |
|---|---|
| Table 14.1.1b | Patient Enrollment and Disposition (Cohort 2) |
| Table 14.1.1c | Patient Enrollment and Disposition (Cohort 3) |
| Table 14.1.1d | Patient Enrollment and Disposition (Cohort 4) |
| Table 14.1.1e | Patient Enrollment and Disposition (Cohort 5) |
| | 1 , , |
| Table 14.1.2.1a | Demographics and Baseline Characteristics (Cohort 1, Response Evaluable Population) |
| Table 14.1.2.1b | Demographics and Baseline Characteristics (Cohort 2, Response Evaluable Population) |
| Table 14.1.2.1c | Demographics and Baseline Characteristics (Cohort 3, Response Evaluable Population) |
| Table 14.1.2.1d | Demographics and Baseline Characteristics (Cohort 4, Response Evaluable Population) |
| Table 14.1.2.1e | Demographics and Baseline Characteristics (Cohort 5, Response Evaluable Population) |
| Table 14.1.2.2a | Demographics and Baseline Characteristics (Cohort 1, Safety Population) |
| Table 14.1.2.2b | Demographics and Baseline Characteristics (Cohort 2, Safety Population) |
| Table 14.1.2.2c | Demographics and Baseline Characteristics (Cohort 3, Safety Population) |
| Table 14.1.2.2d | Demographics and Baseline Characteristics (Cohort 4, Safety Population) |
| Table 14.1.2.2e | Demographics and Baseline Characteristics (Cohort 5, Safety Population) |
| Table 14.1.3.1 | Baseline Disease Characteristics (Cohort 1, Response Evaluable Population) |
| Table 14.1.3.1b | Baseline Disease Characteristics (Cohort 2, Response Evaluable Population) |
| Table 14.1.3.1c | Baseline Disease Characteristics (Cohort 3, Response Evaluable Population) |
| Table 14.1.3.1d | Baseline Disease Characteristics (Cohort 4, Response Evaluable Population) |
| Table 14.1.3.1e | Baseline Disease Characteristics (Cohort 5, Response Evaluable Population) |

| Table 14.1.3.2a Table 14.1.3.2b Table 14.1.3.2c Table 14.1.3.2d Table 14.1.3.2e | Baseline Disease Characteristics (Cohort 1, Safety Population) Baseline Disease Characteristics (Cohort 2, Safety Population) Baseline Disease Characteristics (Cohort 3, Safety Population) Baseline Disease Characteristics (Cohort 4, Safety Population) Baseline Disease Characteristics (Cohort 5, Safety Population) |
|---|---|
| Table 14.1.4.1a | IDH1 and Other Mutations (Cohort 1, Response Evaluable Population) |
| Table 14.1.4.1b | IDH1 and Other Mutations (Cohort 2, Response Evaluable Population) |
| Table 14.1.4.1c | IDH1 and Other Mutations (Cohort 3, Response Evaluable Population) |
| Table 14.1.4.1d | IDH1 and Other Mutations (Cohort 4, Response Evaluable Population) |
| Table 14.1.4.1e | IDH1 and Other Mutations (Cohort 5, Response Evaluable Population) |
| Table 14.1.4.2a | IDH1 and Other Mutations (Cohort 1, Safety Population) |
| Table 14.1.4.2b | IDH1 and Other Mutations (Cohort 2, Safety Population) |
| Table 14.1.4.2c | IDH1 and Other Mutations (Cohort 3, Safety Population) |
| Table 14.1.4.2d | IDH1 and Other Mutations (Cohort 4, Safety Population) |
| Table 14.1.4.2e | IDH1 and Other Mutations (Cohort 5, Safety Population) |
| Table 14.1.5.1a | Prior Therapies (Cohort 1, Response Evaluable Population) |
| Table 14.1.5.1b | Prior Therapies (Cohort 2, Response Evaluable Population) |
| Table 14.1.5.1c | Prior Therapies (Cohort 3, Response Evaluable Population) |
| Table 14.1.5.1d | Prior Therapies (Cohort 4, Response Evaluable Population) |
| Table 14.1.5.1e | Prior Therapies (Cohort 5, Response Evaluable Population) |
| Table 14.1.5.2a | Prior Therapies (Cohort 1, Safety Population) |
| Table 14.1.5.2b | Prior Therapies (Cohort 2, Safety Population) |
| Table 14.1.5.2c | Prior Therapies (Cohort 3, Safety Population) |
| Table 14.1.5.2d | Prior Therapies (Cohort 4, Safety Population) |
| Table 14.1.5.2e | Prior Therapies (Cohort 5, Safety Population) |
| Table 14.1.6a | Medical History (Cohort 1, Safety Population) |
| Table 14.1.6b | Medical History (Cohort 2, Safety Population) |
| Table 14.1.6c | Medical History (Cohort 3, Safety Population) |
| Table 14.1.6d | Medical History (Cohort 4, Safety Population) |
| Table 14.1.6e | Medical History (Cohort 5, Safety Population) |

#### Efficacy/Pharmacokinetic Results (CSR Table Section 14.2) Table 14.2.1a Disease Response Assessment Overall and by Subgroup (Cohort 1, Response Evaluable Population) Table 14.2.1b Disease Response Assessment Overall and by Subgroup (Cohort 2, Response Evaluable Population) Table 14.2.1c Disease Response Assessment Overall and by Subgroup (Cohort 3, Response Evaluable Population) Table 14.2.1d Disease Response Assessment Overall and by Subgroup (Cohort 4, Response Evaluable Population) Table 14.2.1e Disease Response Assessment Overall and by Subgroup (Cohort 5, Response Evaluable Population) Maximum Decrease from Baseline in Tumor Burden (Cohort 1 Figure 14.2.2.1a Single Agent, Response Evaluable Population) Maximum Decrease from Baseline in Tumor Burden (Cohort 1 Figure 14.2.2.2a Combination Therapy, Response Evaluable Population) Figure 14.2.2.1b Maximum Decrease from Baseline in Tumor Burden (Cohort 2 Single Agent, Response Evaluable Population) Maximum Decrease from Baseline in Tumor Burden (Cohort 2 Figure 14.2.2.2b Combination Therapy, Response Evaluable Population) Figure 14.2.2.1c Maximum Decrease from Baseline in Tumor Burden (Cohort 3 Single Agent, Response Evaluable Population) Figure 14.2.2.2c Maximum Decrease from Baseline in Tumor Burden (Cohort 3 Combination Therapy, Response Evaluable Population) Figure 14.2.2.1d Maximum Decrease from Baseline in Tumor Burden (Cohort 4 Single Agent, Response Evaluable Population) Maximum Decrease from Baseline in Tumor Burden (Cohort 4 Figure 14.2.2.2d Combination Therapy, Response Evaluable Population) Figure 14.2.2.1e Maximum Decrease from Baseline in Tumor Burden (Cohort 5, Response Evaluable Population) Time on Treatment (Cohort 1 Single Agent, Safety Population) Figure 14.2.3.1a Time on Treatment (Cohort 1 Combination Therapy, Safety Figure 14.2.3.2a Population) Time on Treatment (Cohort 2 Single Agent, Safety Population) Figure 14.2.3.1b Figure 14.2.3.2b Time on Treatment (Cohort 2 Combination Therapy, Safety Population) Time on Treatment (Cohort 3 Single Agent, Safety Population) Figure 14.2.3.1c Figure 14.2.3.2c Time on Treatment (Cohort 3 Combination Therapy, Safety Population)

Figure 14.2.3.1d

Time on Treatment (Cohort 4 Single Agent, Safety Population)

| Figure 14.2.3.2d | Time on Treatment (Cohort 4 Combination Therapy, Safety Population) |
|---|---|
| Figure 14.2.3.1e | Time on Treatment (Cohort 5, Safety Population) |
| Table 14.2.4a | Progression-Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 1, Response Evaluable Population) |
| Table 14.2.4b | Progression-Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 2, Response Evaluable Population) |
| Table 14.2.4c | Progression-Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 3, Response Evaluable Population) |
| Table 14.2.4d | Progression-Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 4, Response Evaluable Population) |
| Table 14.2.4e | Progression-Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 5, Response Evaluable Population) |
| Table 14.2.5.1<br>Table14.2.5.2 | Overall Survival (Response Evaluable Population)<br>Overall Survival (Safety Population) |
| Figure 14.2.5.3a | Kaplan-Meier Plot of Overall Survival (Cohort 1, Response Evaluable Population) |
| Figure 14.2.5.3b | Kaplan-Meier Plot of Overall Survival (Cohort 2, Response Evaluable Population) |
| Figure 14.2.5.3c | Kaplan-Meier Plot of Overall Survival (Cohort 3, Response Evaluable Population) |
| Figure 14.2.5.3d | Kaplan-Meier Plot of Overall Survival (Cohort 4, Response Evaluable Population) |
| Figure 14.2.5.3e | Kaplan-Meier Plot of Overall Survival (Cohort 5, Response Evaluable Population) |
| Figure 14.2.5.4a | Kaplan-Meier Plot of Overall Survival (Cohort 1, Safety Population) |
| Figure 14.2.5.4b | Kaplan-Meier Plot of Overall Survival (Cohort 2, Safety Population) |
| Figure 14.2.5.4c | Kaplan-Meier Plot of Overall Survival (Cohort 3, Safety Population) |

| Figure 14.2.5.4d | Kaplan-Meier Plot of Overall Survival (Cohort 4, Safety Population) |
|---|---|
| Figure 14.2.5.4e | Kaplan-Meier Plot of Overall Survival (Cohort 5, Safety Population) |
| Figure 14.2.5.5a | Kaplan-Meier Plot of Progression Free Survival (Cohort 1, Response Evaluable Population) |
| Figure 14.2.5.5b | Kaplan-Meier Plot of Progression Free Survival (Cohort 2, Response Evaluable Population) |
| Figure 14.2.5.5c | Kaplan-Meier Plot of Progression Free Survival (Cohort 3, Response Evaluable Population) |
| Figure 14.2.5.5d | Kaplan-Meier Plot of Progression Free Survival (Cohort 4, Response Evaluable Population) |
| Figure 14.2.5.5e | Kaplan-Meier Plot of Progression Free Survival (Cohort 5,<br>Response Evaluable Population) |
| Figure 14.2.5.6a | Kaplan-Meier Plot of Progression Free Survival (Cohort 1, Safety Population) |
| Figure 14.2.5.6b | Kaplan-Meier Plot of Progression Free Survival (Cohort 2, Safety Population) |
| Figure 14.2.5.6c | Kaplan-Meier Plot of Progression Free Survival (Cohort 3, Safety Population) |
| Figure 14.2.5.6d | Kaplan-Meier Plot of Progression Free Survival (Cohort 4, Safety Population) |
| Figure 14.2.5.6e | Kaplan-Meier Plot of Progression Free Survival (Cohort 5, Safety Population) |
| Table 14.2.6a | Serum AFP, CA19-9, CEA (Cohort 2, Response Evaluable Population) |
| Table 14.2.6b | Serum AFP, CA19-9, CEA (Cohort 4, Response Evaluable Population) |
| Figure 14.2.7a | Serum AFP, CA19-9, CEA (Cohort 2, Response Evaluable Population) |
| Figure 14.2.7b | Serum AFP, CA19-9, CEA (Cohort 4, Response Evaluable Population) |
| Table 14.2.8a<br>Table 14.2.8b | EQ-5D-5L Summary (Cohort 1, Response Evaluable Population)<br>EQ-5D-5L Summary (Cohort 2, Response Evaluable Population) |
| Table 14.2.8c | EQ-5D-5L Summary (Cohort 2, Response Evaluable Population) EQ-5D-5L Summary (Cohort 3, Response Evaluable Population) |

| Table 14.2.8d<br>Table 14.2.8e | EQ-5D-5L Summary (Cohort 4, Response Evaluable Population)<br>EQ-5D-5L Summary (Cohort 5, Response Evaluable Population) |
|---|---|
| Figure 14.2.9a | EQ-5D-5L Quality of Life Assessment (Cohort 1, Response Evaluable Population) |
| Figure 14.2.9b | EQ-5D-5L Quality of Life Assessment (Cohort 2, Response Evaluable Population) |
| Figure 14.2.9c | EQ-5D-5L Quality of Life Assessment (Cohort 3, Response Evaluable Population) |
| Figure 14.2.9d | EQ-5D-5L Quality of Life Assessment (Cohort 4, Response Evaluable Population) |
| Figure 14.2.9e | EQ-5D-5L Quality of Life Assessment (Cohort 5, Response Evaluable Population) |
| Table 14.2.10.1a | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 1, PD Population) |
| Table 14.2.10.1b | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 2, PD Population) |
| Table 14.2.10.1c | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 3, PD Population) |
| Table 14.2.10.1d | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 4, PD Population) |
| Table 14.2.10.1e | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 5, PD Population) |
| Table 14.2.10.2a | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 1, PD Population) |
| Table 14.2.10.2b | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 2, PD Population) |
| Table 14.2.10.2c | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 3, PD Population) |
| Table 14.2.10.2d | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 4, PD Population) |
| Table 14.2.10.2e | Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 5, PD Population) |
| Figure 14.2.11.1a<br>Figure 14.2.11.1b<br>Figure 14.2.11.1c | Boxplot of Plasma 2-HG by Time Point (Cohort 1, PD Population)<br>Boxplot of Plasma 2-HG by Time Point (Cohort 2, PD Population)<br>Boxplot of Plasma 2-HG by Time Point (Cohort 3, PD Population) |

| Figure 14.2.11.1d<br>Figure 14.2.11.1e | Boxplot of Plasma 2-HG by Time Point (Cohort 4, PD Population)<br>Boxplot of Plasma 2-HG by Time Point (Cohort 5, PD Population) |
|---|---|
| Figure 14.2.11.2a<br>Figure 14.2.11.2b<br>Figure 14.2.11.2c<br>Figure 14.2.11.2d<br>Figure 14.2.11.2e | Boxplot of Urine 2-HG by Time Point (Cohort 1, PD Population) Boxplot of Urine 2-HG by Time Point (Cohort 2, PD Population) Boxplot of Urine 2-HG by Time Point (Cohort 3, PD Population) Boxplot of Urine 2-HG by Time Point (Cohort 4, PD Population) Boxplot of Urine 2-HG by Time Point (Cohort 5, PD Population) |
| Figure 14.2.11.3 | Boxplot of Tumor 2-HG Assessed by MRS by Time Point (Cohort 1, PD Population) |
| Figure 14.2.11.4 | Boxplot of CSF 2-HG by Time Point (Cohort 1, PD Population) |
| Table 14.2.13a | Summary of Pharmacokinetic Parameters (All Patients on Single Agent Therapy, PK Population) |
| Table 14.2.13b | Summary of Pharmacokinetic Parameters (Cohort 1, PK Population) |
| Table 14.2.13c | Summary of Pharmacokinetic Parameters (Cohort 2, PK Population) |
| Table 14.2.13d | Summary of Pharmacokinetic Parameters (Cohort 3, PK Population) |
| Table 14.2.13e | Summary of Pharmacokinetic Parameters (Cohort 4, PK Population) |
| Table 14.2.13f | Summary of Pharmacokinetic Parameters (Cohort 5, PK Population) |
| Figure 14.2.14.1a | FT-2102 Plasma Concentration over Time (Cohort 1, PK Population) |
| Figure 14.2.14.1b | FT-2102 Plasma Concentration over Time (Cohort 2, PK Population) |
| Figure 14.2.14.1c | FT-2102 Plasma Concentration over Time (Cohort 3, PK Population) |
| Figure 14.2.14.1d | FT-2102 Plasma Concentration over Time (Cohort 4, PK Population) |
| Figure 14.2.14.1e | FT-2102 Plasma Concentration over Time (Cohort 5, PK Population) |
| Figure 14.2.14.2a | FT-2102 Plasma Concentration over Log-Time (Cohort 1, PK Population) |
| Figure 14.2.14.2b | FT-2102 Plasma Concentration over Log-Time (Cohort 2, PK Population) |

| Figure 14.2.14.2c | FT-2102 Plasma Concentration over Log-Time (Cohort 3, PK Population) |
|---|---|
| Figure 14.2.14.2d | FT-2102 Plasma Concentration over Log-Time (Cohort 4, PK |
| F: 140140 | Population) |
| Figure 14.2.14.2e | FT-2102 Plasma Concentration over Log-Time (Cohort 5, PK Population) |
| Figure 14.2.15a | FT-2102 Geometric Mean Plasma Concentration over Nominal |
| | Time (All Patients on Single Agent Therapy, PK Population) |
| Figure 14.2.15b | FT-2102 Geometric Mean Plasma Concentration over Nominal |
| | Time (Cohort 1, PK Population) |
| Figure 14.2.15c | FT-2102 Geometric Mean Plasma Concentration over Nominal |
| | Time (Cohort 2, PK Population) |
| Figure 14.2.15d | FT-2102 Geometric Mean Plasma Concentration over Nominal |
| T: 44645 | Time (Cohort 3, PK Population) |
| Figure 14.2.15e | FT-2102 Geometric Mean Plasma Concentration over Nominal |
| E: 140.150 | Time (Cohort 4, PK Population) |
| Figure 14.2.15f | FT-2102 Geometric Mean Plasma Concentration over Nominal Time (Cohort 5, PK Population) |
| | Time (Conort 3, TR Topulation) |
| Table 14 2 16 1a | |
| Table 14.2.16.1a Table 14.2.16.1b | FT-2102 Exposure (Cohort 1, Response Evaluable Population) |
| Table 14.2.16.1b | FT-2102 Exposure (Cohort 1, Response Evaluable Population)<br>FT-2102 Exposure (Cohort 2, Response Evaluable Population) |
| Table 14.2.16.1b<br>Table 14.2.16.1c | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) |
| Table 14.2.16.1b<br>Table 14.2.16.1c<br>Table 14.2.16.1d | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) |
| Table 14.2.16.1b<br>Table 14.2.16.1c | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) |
| Table 14.2.16.1b<br>Table 14.2.16.1c<br>Table 14.2.16.1d<br>Table 14.2.16.1e | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) |
| Table 14.2.16.1b Table 14.2.16.1c Table 14.2.16.1d Table 14.2.16.1e Table 14.2.16.2a | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) FT-2102 Exposure (Cohort 1, Safety Population) |
| Table 14.2.16.1b Table 14.2.16.1c Table 14.2.16.1d Table 14.2.16.1e Table 14.2.16.2a Table 14.2.16.2b | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) FT-2102 Exposure (Cohort 1, Safety Population) FT-2102 Exposure (Cohort 2, Safety Population) |
| Table 14.2.16.1b Table 14.2.16.1c Table 14.2.16.1d Table 14.2.16.1e Table 14.2.16.2a Table 14.2.16.2b Table 14.2.16.2c | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) FT-2102 Exposure (Cohort 1, Safety Population) FT-2102 Exposure (Cohort 2, Safety Population) FT-2102 Exposure (Cohort 3, Safety Population) |
| Table 14.2.16.1b Table 14.2.16.1c Table 14.2.16.1d Table 14.2.16.1e Table 14.2.16.2a Table 14.2.16.2b Table 14.2.16.2c Table 14.2.16.2c Table 14.2.16.2d Table 14.2.16.2d | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) FT-2102 Exposure (Cohort 1, Safety Population) FT-2102 Exposure (Cohort 2, Safety Population) FT-2102 Exposure (Cohort 3, Safety Population) FT-2102 Exposure (Cohort 4, Safety Population) FT-2102 Exposure (Cohort 5, Safety Population) |
| Table 14.2.16.1b Table 14.2.16.1c Table 14.2.16.1d Table 14.2.16.1e Table 14.2.16.2a Table 14.2.16.2b Table 14.2.16.2c Table 14.2.16.2d Table 14.2.16.2d Table 14.2.16.2e | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) FT-2102 Exposure (Cohort 1, Safety Population) FT-2102 Exposure (Cohort 2, Safety Population) FT-2102 Exposure (Cohort 3, Safety Population) FT-2102 Exposure (Cohort 4, Safety Population) FT-2102 Exposure (Cohort 5, Safety Population) Summary of Azacitidine Exposure (Cohort 1, Safety Population) |
| Table 14.2.16.1b Table 14.2.16.1c Table 14.2.16.1d Table 14.2.16.1e Table 14.2.16.2a Table 14.2.16.2b Table 14.2.16.2c Table 14.2.16.2d Table 14.2.16.2d Table 14.2.17a Table 14.2.17a | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) FT-2102 Exposure (Cohort 1, Safety Population) FT-2102 Exposure (Cohort 2, Safety Population) FT-2102 Exposure (Cohort 3, Safety Population) FT-2102 Exposure (Cohort 4, Safety Population) FT-2102 Exposure (Cohort 5, Safety Population) Summary of Azacitidine Exposure (Cohort 1, Safety Population) Summary of Nivolumab Exposure (Cohort 2, Safety Population) |
| Table 14.2.16.1b Table 14.2.16.1c Table 14.2.16.1d Table 14.2.16.1e Table 14.2.16.2a Table 14.2.16.2b Table 14.2.16.2c Table 14.2.16.2d Table 14.2.16.2d Table 14.2.16.2e | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) FT-2102 Exposure (Cohort 1, Safety Population) FT-2102 Exposure (Cohort 2, Safety Population) FT-2102 Exposure (Cohort 3, Safety Population) FT-2102 Exposure (Cohort 4, Safety Population) FT-2102 Exposure (Cohort 5, Safety Population) Summary of Azacitidine Exposure (Cohort 1, Safety Population) Summary of Nivolumab Exposure (Cohort 2, Safety Population) Summary of Gemcitabine and Cisplatin Exposure (Cohort 3, |
| Table 14.2.16.1b Table 14.2.16.1c Table 14.2.16.1d Table 14.2.16.1e Table 14.2.16.2a Table 14.2.16.2b Table 14.2.16.2c Table 14.2.16.2d Table 14.2.16.2d Table 14.2.17a Table 14.2.17a | FT-2102 Exposure (Cohort 1, Response Evaluable Population) FT-2102 Exposure (Cohort 2, Response Evaluable Population) FT-2102 Exposure (Cohort 3, Response Evaluable Population) FT-2102 Exposure (Cohort 4, Response Evaluable Population) FT-2102 Exposure (Cohort 5, Response Evaluable Population) FT-2102 Exposure (Cohort 1, Safety Population) FT-2102 Exposure (Cohort 2, Safety Population) FT-2102 Exposure (Cohort 3, Safety Population) FT-2102 Exposure (Cohort 4, Safety Population) FT-2102 Exposure (Cohort 5, Safety Population) Summary of Azacitidine Exposure (Cohort 1, Safety Population) Summary of Nivolumab Exposure (Cohort 2, Safety Population) |

# Displays of Adverse Events (CSR Section 14.3.1)

| Table 14.3.1.1a | Summary of Treatment-Emergent Adverse Events, Overall and by Dose Group (Cohort 1, Safety Population) |
|---|---|
| Table 14.3.1.1b | Summary of Treatment-Emergent Adverse Events, Overall and by Dose Group (Cohort 2, Safety Population) |
| Table 14.3.1.1c | Summary of Treatment-Emergent Adverse Events, Overall and by Dose Group (Cohort 3, Safety Population) |
| Table 14.3.1.1d | Summary of Treatment-Emergent Adverse Events, Overall and by Dose Group (Cohort 4, Safety Population) |
| Table 14.3.1.1e | Summary of Treatment-Emergent Adverse Events, Overall and by Dose Group (Cohort 5, Safety Population) |
| Table 14.3.1.a | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (All Patients Receiving Single Agent<br>Therapy, Safety Population) |
| Table 14.3.1.b | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (All Patients Receiving Combination<br>Therapy, Safety Population) |
| Table 14.3.1.c | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (All Patients, Safety Population) |
| Table 14.3.1.d | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 1, Safety Population) |
| Table 14.3.1.e | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 2, Safety Population) |
| Table 14.3.1.2f | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 3, Safety Population) |
| Table 14.3.1.g | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 4, Safety Population) |
| Table 14.3.1.h | Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term (Cohort 5, Safety Population) |
| Table 14.3.1.3a | Treatment-Emergent Adverse Events Related to FT-2102 by<br>MedDRA System Organ Class and Preferred Term (Cohort 1,<br>Safety Population) |
| Table 14.3.1.3b | Treatment-Emergent Adverse Events Related to FT-2102 by<br>MedDRA System Organ Class and Preferred Term (Cohort 2,<br>Safety Population) |
| Table 14.3.1.3c | Treatment-Emergent Adverse Events Related to FT-2102 by<br>MedDRA System Organ Class and Preferred Term (Cohort 3,<br>Safety Population) |

| Table 14.3.1.3d | Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 4, |
|---|---|
| Table 14.3.1.3e | Safety Population) Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 5, Safety Population) |
| Table 14.3.1.4a | Severe Treatment-Emergent Adverse Events by MedDRA System<br>Organ Class and Preferred Term (Cohort 1, Safety Population) |
| Table 14.3.1.4b | Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Cohort 2, Safety Population) |
| Table 14.3.1.4c | Severe Treatment-Emergent Adverse Events by MedDRA System<br>Organ Class and Preferred Term (Cohort 3, Safety Population) |
| Table 14.3.1.4d | Severe Treatment-Emergent Adverse Events by MedDRA System<br>Organ Class and Preferred Term (Cohort 4, Safety Population) |
| Table 14.3.1.4e | Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Cohort 5, Safety Population) |
| Table 14.3.1.5a | TEAEs by MedDRA Preferred Term (Cohort 1, Safety Population) |
| Table 14.3.1.5b | TEAEs by MedDRA Preferred Term (Cohort 2, Safety Population) |
| Table 14.3.1.5c | TEAEs by MedDRA Preferred Term (Cohort 3, Safety Population) |
| Table 14.3.1.5d | TEAEs by MedDRA Preferred Term (Cohort 4, Safety Population) |
| Table 14.3.1.5e | TEAEs by MedDRA Preferred Term (Cohort 5, Safety Population) |
| Listings of Deaths, Se | erious Adverse Events, and Other Significant Events (CSR Section 14.3.2) |
| Table 14.3.2.1 | Listing of Deaths |
| Table 14.3.2.2 | Listing of Serious Adverse Events |
| Table 14.3.2.3 | Listing of Discontinuations Due to Adverse Events |
| Table 14.3.2.4 | Listing of Dose-Limiting Toxicities |
| Abnormal Laboratory Value Listings (CSR Section 14.3.4) | |
| Table 14.3.4.1 | Listing of Abnormal Laboratory Values |
| Table 14.3.4.2 | Listing of Laboratory Values with CTCAE Severity ≥Grade 3 |
| Table 14.3.4.3 | Listing of Liver Function Tests of Potential Concern |
| Other Safety Tabulations (CSR Section 14.3.5) | |
| Table 14.3.5.1a | Summary and Change from Baseline for Hematology and<br>Coagulation Parameters by Time Point, Overall and by Dose<br>Group (Cohort 1, Safety Population) |

| Table 14.3.5.1b | Summary and Change from Baseline for Hematology and<br>Coagulation Parameters by Time Point, Overall and by Dose<br>Group (Cohort 2, Safety Population) |
|---|---|
| Table 14.3.5.1c | Summary and Change from Baseline for Hematology and Coagulation Parameters by Time Point, Overall and by Dose Group (Cohort 3, Safety Population) |
| Table 14.3.5.1d | Summary and Change from Baseline for Hematology and Coagulation Parameters by Time Point, Overall and by Dose Group (Cohort 4, Safety Population) |
| Table 14.3.5.1e | Summary and Change from Baseline for Hematology and Coagulation Parameters by Time Point, Overall and by Dose Group (Cohort 5, Safety Population) |
| Table 14.3.5.2a | Summary and Change from Baseline for Chemistry Parameters by Time Point, Overall and by Dose Group (Cohort 1, Safety Population) |
| Table 14.3.5.2b | Summary and Change from Baseline for Chemistry Parameters by Time Point, Overall and by Dose Group (Cohort 2, Safety Population) |
| Table 14.3.5.2c | Summary and Change from Baseline for Chemistry Parameters by Time Point, Overall and by Dose Group (Cohort 3, Safety Population) |
| Table 14.3.5.2d | Summary and Change from Baseline for Chemistry Parameters by Time Point, Overall and by Dose Group (Cohort 4, Safety Population) |
| Table 14.3.5.2e | Summary and Change from Baseline for Chemistry Parameters by Time Point, Overall and by Dose Group (Cohort 5, Safety Population) |
| Table 14.3.6.1a | Shifts from Baseline to Worst Value on Study in Hematology,<br>Overall and by Dose Group (Cohort 1, Safety Population) |
| Table 14.3.6.1b | Shifts from Baseline to Worst Value on Study in Hematology,<br>Overall and by Dose Group (Cohort 2, Safety Population) |
| Table 14.3.6.1c | Shifts from Baseline to Worst Value on Study in Hematology,<br>Overall and by Dose Group (Cohort 3, Safety Population) |
| Table 14.3.6.1d | Shifts from Baseline to Worst Value on Study in Hematology,<br>Overall and by Dose Group (Cohort 4, Safety Population) |
| Table 14.3.6.1e | Shifts from Baseline to Worst Value on Study in Hematology,<br>Overall and by Dose Group (Cohort 5, Safety Population) |
| Table 14.3.6.2a | Shifts from Baseline to Worst Value on Study in Chemistry,<br>Overall and by Dose Group (Cohort 1, Safety Population) |

| Table 14.3.6.2b Table 14.3.6.2c | Shifts from Baseline to Worst Value on Study in Chemistry,<br>Overall and by Dose Group (Cohort 2, Safety Population)<br>Shifts from Baseline to Worst Value on Study in Chemistry, |
|---|---|
| Table 14.3.6.2d | Overall and by Dose Group (Cohort 3, Safety Population) Shifts from Baseline to Worst Value on Study in Chemistry, |
| Table 14.3.6.2e | Overall and by Dose Group (Cohort 4, Safety Population) Shifts from Baseline to Worst Value on Study in Chemistry, Overall and by Dose Group (Cohort 5, Safety Population) |
| Table 14.3.7a | Summary of Liver Function Test Results (All Patients Receiving Single Agent Therapy, Safety Population) |
| Table 14.3.7b | Summary of Liver Function Test Results (Cohort 1, Safety Population) |
| Table 14.3.7c | Summary of Liver Function Test Results (Cohort 2, Safety Population) |
| Table 14.3.7d | Summary of Liver Function Test Results (Cohort 3, Safety Population) |
| Table 14.3.7e | Summary of Liver Function Test Results (Cohort 4, Safety Population) |
| Table 14.3.7f | Summary of Liver Function Test Results (Cohort 5, Safety Population) |
| Table 14.3.8a | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 1, Safety Population) |
| Table 14.3.8b | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 2, Safety Population) |
| Table 14.3.8c | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 3, Safety Population) |
| Table 14.3.8d | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 4, Safety Population) |
| Table 14.3.8e | Summary and Change from Baseline for Vital Signs by Time Point, Overall and by Dose Group (Cohort 5, Safety Population) |
| Table 14.3.9a | Electrocardiogram Results (Cohort 1, Safety Population) |
| Table 14.3.9b | Electrocardiogram Results (Cohort 2, Safety Population) |
| Table 14.3.9c | Electrocardiogram Results (Cohort 3, Safety Population) |
| Table 14.3.9d | Electrocardiogram Results (Cohort 4, Safety Population) |
| Table 14.3.9e | Electrocardiogram Results (Cohort 5, Safety Population) |

| Table 14.3.11a | Concomitant Medications (Cohort 1, Safety Population) |
|---|---|
| Table 14.3.11b | Concomitant Medications (Cohort 2, Safety Population) |
| Table 14.3.11c | Concomitant Medications (Cohort 3, Safety Population) |
| Table 14.3.11d | Concomitant Medications (Cohort 4, Safety Population) |
| Table 14.3.11e | Concomitant Medications (Cohort 5, Safety Population) |
| 8.2. Data Li | stings to be Generated |
| Discontinued Patient | s (CSR Appendix 16.2.1) |
| Listing 16.2.1.1 | Study Completion Status |
| Listing 16.2.1.2 | Pre-Screening Consent |
| Listing 16.2.1.3 | Enrollment Protocol Deviations (CSR Appendix 16.2.2) |
| Listing 16.2.2.1 | Inclusion and Exclusion Criteria |
| Listing 16.2.2.2 | Protocol Violations |
| Patients Excluded fro | om the Efficacy Analysis (CSR Appendix 16.2.3) |
| Listing 16.2.3.1 | Analysis Sets |
| Demographic and Ba | seline Characteristics (CSR Appendix 16.2.4) |
| Listing 16.2.4.1 | Demographics and Baseline Characteristics |
| Listing 16.2.4.2 | Baseline Disease Data and Cancer Diagnosis |
| Listing 16.2.4.3 | IDH1 Mutation and Other Mutations |
| Listing 16.2.4.4 | Medical History |
| Listing 16.2.4.5 | Prior Anti-Cancer Therapies |
| Listing 16.2.4.6 | Prior Radiotherapy |
| Listing 16.2.4.7 | Major Surgical Tumor Resections |
| Listing 16.2.4.8 | Child-Pugh Score |
| Listing 16.2.4.9 | Hepatitis B and C |
| Listing 16.2.4.10 | Archival Tumor Tissue |
| Compliance and/or I | Orug Concentration Data (CSR Appendix 16.2.5) |
| Listing 16.2.5.1 | FT-2102 Administration |
| Listing 16.2.5.2 | Drug Accountability |
| Listing 16.2.5.3 | Azacitidine, Nivolumab, Cisplatin, and Gemcitibine |
| | Administration |
| Listing 16.2.5.4 | Pharmacokinetic Concentrations |
| Listing 16.2.5.5 | Pharmacokinetic Parameters |
| Individual Efficacy R | esponse Data (CSR Appendix 16.2.6) |
| Listing 16.2.6.1 | Target Lesions (RECIST) |
| Listing 16.2.6.2 | Non-Target and New Lesions (RECIST) |
| Listing 16.2.6.3 | Measurable Lesions (RANO) |

| Listing 16.2.6.4<br>Listing 16.2.6.5<br>Listing 16.2.6.6<br>Listing 16.2.6.7 | Non-Measurable and New Lesions (RANO) Response Assessment (RECIST) Response Assessment (RANO and LGG RANO) Response Assessment (Cheson) |
|---|---|
| Listing 16.2.6.8<br>Listing 16.2.6.9<br>Listing 16.2.6.10 | Survival Status Serum AFP, CA19-9, CEA EQ5D-5L Quality of Life |
| Listing 16.2.6.11<br>Listing 16.2.6.12<br>Listing 16.2.6.13 | 2-HG MRS Assessments Archival Tumor Tissue and Tumor Biopsy Pharmacogenomics Samples |
| AssessmentAdverse E | Event Listings (CSR Appendix 16.2.7) |
| Listing 16.2.7.1<br>Listing 16.2.7.2 | Adverse Events by Patient and Verbatim Term<br>Adverse Events by Patient and MedDRA System Organ Class and<br>Preferred Term |
| Listing 16.2.7.3 | Adverse Events by MedDRA System Organ Class, Preferred Term, Cohort, and Patient |
| Listings of Individual | Laboratory Measurements by Patient (CSR Appendix 16.2.8) |
| Listing 16.2.8.1<br>Listing 16.2.8.2<br>Listing 16.2.8.3<br>Listing 16.2.8.4<br>Listing 16.2.8.5<br>Listing 16.2.8.6 | Laboratory Results: Hematology Laboratory Results: Chemistry Laboratory Results: Urinalysis Laboratory Results: Coagulation Laboratory Normal Ranges Laboratory Results: Other Screening Tests and Pregnancy |
| Other Safety Listings (CSR Appendix 16.2.9) | |
| Listing 16.2.9.1<br>Listing 16.2.9.2<br>Listing 16.2.9.3<br>Listing 16.2.9.4<br>Listing 16.2.9.5<br>Listing 16.2.9.6<br>Listing 16.2.9.7 | Vital Signs Physical Examinations Electrocardiogram Results Prior and Concomitant Medications Concomitant Procedures Systemic Steroid Dosing ECOG Performance Status |

## 9. TABLE AND FIGURE SHELLS


Table 14.1.1a

#### Patient Enrollment and Disposition (Cohort 1)

| Disposition | Statistic | Cohort 1A:<br>FT-2102<br>N (%) | Cohort 1B:<br>FT-2102 + AZA<br>N (%) | Cohort 1:<br>Overall<br>N (%) | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Total Number of Patients | | | | |
| | | | | | Screened | n | XX | XX | XX |
| Screen Failures <sup>1</sup> | n (%) | xx (xx) | xx (xx) | xx (xx) | | | | | |
| Enrolled <sup>1</sup> | n (%) | xx (xx) | xx (xx) | xx (xx) | | | | | |
| Dosed <sup>2</sup> | n (%) | xx (xx) | xx (xx) | xx (xx) | | | | | |
| Currently ongoing <sup>3</sup> | n (%) | xx (xx) | xx (xx) | xx (xx) | | | | | |
| Discontinued treatment <sup>3</sup> | | | | | | | | | |
| Discontinued study participation <sup>3</sup> | | | | | | | | | |
| Study Populations <sup>2</sup> | | | | | | | | | |
| Safety | n (%) | | | | | | | | |
| DLT Evaluable | n (%) | | | | | | | | |
| Response Evaluable | n (%) | | | | | | | | |
| PK Analysis Set | n (%) | | | | | | | | |
| PD Analysis Set | 11 (0) | | | | | | | | |
| Primary Reason for Discontinuation of Treatment <sup>3</sup> | n (%) | | | | | | | | |
| Adverse Event | n (%) | | | | | | | | |
| Death | n (%) | | | | | | | | |
| Withdrew Consent | n (%) | | | | | | | | |
| Lost to Follow-up | n (%) | | | | | | | | |
| Patient Noncompliance | n (%) | | | | | | | | |
| Discontinuation of Study by Sponsor | n (%) | | | | | | | | |
| Protocol Violation | n (%) | | | | | | | | |
| Physician Decision | n (%) | | | | | | | | |
| Protocol Defined Disease Progression | 11 (0) | | | | | | | | |

DATE: HH:MM/DDMMMYYYY

Primary Reason for Discontinuation of Study Participation<sup>3</sup> Death n (%) Permanent Withdrawal of Consent n (%) Lost to Follow-up n (%) Patient Noncompliance/ Protocol Violation(s) n (%) Discontinuation of Study by Sponsor n (%) Physician Decision n (%) Pregnancy n (%) Protocol Defined Disease Progression n (%) Other n (%)

Source: Data Listing 16.2.x

Programming Note:

Repeat table for Cohorts 2-5.

<sup>1</sup> Percentage based on the number screened.

<sup>&</sup>lt;sup>2</sup> Percentage based on the number enrolled.

<sup>&</sup>lt;sup>3</sup> Percentage based on the number dosed.

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

#### Table 14.1.2.1a

Demographics and Baseline Characteristics (Cohort 1, Response Evaluable Population)

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|---|---|---|---|---|
| Demographics | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| | | (N = ) | (N = ) | (N = ) |
| Age at consent (years) | n | | | |
| nge at consone (years) | mean | | | |
| | SD | | | |
| | median | | | |
| | min - max | | | |
| Age category (years) | | | | |
| 18-40 | n (%) | | | |
| 41-59 | n (%) | | | |
| >60 | n (%) | | | |
| Sex at birth | | | | |
| Male | n (%) | | | |
| Female | n (%) | | | |
| Of childbearing potential | n (%) | | | |
| Post-menopausal | n (%) | | | |
| Sterilized | n (응) | | | |
| Race | | | | |
| American Indian or Alaska Native | n (%) | | | |
| Asian | n (%) | | | |
| Black or African American | n (%) | | | |
| Native Hawaiian or Other Pacific Islander | n (%) | | | |
| White | n (%) | | | |
| Other<br>Not Reported | n (%) | | | |
| Ethnicity<br>Hispanic<br>Not Hispanic | | | | |
| Not reported | n (%) | | | |

| Height (cm) | | n<br>mean<br>SD<br>median<br>min - max |
|---|---|---|
| Weight (kg) | | n<br>mean<br>SD<br>median<br>min - max |
| BMI (kg/m^2) | | n<br>mean<br>SD<br>median<br>min - max |
| ECOG Score | 0<br>1<br>2<br>3<br>4 | n (%) n (%) n (%) n (%) n (%) |
| Hepatitis B Status<br>Negative<br>Positive | | n (%)<br>n (%) |
| Hepatitis C Status<br>Negative<br>Positive | | n (%)<br>n (%) |
| IDH1 Mutation Subtype R132C R132H R132S R132L R132G Other Unknown | | n (%) |

FORMA Therapeutics 2102-ONC-102 Statistical Analysis Plan 28 June 2019, Version 2.0

DATE: HH:MM/DDMMMYYYY

Programming Note: Repeat for Cohorts 2-5

Programming Note: Use this shell for 14.1.2.2 (Safety Population)

dential Page 1 of x

### Table 14.1.3.1a

# Baseline Disease Characteristics (Cohort 1, Response Evaluable Population)

| Parameter | Statistic | Cohort 1A: | Cohort 1B: | Cohort 1: |
|---|---|---|---|---|
| | Statistic | FT-2102<br>(N = ) | FT-2102 + AZA $(N = )$ | Overall (N = ) |
| | | (14 ) | (24 ) | (14 ) |
| Current glioma diagnosis | | | | |
| Diffuse astrocytoma, IDH mutant | n (%) | | | |
| Diffuse astrocytoma, NOS | n (%) | | | |
| Anaplastic astrocytoma, IDH mutant | n (%) | | | |
| Anaplastic astrocytoma, NOS | n (%) | | | |
| Glioblastoma, IDH mutant | n (%) | | | |
| Glioblastoma, NOS | n (%) | | | |
| Oligodendroglioma, IDH mutant | n (%) | | | |
| Oligodendroglioma, NOS | n (%) | | | |
| Anaplastic oligodendroglioma, IDH-mutant | n (%) | | | |
| Anaplastic oligodendroglioma, NOS | n (%) | | | |
| Oligoastrocytoma, NOS | n (%) | | | |
| Anaplastic oligoastrocytoma, NOS | n (%) | | | |
| Pilocytic astrocytoma | n (%) | | | |
| Pilomyxoid astrocytoma | n (%) | | | |
| Subependymal giant cell astrocytoma | n (%) | | | |
| Pleomorphic xanthoastrocytoma | n (%) | | | |
| Anaplastic pleomorphic xanthoastrocytoma | n (%) | | | |
| Other | n (%) | | | |
| Initial glioma diagnosis | | | | |
| Diffuse astrocytoma, IDH mutant | n (%) | | | |
| Diffuse astrocytoma, NOS | n (%) | | | |
| Anaplastic astrocytoma, IDH mutant | n (%) | | | |
| Anaplastic astrocytoma, NOS | n (%) | | | |
| Glioblastoma, IDH mutant | n (%) | | | |
| Glioblastoma, NOS | n (%) | | | |
| Oligodendroglioma, IDH mutant | n (%) | | | |
| Oligodendroglioma, NOS | n (%) | | | |
| Anaplastic oligodendroglioma, IDH-mutant | n (%) | | | |
| Anaplastic oligodendroglioma, NOS | n (%) | | | |

| Oligoastrocytoma, NOS | n (%) |
|---|---|
| Anaplastic oligoastrocytoma, NOS | n (%) |
| Pilocytic astrocytoma | n (%) |
| Pilomyxoid astrocytoma | n (%) |
| Subependymal giant cell astrocytoma | n (%) |
| Pleomorphic xanthoastrocytoma | n (%) |
| Anaplastic pleomorphic xanthoastrocytoma | n (%) |
| Other | n (%) |
| Years since initial diagnosis | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Grade at initial diagnosis | |
| I | n (%) |
| II | n (%) |
| III | n (%) |
| IV | n (%) |
| Months since recurrence | n |
| Months since recurrence | n<br>mean |
| Months since recurrence | |
| Months since recurrence | mean |
| Months since recurrence | mean<br>SD |
| Months since recurrence | mean<br>SD<br>median |
| Months since recurrence Current grade | mean<br>SD<br>median |
| | mean<br>SD<br>median |
| Current grade | mean<br>SD<br>median<br>min - max |
| Current grade | mean<br>SD<br>median<br>min - max<br>n (%) |
| Current grade I II III IV | mean SD median min - max n (%) n (%) |
| Current grade I II | mean SD median min - max n (%) n (%) n (%) |
| Current grade I II III IV | mean<br>SD<br>median<br>min - max<br>n (%)<br>n (%)<br>n (%)<br>n (%) |
| Current grade I II III IV | mean<br>SD<br>median<br>min - max<br>n (%)<br>n (%)<br>n (%)<br>n (%) |
| Current grade I II III IV Unknown/ NA | mean<br>SD<br>median<br>min - max<br>n (%)<br>n (%)<br>n (%)<br>n (%) |
| Current grade I II III IV Unknown/ NA Baseline steroids | mean SD median min - max n (%) n (%) n (%) n (%) n (%) |
| Current grade I II III IV Unknown/ NA Baseline steroids Yes | mean SD median min - max n (%) n (%) n (%) n (%) n (%) |
| Current grade I II III IV Unknown/ NA Baseline steroids Yes No Prior therapies | mean SD median min - max n (%) n (%) n (%) n (%) n (%) |
| Current grade I II III IV Unknown/ NA Baseline steroids Yes No | mean SD median min - max n (%) n (%) n (%) n (%) n (%) |
| Current grade I II III IV Unknown/ NA Baseline steroids Yes No Prior therapies | mean SD median min - max n (%) n (%) n (%) n (%) n (%) n (%) |

| Number of prior regimens | n |
|--------------------------|-----------|
| | mean |
| | SD |
| | median |
| | min - max |
| Prior regimen categories | |
| 1 | n (%) |
| 2 | n (%) |
| 3 | n (%) |
| >3 | n (%) |
| Prior IDH1 therapy | |
| Yes | n (%) |
| No | n (%) |
| Prior radiation | |
| Yes | n (%) |
| No | n (%) |
| Prior tezolomide | |
| Yes | n (%) |
| No | n (%) |

Programming note: repeat for 14.1.3.2a (Safety Population)


Table 14.1.3.1b

# Baseline Disease Characteristics (Cohort 2, Response Evaluable Population)

| | | Cohort 2A: | Cohort 2B: | Cohort 2: |
|---|---|---|---|---|
| Parameter | Statistic | FT-2102 | FT-2102 +<br>Nivolumab<br>(N = ) | Overall |
| | | (N = ) | | (N = ) |
| Hepatobiliary Cancer (HBC) Diagnosis | | | | |
| Hepatocellular carcinoma | n (%) | | | |
| Fibrolamellar | n (%) | | | |
| Clear Cell | n (%) | | | |
| Other | n (%) | | | |
| Gallbladder carcinoma | n (%) | | | |
| Intrahepatic cholangiocarcinoma | n (%) | | | |
| Extraheptic cholangiocarcinoma | n (%) | | | |
| Biliary tumor NOS | n (%) | | | |
| - | | | | |
| Current Stage | | | | |
| I | n (%) | | | |
| IA | n (%) | | | |
| IB | n (%) | | | |
| IIA | n (%) | | | |
| IIB | n (%) | | | |
| IIIA | n (%) | | | |
| IIIB | n (%) | | | |
| IVA | n (%) | | | |
| IVB | n (%) | | | |
| NA | n (%) | | | |
| Grade at Initial Diagnosis | | | | |
| Gx | n (%) | | | |
| G1 | n (%) | | | |
| G2 | n (%) | | | |
| G3 | n (%) | | | |
| G4 | n (%) | | | |
| Unknown | n (%) | | | |
| Not Applicable | n (%) | | | |

| Years since initial diagnosis | n<br>mean<br>SD<br>median<br>min - max |
|---|---|
| Months since recurrence | n<br>mean<br>SD<br>median<br>min - max |
| Fibrosis | |
| F0 | n (%) |
| F1 | n (%) |
| Current TNM Staging: Primary Tumor (T) | |
| Tx | n (%) |
| TO | n (%) |
| Tis | n (%) |
| T1 | n (%) |
| T2 | n (왕) |
| T3 | n (%) |
| T4 | n (%) |
| NA | n (%) |
| Current TNM Staging: Lymph Node (N) | |
| Nx | n (%) |
| NO | n (%) |
| N1 | n (%) |
| NA | n (%) |
| Current TNM Staging: Metastasis (M) | |
| M0 | n (%) |
| M1 | n (%) |
| NA | n (%) |
| | ( - / |
| Initial TNM Staging: Primary Tumor (T) | |
| Tx | n (%) |
| TO | n (%) |
| Tis | n (%) |

| T1 T2 T3 T4 NA Initial TNM Staging: Lymph Node (N) | n (%) n (%) n (%) n (%) n (%) |
|---|---|
| T3 T4 NA Initial TNM Staging: Lymph Node (N) | n (%)<br>n (%) |
| T4 NA Initial TNM Staging: Lymph Node (N) | n (%) |
| NA Initial TNM Staging: Lymph Node (N) | |
| Initial TNM Staging: Lymph Node (N) | n (%) |
| Nv | |
| | n (왕) |
| NO | n (왕) |
| N1 | n (왕) |
| NA | n (%) |
| Initial TNM Staging: Metastasis (M) | |
| MO | n (%) |
| M1 | n (%) |
| NA | n (%) |
| 1411 | 11 (0) |
| Number of prior regimens | n |
| . , | mean |
| | SD |
| | median |
| | min - max |
| Prior regimen categories | |
| 1 | n (%) |
| 2 | n (%) |
| 3 | n (왕) |
| >3 | n (왕) |
| D / TDW1 /1 | |
| Prior IDH1 therapy | - (0) |
| Yes<br>No | n (%) |
| NO | n (%) |
| Child-Pugh Score | n |
| 0 | mean |
| | SD |
| | median |
| | min - max |
| Child-Pugh Category | |
| A | n (%) |
| В | n (%) |

FORMA Therapeutics 2102-ONC-102 Statistical Analysis Plan 28 June 2019, Version 2.0

| С | n (%) | |
|---|---|---|
| Programming note: repeat for 14.1.3.2b | (Safety Population) | |
| PROGRAM NAME: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DATE: HH:MM/DDMMMYYYY |


### Table 14.1.3.1c

# Baseline Disease Characteristics (Cohort 3, Response Evaluable Population)

| | | Cohort 3A: | Cohort 3B: | Cohort 3: |
|---|---|---|---|---|
| Parameter | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| | | (N = ) | (N = ) | (N = ) |
| Chondrosarcoma diagnosis | | | | |
| Differentiated | n (%) | | | |
| Mesenchymal | n (%) | | | |
| Clear cell | n (%) | | | |
| Unknown | n (%) | | | |
| Other | n (%) | | | |
| Current Stage | | | | |
| Tx | n (%) | | | |
| TO | n (%) | | | |
| T1 | n (%) | | | |
| T1a | n (%) | | | |
| T1b | n (%) | | | |
| Т2 | n (%) | | | |
| T2b | n (%) | | | |
| Т3 | n (%) | | | |
| T3a | n (%) | | | |
| T3b | n (%) | | | |
| Т4 | n (%) | | | |
| Stage at initial diagnosis | | | | |
| Tx | n (%) | | | |
| TO | n (%) | | | |
| T1 | n (%) | | | |
| T1a | n (%) | | | |
| T1b | n (%) | | | |
| Т2 | n (%) | | | |
| T2b | n (%) | | | |
| Т3 | n (%) | | | |
| T3a | n (%) | | | |
| T3b | n (%) | | | |

| Т4 | n (%) |
|----------------------------------------|----------------|
| Current grade | |
| Gx | n (%) |
| G1 | n (%) |
| G2 | n (%) |
| G3 | n (%) |
| G4 | n (%) |
| Unknown | n (%) |
| Not Applicable | n (%) |
| Grade at Initial Diagnosis | |
| Gx | n (%) |
| G1 | n (%) |
| G2 | n (%) |
| G3 | n (%) |
| Unknown | n (%) |
| Not Applicable | n (%) |
| Years since initial diagnosis | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Months since recurrence | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Current TNM Staging: Primary Tumor (T) | |
| Tx | n (%) |
| TO | n (%) |
| T1 | n (%) |
| T1a | n (%) |
| T1b | n (%) |
| T2 | n (%) |
| T2a | n (%) |
| m01 | |
| T2b | n (%) |
| Т3 | n (%)<br>n (%) |
| | n (%) |

| T3b<br>T4<br>T4a<br>T4b<br>NA | n (%) n (%) n (%) n (%) n (%) |
|---|---|
| Current TNM Staging: Lymph Node (N) Nx N0 N1 NA | n (%)<br>n (%)<br>n (%)<br>n (%) |
| Current TNM Staging: Metastasis (M) M0 M1 M1a M1b | n (%)<br>n (%)<br>n (%)<br>n (%) |
| Initial TNM Staging: Primary Tumor (T) Tx T0 T1 T1a T1b T2 T2a T2b T3 T3a T3b T4 T4a T4b NA | n (%) |
| Initial TNM Staging: Lymph Node (N) Nx N0 N1 NA | n (%)<br>n (%)<br>n (%)<br>n (%) |
| Initial TNM Staging: Metastasis (M) | |

| MO | n (%) |
|--------------------------|-----------|
| M1 | n (%) |
| M1a | n (%) |
| M1b | n (%) |
| Number of prior regimens | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Prior regimen categories | |
| 1 | n (%) |
| 2 | n (%) |
| 3 | n (%) |
| >3 | n (%) |
| Prior IDH1 therapy | |
| Yes | n (%) |
| No | n (%) |

Programming note: repeat for 14.1.3.2c (Safety Population)


### Table 14.1.3.1d

# Baseline Disease Characteristics (Cohort 4, Response Evaluable Population)

| | | Cohort 4A: | Cohort 4B: | Cohort 4: |
|---|---|---|---|---|
| Parameter | Statistic | FT-2102 | FT-2102 +<br>GemCis | Overall |
| | | (N = ) | (N = ) | (N = ) |
| Commant Stars | | | | |
| Current Stage<br>I | - (0) | | | |
| IA | n (%) | | | |
| | n (%) | | | |
| IB | n (%) | | | |
| IIA | n (%) | | | |
| IIB | n (%) | | | |
| IIIA | n (%) | | | |
| IIIB | n (%) | | | |
| IVA | n (%) | | | |
| IVB | n (%) | | | |
| NA | n (%) | | | |
| Initial Stage | | | | |
| I | n (%) | | | |
| IA | n (%) | | | |
| IB | n (%) | | | |
| IIA | n (%) | | | |
| IIB | n (%) | | | |
| IIIA | n (%) | | | |
| IIIB | n (%) | | | |
| IVA | n (%) | | | |
| IVB | n (%) | | | |
| NA | n (%) | | | |
| Current Grade | | | | |
| Gx | n (%) | | | |
| G1 | n (%) | | | |
| G2 | n (%) | | | |
| G3 | n (%) | | | |
| Unknown | n (%) | | | |
| Not Applicable | n (%) | | | |
| wer whatteante | 11 ('0) | | | |

| Grade at Initial Diagnosis | |
|------------------------------------------|-----------|
| Gx | n (%) |
| G1 | n (%) |
| G2 | n (%) |
| G3 | n (%) |
| Unknown | n (%) |
| Not Applicable | n (%) |
| Years since initial diagnosis | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Months since recurrence | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Current TNM Staging: Primary Tumor (T) | |
| Tx | n (응) |
| TO | n (응) |
| Tis | n (응) |
| T1 | n (%) |
| T2 | n (%) |
| T3 | n (%) |
| T4 | n (%) |
| NA | n (%) |
| Company Mills Observer Towards Nada (NI) | |
| Current TNM Staging: Lymph Node (N) | - (0) |
| Nx | n (%) |
| NO | n (%) |
| N1 | n (%) |
| NA | n (%) |
| Current TNM Staging: Metastasis (M) | |
| M0 | n (%) |
| M1 | n (%) |
| NA | n (%) |
| 1411 | 11 (.0) |

| Initial TNM Staging: Primary Tumor (T) | |
|----------------------------------------|-----------------|
| Tx | n (%) |
| TO | n (%) |
| Tis | n (%) |
| T1 | n (%) |
| Т2 | n (%) |
| T3 | n (%) |
| T4 | n (%) |
| NA | n (%) |
| Initial TNM Staging: Lymph Node (N) | |
| Nx | n (%) |
| NO | n (%) |
| N1 | n (%) |
| NA | n (%) |
| Initial TNM Staging: Metastasis (M) | |
| M0 | n (%) |
| M1 | n (%) |
| NA | n (%) |
| M | 11 (%) |
| Number of prior regimens | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Prior regimen categories | |
| 1 | n (%) |
| 2 | n (%) |
| 3 | n (%) |
| >3 | n (%) |
| Prior INU1 therapy | |
| Prior IDH1 therapy | n (%) |
| Yes | n (%) |
| | n (%)<br>n (%) |
| Yes | |
| Yes<br>No | n (%) |
| Yes<br>No | n (%) |
| Yes<br>No | n (%) n mean |
| Yes<br>No | n (%) n mean SD |

| Child-Pugh Category | |
|---------------------|-------|
| A | n (%) |
| В | n (%) |
| _ C | n (%) |

Programming note: repeat for 14.1.3.2d (Safety Population)


Protocol 2102-ONC-102

Table 14.1.3.1e

# Baseline Disease Characteristics (Cohort 5, Response Evaluable Population)

| | | Cohort 5: |
|-------------------------------|-----------|-----------|
| Parameter | Statistic | Overall |
| | | N (%) |
| Current Stage | | |
| I | n (%) | |
| IA | n (%) | |
| IB | n (%) | |
| IIA | n (%) | |
| IIB | n (%) | |
| IIIA | n (%) | |
| IIIB | n (%) | |
| IVA | n (%) | |
| IVB | n (%) | |
| NA | n (%) | |
| Initial Stage | | |
| I | n (%) | |
| IA | n (%) | |
| IB | n (%) | |
| IIA | n (%) | |
| IIB | n (%) | |
| IIIA | n (%) | |
| IIIB | n (%) | |
| IVA | n (%) | |
| IVB | n (%) | |
| NA | n (%) | |
| Years since initial diagnosis | n | |
| - | mean | |
| | SD | |
| | median | |
| | min - max | |
| Months since recurrence | n | |

| | mean<br>SD<br>median<br>min - max |
|---|---|
| Current TNM Staging: Primary Tumor (T) Tx T0 Tis T1 T2 T3 T4 NA | n (%) |
| Current TNM Staging: Lymph Node (N) Nx N0 N1 N2 N3 | n (%) n (%) n (%) n (%) n (%) n (%) |
| Current TNM Staging: Metastasis (M) M0 M1 NA | n (%)<br>n (%)<br>n (%) |
| <pre>Initial TNM Staging: Primary Tumor (T) Tx T0 Tis T1 T2 T3 T4 NA</pre> | n (%) |
| <pre>Initial TNM Staging: Lymph Node (N) Nx N0</pre> | n (%)<br>n (%) |

DATE: HH:MM/DDMMMYYYY

| N1 | n (%) |
|-------------------------------------|-----------|
| N2 | n (%) |
| N3 | n (%) |
| NA | n (%) |
| Initial TNM Staging: Metastasis (M) | |
| M0 | n (%) |
| M1 | n (%) |
| NA | n (%) |
| Number of prior regimens | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Prior regimen categories | |
| 1 | n (%) |
| 2 | n (%) |
| 3 | n (%) |
| >3 | n (%) |
| <i>7</i> 3 | 11 (%) |
| Prior IDH1 therapy | |
| Yes | n (%) |
| No | n (%) |
| Child-Pugh Score | n |
| | mean |
| | SD |
| | median |
| | min - max |
| Child-Pugh Category | |
| A | n (%) |
| В | n (%) |
| С | n (%) |

Programming note: repeat for 14.1.3.2e (Safety Population)

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

#### Table 14.1.4.1a

### IDH1 and Other Mutations (Cohort 1, Response Evaluable Population)

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|-----------------------|-----------|------------|---------------|-----------|
| Parameter | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| | | (N = ) | (N = ) | (N = ) |
| IDH1 Mutation Subtype | | | | |
| R132C | n (%) | | | |
| R132H | n (%) | | | |
| R132S | n (%) | | | |
| R132L | n (%) | | | |
| R132G | n (%) | | | |
| Other | n (%) | | | |
| Unknown | n (%) | | | |
| Other mutations | | | | |
| ABL1 | n (%) | | | |
| ABL2 | n (%) | | | |
| ARID1A | n (%) | | | |
| ARID2 | n (%) | | | |
| AXIN1 | n (%) | | | |
| (etc.) | n (%) | | | |

#### Programming notes:

For other mutations show all mutations where at least 1 patient had the mutation. List them in alphabetical order. If a patient notes a mutation in the other, specify field then also show that mutation in this list.

Repeat for Cohorts 2-5
Repeat for 14.1.4.2a-14.1.4.2e (Safety population)


DATE: HH:MM/DDMMMYYYY

Protocol 2102-ONC-102

Table 14.1.5a

Prior Therapies (Cohort 1, Response Evaluable Population)

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|--------------|-----------|------------|---------------|-----------|
| Parameter | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| | | (N = ) | (N = ) | (N = ) |
| Drug class 1 | n (%) | | | |
| ATC text 1 | n (%) | | | |
| ATC text 2 | n (%) | | | |
| ATC text 3 | n (%) | | | |
| etc. | n (%) | | | |
| Drug class 2 | n (%) | | | |
| ATC text 1 | n (%) | | | |
| ATC text 2 | n (%) | | | |
| ATC text 3 | n (%) | | | |
| etc. | n (%) | | | |

.

Repeat for Cohorts 2-5 (Response Evaluable Population) Repeat for 14.1.5.2a-e (Safety Population)

Note: Prior anti-cancer therapy medications are coded with the WHO Drug version March 2018.

DATE: HH:MM/DDMMMYYYY

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Table 14.1.6a

### Medical History (Cohort 1, Safety Population)

| Parameter | Statistic | Cohort 1A:<br>FT-2102 | Cohort 1B:<br>FT-2102 + AZA | Cohort 1:<br>Overall |
|---|---|---|---|---|
| | | (N = ) | (N = ) | (N = ) |
| OC | n (%) | | | |
| PT1 | n (%) | | | |
| PT2 | n (%) | | | |
| PT3 | n (%) | | | |
| etc. | n (%) | | | |
| SOC2 | n (%) | | | |
| PT1 | n (%) | | | |
| PT2 | n (%) | | | |
| PT3 | n (%) | | | |
| etc. | n (%) | | | |

Repeat for Cohorts 2-5

Note: Medical Histories are coded with the MedDRA version 21.0.


### Table 14.2.1a

Disease Response Assessment Overall and by Subgroups (Cohort 1, Response Evaluable Population)

| Parameter | Statistic | Cohort 1A:<br>FT-2102<br>(N = ) | Cohort 1B:<br>FT-2102 + AZA<br>(N = ) | Cohort 1: Overall (N = ) |
|---|---|---|---|---|
| Best overall response | n (%) | | | |
| Complete response (CR) | n (%) | | | |
| Partial response (PR) | n (%) | | | |
| Minor response (MR) | n (%) | | | |
| Stable disease (SD) | n (%) | | | |
| Progression (PD) | n (%) | | | |
| Not evaluable | n (%) | | | |
| Overall response rate (ORR) | n (%) | | | |
| ORR by subgroups: | | | | |
| Gender | | | | |
| Male | | | | |
| Responder | n (%) | | | |
| Non-Responder | n (%) | | | |
| Female | | | | |
| Responder | n (%) | | | |
| Non-Responder | n (%) | | | |
| Race (Caucasian yes/ no) | | | | |
| Caucasian | | | | |
| Responder | n (%) | | | |
| Non-Responder | n (%) | | | |
| Non-Caucasian | | | | |
| Responder | n (%) | | | |
| Non-Responder | n (%) | | | |
| Baseline ECOG<br>0/1 | | | | |
| Responder | n (%) | | | |

| | | | (0) |
|-------|-----------------------------------------|----|-------|
| 2 | Non-Responder | n | (응) |
| ۷ | Responder | n | (왕) |
| | Non-Responder | | (응) |
| | non Noopondor | | ( 0 ) |
| Age C | ategory | | |
| 18 | -40 | | |
| | Responder | n | (%) |
| | Non-Responder | n | (%) |
| 41 | -59 | | |
| | Responder | n | (응) |
| | Non-Responder | n | (응) |
| >= | 60 | | |
| | Responder | | (응) |
| | Non-Responder | n | (응) |
| Drion | thorany | | |
| | therapy<br>rgery only | | |
| Su | Responder | n | (왕) |
| | Non-Responder | | (응) |
| S11 | rgery and medication | 11 | ( 0) |
| 54 | Responder | n | (응) |
| | Non-Responder | | (응) |
| | Non Responder | | ( 0 ) |
| Numbe | r of prior regimens | | |
| 1 | | | |
| | Responder | n | (왕) |
| | Non-Responder | n | (응) |
| 2 | | | |
| | Responder | n | (응) |
| | Non-Responder | n | (왕) |
| 3 | | | |
| | Responder | | (응) |
| | Non-Responder | n | (%) |
| >3 | | | |
| | Responder | | (응) |
| | Non-Responder | n | (%) |
| Prior | IDH1 therapy | | |
| Ye | | | |
| | Responder | n | (응) |
| | Non-Responder | | (왕) |
| | ± * | | / |

| No | | | |
|--------|-------------------|----|-------|
| | Responder | n | (응) |
| | Non-Responder | n | (응) |
| Prior | temozolomide | | |
| Ye | s | | |
| | Responder | n | (%) |
| | Non-Responder | n | (%) |
| No | | | |
| | Responder | n | (왕) |
| | Non-Responder | n | (응) |
| Prior | radiation therapy | | |
| Ye | | | |
| 10. | Responder | n | (응) |
| | Non-Responder | | (왕) |
| No | <del>-</del> | | ( 0 ) |
| 2.0 | Responder | n | (응) |
| | Non-Responder | | (왕) |
| | Non Responder | 11 | ( 0 ) |
| Baseli | ine steroids | | |
| Ye | s | | |
| | Responder | n | (%) |
| | Non-Responder | n | (왕) |
| No | | | |
| | Responder | n | (응) |
| | Non-Responder | n | (%) |
| Baseli | ine tumor grade | | |
| I | ine camer grade | | |
| _ | Responder | n | (응) |
| | Non-Responder | n | |
| II | | 11 | ( 0 ) |
| | Responder | n | (응) |
| | Non-Responder | n | |
| II | | | ( - , |
| | Responder | n | (왕) |
| | Non-Responder | n | |
| IV | <del>-</del> | | , - / |
| | Responder | n | (응) |
| | Non-Responder | n | |

| IDH mutation subtype | | |
|----------------------|------|-----|
| R132H | | |
| Responder | n | (응) |
| Non-Responder | n | (응) |
| R132C | | |
| Responder | n | (응) |
| Non-Responder | n | (응) |
| other R132 subtype | es : | |
| Responder | n | (응) |
| Non-Responder | n | (응) |

Repeat for Cohorts 2-5

Programming note: for cohorts 2 and 4, refer to SAP for cohort-specific subgroups to add to the table, not shown in this shell.

For cohorts 2 and higher, remove MR as a response option.

DATE: HH:MM/DDMMMYYYY

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Figure 14.2.2.1a

Best Percent Change from Baseline in Tumor Burden (Cohort 1 Single Agent, Response Evaluable Population)



Note: Baseline is the last imaging assessment performed before the patient's first dose of FT-2102.

Note: Best percent change is defined as maximum percentage reduction or minimum percentage increase at a single time point of the patient's tumor burden post first dose of study drug.

Programming note: color code the bars by best overall response

Programming note: Y-axis should be labeled "Maximum Decrease from Baseline (%)"

Programming note: for Cohort 1, reference line should be at -50% for Cohort 1, and -30% for other cohorts.

Programming note: Repeat for 14.2.2.2a-e (Combination Therapy)

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

### Figure 14.2.3.1a

### Time on Treatment (Cohort 1 Single Agent, Safety Population)



Programming note: Repeat for 14.2.3.2a-e (Time on Treatment Combination Therapy)

Programming note: color code by appropriate best overall response criteria, depending on Cohort being summarized. This figure is for example only, the response categories used above are not to be used, follow appropriate disease-based response criteria.

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Table 14.2.4a

Progression Free Survival, Time to Progression, Duration of Response, and Time to Response (Cohort 1, Response Evaluable Population)

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|-----------|-----------|------------|---------------|-----------|
| Parameter | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| | | (N = ) | (N = ) | (N = ) |

Progression free survival (PFS; weeks) Patients with event n (%) Censored Patients n (%) PFS median 95% CI for median 25-75%ile min - max Time to progression (TTP; weeks) Patients with event n (%) Censored Patients n (%) TTP median 95% CI for median 25-75%ile min - max Duration of response (DOR; weeks) Patients with event n (응) Censored Patients n (%) DOR n median 95% CI for median 25-75%ile min - max Time to response (TTR; weeks) TTR n median 95% CI for median 25-75%ile min - max

Repeat for Cohorts 2-5

DATE: HH:MM/DDMMMYYYY

Note: Progression Free Survival (PFS) is defined as the time from the date of the first dose to the date of disease progression or death, whichever is sooner. Time to Progression (TTP) is defined as the time from the date of the first dose to the date of disease progression. Duration of Response (DOR) is defined as the time from the date of the first CR, PR, or MR response to the date of disease progression. Time to Response (TTR) is defined as the time from the date of first dose to the date of first CR, PR or MR response.


Protocol 2102-ONC-102 Table 14.2.5.1

Overall Survival (Response Evaluable Population)

| Parameter | Statistic | FT-2102 | FT-2102 combination | Overall |
|-----------|-----------|---------|---------------------|---------|
| 9 | | (N = ) | (N = ) | (N = ) |

```
Cohort 1
  Overall survival (weeks)
     Patients with event
                                                       n (%)
     Censored Patients
                                                       n (%)
     OS
                                                       median
                                                       95% CI for median
                                                      25-75%ile
                                                      min - max
Event free Rate (95% CI)
     3 months
                                                       응 (응, 응)
                                                       용(용,용)
     6 months
     9 months
                                                       응 (응, 응)
                                                       용(용,용)
     12 months
Cohort 2
 Overall survival (weeks)
     Patients with event
                                                       n (%)
     Censored Patients
                                                       n (%)
     OS
                                                       median
                                                       95% CI for median
                                                      25-75%ile
                                                      min - max
Event free Rate (95% CI)
     3 months
                                                      응(응,용)
     6 months
                                                       용(용,용)
                                                       응(응,용)
     9 months
                                                       응 (응, 응)
     12 months
Cohort 3
  Overall survival (weeks)
```

```
Patients with event
                                                       n (%)
     Censored Patients
                                                       n (%)
                                                       median
                                                       95% CI for median
                                                       25-75%ile
                                                       min - max
Event free Rate (95% CI)
     3 months
                                                       응 (응, 응)
     6 months
                                                       응 (응, 응)
                                                       응 (응, 응)
     9 months
                                                       응 (응, 응)
     12 months
Cohort 4
 Overall survival (weeks)
     Patients with event
                                                       n (%)
                                                       n (%)
     Censored Patients
     OS
                                                       median
                                                       95% CI for median
                                                       25-75%ile
                                                       min - max
Event free Rate (95% CI)
     3 months
                                                       응(응,응)
                                                       응 (응, 응)
     6 months
                                                       응 (응, 응)
     9 months
                                                       응(응,응)
     12 months
Cohort 5
 Overall survival (weeks)
     Patients with event
                                                       n (%)
     Censored Patients
                                                       n (%)
                                                       n
                                                       median
                                                       95% CI for median
                                                       25-75%ile
                                                       min - max
Event free Rate (95% CI)
                                                       용 (용,용)
     3 months
                                                       응 (응, 응)
     6 months
                                                       응(응,응)
     9 months
                                                       응(응,응)
     12 months
```

FORMA Therapeutics 2102-ONC-102 Statistical Analysis Plan 28 June 2019, Version 2.0

Programming note: repeat for 14.2.5.2 (Safety Population)

DATE: HH:MM/DDMMMYYYY

Note: Overall Survival (OS) is defined as the time from the date of the first dose to the date of death.

0

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Table 14.2.5.3a

Kaplan-Meier Plot of Overall Survival (Cohort 1, Response Evaluable Population)



Program: EXAMPLE.sas Run: 25SEP2013 09:40, Dataset: SASHELP.BMT

13

11

21

Treatment 2

45

Note: Overall Survival (OS) is defined as the time from the date of the first dose to the date of death.

10

Programming note: Present different lines for single agent and combination arms, rather than treatments. Repeat for cohorts 2-5.

Repeat for 14.2.5.4a-e Overall Survival(Safety Population), 14.2.5.5a-e Progression Free Survival (Response Evaluable Population), 14.2.5.6a-e Progression Free Survival (Safety Population)

Protocol 2102-ONC-102

rtial Page 1 of x

### Table 14.2.6a

# Serum AFP, CA19-9, and CEA (Cohort 2, Safety Population)

| | | Cohort 2A: | | | Cohort 2B: | | | Cohort 2: | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Statisti<br>c | | FT-2102 (N = ) | | | FT-2102 + AZA $(N = )$ | | | Overall | |
| | | | | | | | | | (N = ) | |
| | | Value | Change<br>from BL | Pct. Chg<br>fr BL | Value | Change<br>from BL | Pct. Chg<br>fr BL | Value | Change<br>from BL | Pct. Chg fr<br>BL |
| Serum AFP | | | | | | | | | | |
| Pre-Dose C1 | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | XX.X |
| | median | XX | XX | XX | XX | XX | XX | xx | XX | XX |
| | min - | xx - | | | xx - | | | xx - | | |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| C3 | n | XX | XX | xx | XX | XX | xx | XX | XX | XX |
| | mean | xx | XX | XX | XX | XX | XX | xx | XX | XX |
| | SD | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x | XX.X | XX.X |
| | median | xx | XX | XX | XX | XX | XX | xx | XX | XX |
| | min - | xx - | | | xx - | | | xx - | | |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| (continue for | | | | | | | | | | |
| all cycles | | | | | | | | | | |
| present in data) | n | xx | XX | XX | XX | XX | XX | xx | XX | XX |
| <u>.</u> | mean | xx | XX | XX | XX | XX | XX | xx | XX | XX |
| | SD | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x | XX.X | XX.X |
| | median | xx | XX | XX | xx | XX | XX | xx | XX | XX |
| | min - | xx - | | | xx - | | | xx - | | |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| CA19-9 | | | | | | | | | | |
| Pre-Dose C1 | n | XX | xx | xx | XX | xx | xx | XX | xx | xx |
| | mean | xx | xx | XX | xx | XX | XX | xx | XX | XX |
| | SD | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | | xx - | | | xx - | | - |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | xx | xx - xx | xx - xx |

| C3 | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
|---|---|---|---|---|---|---|---|---|---|---|
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | | xx - | | | xx - | | |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| (continue for all cycles | | | | | | | | | | |
| present in data) | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | | xx - | | | xx - | | |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| CEA | | | | | | | | | | |
| Pre-Dose C1 | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | | xx - | | | xx - | | |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| C3 | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | | xx - | | | xx - | | |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| (continue for all cycles | | | | | | | | | | |
| present in data) | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | | xx - | | | XX - | | |
| | max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |

Programming note: repeat for Cohort 4

DATE: HH:MM/DDMMMYYYY

Note: BL = baseline.

Note: Baseline is defined as the most recent measurement prior to the first administration of study drug.
FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Figure 14.2.7a

Serum AFP, CA19-9, and CEA (Cohort 2, Response Evaluable Population)



Programming note; Different colors indicate single agent and combination therapy. Please include legend indicating this. Programming note; please include value and unit on Y-axis
Programming note: via proc SGPANEL, matrix to include Serum AFP, CA19-9, and CEA on a single page.

Repeat for Cohort 4


Protocol 2102-ONC-102

Table 14.2.8a

# EQ-5D-5L Summary (Cohort 1, Response Evaluable Set)

| | | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|---|---|---|---|---|---|
| Dimension | Level | Statistic | FT-2102 | FT-2102<br>combination | Overall |
| Visit | | | (N = ) | (N = ) | (N = ) |
| Mobility | | | | | |
| C1 | 1 (no problems) | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 2 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 3 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 4 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 5 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | Total | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | Number reporting some problems | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | Change from BL in number reporting some problems | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| C3 | 1 (no problems) | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 2 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 3 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 4 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 5 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | Total | n (%) | xx (xx.x% | ) | xx (xx.x%) |
| | Number reporting some problems | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | Change from BL in number reporting some problems | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| Treatment Termination | 1 (no problems) | n (응) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |
| | 2 | n (%) | xx (xx.x% | ) xx (xx.x%) | xx (xx.x%) |

DATE: HH:MM/DDMMMYYYY

| 3 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|
| 4 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 5 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number reporting some problems | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Change from BL in number reporting some problems | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Continue for other EQ-5D dimensions

### BL = baseline

Repeat for Cohorts 2-5

Note: Baseline is defined as the most recent measurement prior to the first administration of study drug.

Source: Data Listing 16.2.x

Protocol 2102-ONC-102
Figure 14.2.9a

EQ-5D-5L Quality of Life Assessment (Cohort 1, Response Evaluable Population)



### Programming notes:

TRT will be displayed at the top left of the page, or of each graph that is presented on the page, whichever is most expedient. Y-axis label is "Percent".

Bars will be shaded as shown in the legend.

All panels (Mobility, Self-care, Usual Activities, Pain/Discomfort and Anxiety/Depression) will be presented in a 2x3 matrix on a single page. (Programmer can use SGPANEL)


Table 14.2.10.1a

Summary of 2-HG, Change from Baseline, and Percent Change from Baseline (Cohort 1, PD Population)

| | | | | Cohort 12 | A: | | Cohort 1B | : | | Cohort 1 | : |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Time<br>Point | Statistic | | FT-2102 | | | FT-2102 + A | AZA | | Overall | - |
| | | | | (N = ) | | | (N = ) | | | (N = ) | |
| | | | Value | Change<br>from BL | Pct. Chg<br>fr BL | Value | Change<br>from BL | Pct.<br>Chg fr<br>BL | Value | Change<br>from BL | Pct. Chg<br>fr BL |
| 2-HG Plasma | Pre- | | | | | | | | | | |
| C1D1 | dose | n<br>mean<br>SD<br>median | xx<br>xx<br>xx.x<br>xx | xx<br>xx<br>xx.x<br>xx | xx<br>xx<br>xx.x<br>xx | xx<br>xx<br>xx.x<br>xx | xx<br>xx<br>xx.x<br>xx | xx<br>xx<br>xx.x<br>xx | xx<br>xx<br>xx.x<br>xx | xx<br>xx<br>xx.x<br>xx | xx<br>xx<br>xx.x<br>xx |
| | | min - max | xx - | xx - xx | xx - xx | xx - | xx - xx | xx - xx | xx - | xx - xx | xx - xx |
| C1D2 | 4 hours Pre- dose | n mean SD median min - max n mean | xx<br>xx<br>xx.x<br>xx<br>xx -<br>xx | xx<br>xx<br>xx.x<br>xx<br>xx<br>xx - xx | xx<br>xx<br>xx.x<br>xx<br>xx<br>xx - xx | xx<br>xx<br>xx.x<br>xx<br>xx<br>xx -<br>xx | xx<br>xx<br>xx.x<br>xx<br>xx<br>xx - xx | xx<br>xx<br>xx.x<br>xx<br>xx<br>xx - xx | xx<br>xx<br>xx.x<br>xx<br>xx -<br>xx | xx<br>xx<br>xx.x<br>xx<br>xx - xx | xx<br>xx<br>xx.x<br>xx<br>xx<br>xx |
| | | SD<br>median<br>min - max | xx.x<br>xx<br>xx -<br>xx | xx.x<br>xx<br>xx - xx | xx.x<br>xx<br>xx - xx | xx.x<br>xx<br>xx -<br>xx | xx.x<br>xx<br>xx - xx | xx - xx | xx.x<br>xx<br>xx -<br>xx | xx.x<br>xx<br>xx - xx | xx.x<br>xx<br>xx - xx |
| (continu e for all cycle/ days and time points) | | n | xx | xx | XX | xx | xx | XX | xx | xx | xx |
| POTITCS) | | | | | | | | | | | |
| | | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |

| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
|---|---|---|---|---|---|---|---|---|---|---|
| | median | xx<br>xx - | XX | XX | xx<br>xx - | XX | XX | xx - | XX | XX |
| | min - max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| C3 | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | xx.x | xx.x | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X | xx.x |
| | median | xx<br>xx - | XX | XX | xx<br>xx - | XX | XX | xx<br>xx - | XX | XX |
| | min - max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| (continu e for all cycles present in | | | | | | | | | | |
| data) | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | xx<br>xx - | XX | XX | xx<br>xx - | XX | XX | xx<br>xx - | XX | XX |
| | min - max | XX | xx - xx | xx - xx | xx | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| 2-HG CSF<br>(present all days/ | | | | | | | | | | |
| times) | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | xx<br>xx - | XX | XX | xx<br>xx - | XX | XX | xx<br>xx - | XX | XX |
| | min - max | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| 2-HG Urine<br>(present all days/ | n | XX | XX | XX | xx | XX | XX | XX | xx | XX |
| times) | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | XX | XX | XX | XX | XX | XX |

BL = Baseline

Programming note: repeat for

Cohorts 2-5

Note: Baseline is defined as the most recent measurement prior to the first administration of study drug.


Table 14.2.10.2a

# Summary of 2-HG, Change from Baseline, and Percent Change from Baseline by Subgroup (Cohort 1, PD Population)

| | | | | Cohort 1 | lA: | | Cohort 1 | 3: | | Cohort 1 | : |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Time<br>Point | Statistic | | FT-210 | 2 | | FT-2102 + | AZA | | Overall | |
| | | | | (N = | ) | | (N = ) | | | (N = ) | |
| | | | | Change<br>from | Pct. Chg | | Change | Pct. Chg | | Change | Pct. Chg |
| 2-HG Plasma | | | Value | BL | fr BL | Value | from BL | fr BL | Value | from BL | fr BL |
| C1D1 | Descri | | | | | | | | | | |
| Male | Pre-<br>dose | n | xx | XX | XX | XX | XX | XX | XX | XX | XX |
| TIGIC | dobe | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | SD | XX.X | XX.X | xx.x | XX.X | XX.X | xx.x | XX.X | xx.x | XX.X |
| | | median | XX | XX | XX | XX | xx | xx | XX | xx | xx |
| | | modium | xx - | xx - | | xx - | | | xx - | | |
| | | min - max | XX | XX | xx - xx | XX | xx - xx | xx - xx | XX | XX - XX | xx - xx |
| | Pre- | | | | | | | | | | |
| Female | dose | n | XX | xx | XX | XX | XX | XX | XX | XX | XX |
| | | mean | XX | xx | XX | xx | xx | XX | xx | xx | XX |
| | | SD | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x |
| | | median | XX | xx | XX | xx | xx | XX | xx | xx | XX |
| | | | xx - | xx - | | xx - | | | xx - | | |
| | | min - max | XX | XX | xx - xx | XX | xx - xx | XX - XX | XX | XX - XX | xx - xx |
| Male | 4 hours | n | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| | | mean | XX | xx | XX | xx | xx | XX | xx | xx | XX |
| | | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| | | median | xx<br>xx - | xx<br>xx - | XX | xx - | xx | xx | xx<br>xx - | xx | xx |
| | | min - max | XX | XX | xx - xx | XX | xx - xx | xx - xx | xx | xx - xx | xx - xx |
| Female | 4 hours | n | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| | | mean | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| | | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

| | median | XX | XX | XX | XX | XX | XX | XX | XX | XX |
|---|---|---|---|---|---|---|---|---|---|---|
| | | XX - | xx - | | xx - | | | xx - | | |
| | min - max | XX | XX | xx - xx | XX | xx - xx | XX - XX | XX | xx - xx | XX - XX |
| C1D1 | | | | | | | | | | |
| Predose | n | XX | xx | XX | xx | xx | XX | xx | xx | XX |
| Male | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | xx | XX | XX | XX | XX | XX |
| | | xx - | xx - | | xx - | | | xx - | | |
| | min - max | XX | XX | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| Female | n | XX | XX | xx | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | xx | XX | XX | XX | XX | XX |
| | | xx - | xx - | | xx - | | | xx - | | |
| | min - max | XX | XX | xx - xx | XX | xx - xx | xx - xx | XX | xx - xx | xx - xx |
| etc. | | | | | | | | | | |

BL = Baseline

Programming note: continue for all

subgroups

Programming note: repeat for Cohorts

2-5

DATE: HH:MM/DDMMMYYYY

Note: Baseline is defined as the most recent measurement prior to the first administration of study drug.

Protocol 2102-ONC-102
Figure 14.2.11.1a

Plasma 2-HG by Time Point (Cohort 1, PD Population)



Programming note; Different colors indicate single agent and combination therapy. Please include legend indicating this. Programming note; please include value and unit on Y-axis

Repeat for Cohorts 2-5.

Repeat for Figure 14.2.11.2 Urine 2-HG, Figure 14.2.11.3 MRS 2-HG, and Figure 14.2.11.4 CSF 2-HG


Table 14.2.12a

| Summary | of | Phamacokinetic | Concentration | over | Time | (Cohort 1 | , Pharmacokinetic | Population) |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|-------------------|-----------|------------|---------------|-----------|
| | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| Visit, Time Point | | (N = ) | (N = ) | (N = ) |

Cycle 1, 1 Hour n mean SD CV (%) Geometric mean Geometric SD median min - max Cycle 1, 2 Hours mean SD Geometric mean Geometric SD median min - max Cycle 1, 4 Hours n mean Geometric mean Geometric SD median min - max Etc. for all time points and overall n mean SD Geometric mean Geometric SD

median min - max

Repeat for Cohorts 2-5 )  $Programming \ note: \ summarize \ all \ cycles \ where \ n \ is \ 3 \ or \ more.$ 


Table 14.2.13a

# Summary of Phamacokinetic Parameters (All Patients on Single Agent Therapy, Pharmacokinetic Population)

AUC0-24

n

mean SD

CV (%)

Geometric mean Geometric SD

median min - max

median min - max

Etc. for all parameters

n mean

geometric mean geometric SD

median min - max

Repeat for Cohorts 1-5

)

Programming note: summarize all cycles where n is 3 or more.

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Table 14.2.14.1a

Geometric Mean FT-2102 Plasma Concentration over Time (Cohort 1, PK Population)



Note: Only one line is needed. Plot geometric mean and use geometric SD for error bars.

# Repeat for:

Figure 14.2.14.1 Cohorts 2-5

Figure 14.2.14.2 FT-2102 Plasma Concentration over Log-Time (Cohort 1, PK Population), but modify x axis so that it is on the

og scale.

Figure 14.2.15a-f FT-2102 Geometric Mean Plasma Concentration over Nominal Time (PK Population)

| FORMA Therapeutics Protocol 2102-ONC-102 | Confidential | | | Page 1 of x |
|---|---|---|---|---|
| Protocol 2102-UNC-102 | Table 14.2.16 | .1a | | |
| | Summary of FT-2102 Expos | ure (Cohort 1) | | |
| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
| Visit | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| Parameter | | (N = ) | (N = ) | (N = ) |
| Overall | | | | |
| Duration of FT-2102 exposure (days) | n<br>mean<br>SD<br>median<br>min - max | | | |
| Total dose FT-2102 taken (mg) | n<br>mean<br>SD<br>median<br>min - max | | | |
| Percent compliance | n<br>mean<br>SD<br>median<br>min - max | | | |
| C1 Duration of FT-2102 exposure (days) | n<br>mean<br>SD<br>median<br>min - max | | | |
| Total dose FT-2102 taken (mg) | n<br>mean<br>SD<br>median<br>min - max | | | |

DATE: HH:MM/DDMMMYYYY

Percent compliance

n mean SD median min - max

(etc. Summarize all cycles where there are 3 or more Patients overall).

Repeat for Cohorts 2-5

Repeat for 14.2.16.2 (Safety Population)


Table 14.2.17a

Summary of Azacitidine Exposure (Cohort 1, Safety Population)

Cohort 1B: Visit Statistic FT-2102 + AZA (N = )Parameter Overall Duration of azacitidine exposure (days) n mean SD median min - max Number of doses of azacitidine n mean median

Number of patients with azacitidine dose interruptions

mean
SD
median
min - max

min - max

| Adverse Event | n (%) |
|----------------------------------------|-------|
| Other | n (%) |
| per of Patients with Dose Modification | as |
| e Reduced | n (%) |
| e Increased | n (%) |
| e Held | n (%) |
| e Withdrawn | n (%) |

Repeat for Cohorts 2-4, per appropriate combo drug

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Table 14.3.1.1a

### Summary of Adverse Events (Cohort 1, Safety Population)

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|---|---|---|---|---|
| Parameter | Statistic | FT-2102 | FT-2102 +<br>AZA | Overall |
| | | (N = ) | (N = ) | (N = ) |
| Patients with any AE | n (%) | | | |
| Patients with any TEAE | n (%) | | | |
| Patients with any Grade 3 or greater TEAE | n (%) | | | |
| Patients with any Grade 4 or greater TEAE | n (%) | | | |
| Patients with any Grade 5 TEAE | n (%) | | | |
| Patients with DLT | n (%) | | | |
| Patients with SAE | n (%) | | | |
| Patients with treatment emergent SAE | n (%) | | | |
| Patients with FT-2102 related TEAE | n (%) | | | |
| Patients with azacitidine related TEAE | n (%) | | | |
| Deticate with DM 2102 related treatment amount CAD | - (8) | | | |
| Patients with FT-2102 related treatment emergent SAE | n (%) | | | |
| Patients with TEAE related to FT-2102 resulting in dose interruption | n (%) | | | |
| Patients with TEAE related to FT-2102 resulting in dose withdrawal | . (0) | | | |
| Withdrawai | n (%) | | | |
| Patients with TEAE related to FT-2102 resulting in dose reduction | n (%) | | | |
| Patients with TEAE related to azacitidine resulting in dose | (0) | | | |
| interruption | n (%) | | | |
| Patients with TEAE related to azacitidine resulting in dose withdrawal | n (%) | | | |
| Patients with TEAE related to azacitidine resulting in dose reduction | n (응) | | | |

# Repeat for Cohorts 2-5

Programming note: when programming tables for cohorts 2-5, substitute the appropriate combination agent for the cohort. Cohorts 1 & 3 have azacitidine, cohort 2 has nivolumab, cohort 4 has gem/cis, cohort 5 has no combination therapy.

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Table 14.3.1.2a

## Treatment Emergent Adverse Events by MedDRA SOC and PT (Cohort 1, Safety Population)

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|---|---|---|---|---|
| System Organ Class (SOC) | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| Preferred Term (PT) | | (N = ) | (N = ) | (N = ) |
| SOC 1 | n (%) | | | |
| PT 1 | n (%) | | | |
| PT 2 | n (%) | | | |
| PT 3 | n (%) | | | |
| PT 4 | n (%) | | | |
| etc. for all terms | n (%) | | | |
| SOC 2 | n (%) | | | |
| PT 1 | n (%) | | | |
| PT 2 | n (%) | | | |
| PT 3 | n (%) | | | |
| PT 4 | n (%) | | | |
| etc. for all terms | n (%) | | | |

Repeat for Cohorts 2-5

Programming note: repeat for:

Table 14.3.1.3: Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Safety Population)
Table 14.3.1.4: Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Cohort 1, Safety Population)
Table 14.3.1.5: Severe Treatment-Emergent Adverse Events Related to FT-2102 by MedDRA System Organ Class and Preferred Term (Cohort 1, Safety Population)


Table 14.3.1.6a

Treatment Emergent Adverse Events by MedDRA Preferred Term (Cohort 1, Safety Population)

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|---------------------|-----------|------------|---------------|-----------|
| | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| Preferred Term (PT) | | (N = ) | (N = ) | (N = ) |
| PT 1 | n (%) | | | |
| PT 2 | n (%) | | | |
| PT 3 | n (%) | | | |
| PT 4 | n (%) | | | |
| etc. for all terms | n (%) | | | |

Repeat for Cohorts 2-5

Programming note: sort preferred terms from most frequent to least frequent, based on the overall column.

DATE: HH:MM/DDMMMYYYY

Note: Patients are counted once in each SOC and PT. Adverse Events are coded with the MedDRA version 21.0.


DATE: HH:MM/DDMMMYYYY

Table 14.3.2.1

Listing of Deaths (Safety Population)

Cohort Patient Date of Last Dose Date of Death Rel Day Primary Cause of Death AE #


Table 14.3.2.2

Listing of Serious Adverse Events (Safety Population)

| | | | Start | Stop | CTCAE | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Verbatim | Date/ | Date/ | Grade/ | | Relationship to | Action Taken with | Other Action |
| Cohort | Patient | Term | Rel Day | Rel Day | SAE | Outcome | Drug | Study Drug | Taken |

FT-2102: unrelated FT-2102: None

Aza: Drug

Aza: related interrupted

Programming note: in relationship and action columns, precede the information with the drug name being given in combination with FT-2102.

DATE: HH:MM/DDMMMYYYY

Note: The combination drug is Azacitidine in cohort 1b and 3b, Nivolumab in cohort 2b, and Gemcitibine + Cisplatin in cohort 4b.

<sup>1</sup> Relationship to Drug: None, REM = Remote, POS= Possible, PROB= Probable, DEF= Definite and NA= Not Applicable

<sup>&</sup>lt;sup>2</sup> Action Taken with Study Drug: None = Dose Not Changed; INT = Dose Interrupted; RED = Dose Reduced; WD = Drug Withdrawn.


Table 14.3.2.3

Listing of Adverse Events Resulting in Drug Interruptions or Withdrawals (Safety Population)

| Cohort | Patient | Verbati<br>m Term | Start<br>Date/<br>Rel Day | Stop<br>Date/<br>Rel Day | CTCAE<br>Grade | SAE | Outcome | Relationship to<br>Drug | Action Taken<br>with Study Drug | Other Action<br>Taken |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | FT-2102:<br>definite | FT-2102: Drug<br>Withdrawn | |

Programming note: in relationship and action columns, precede the information with the drug name being given in combination with FT-2102.

DATE: HH:MM/DDMMMYYYY

Note: The combination drug is Azacitidine in cohort 1b and 3b, Nivolumab in cohort 2b, and Gemcitibine + Cisplatin in cohort 4b.

- 1 Relationship to Drug: None, REM = Remote, POS= Possible, PROB= Probable, DEF= Definite and NA= Not Applicable
- <sup>2</sup> Action Taken with Study Drug: None = Dose Not Changed; INT = Dose Interrupted; RED = Dose Reduced; WD = Drug Withdrawn.


Table 14.3.2.4

Listing of Dose Limiting Toxicities (Safety Population)

| Cohort | Patient | Verbatim<br>Term | Start<br>Date/<br>Rel Day | Stop<br>Date/<br>Rel Day | CTCAE<br>Grade | SAE | Outcome | Relationship to<br>Drug | Action Taken<br>with Study Drug | Other Action<br>Taken |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | FT-2102:<br>definite | FT-2102: Drug<br>Withdrawn | |

Programming note: in relationship and action columns, precede the information with the drug name being given in combination with FT-2102.

Note: The combination drug is Azacitidine in cohort 1b and 3b, Nivolumab in cohort 2b, and Gemcitibine + Cisplatin in cohort 4b.

<sup>&</sup>lt;sup>1</sup> Relationship to Drug: None, REM = Remote, POS= Possible, PROB= Probable, DEF= Definite and NA= Not Applicable

<sup>&</sup>lt;sup>2</sup> Action Taken with Study Drug: None = Dose Not Changed; INT = Dose Interrupted; RED = Dose Reduced; WD = Drug Withdrawn.


Table 14.3.4.1

Listing of Abnormal Laboratory Values (Safety Population)

CTCAE Laboratory Sample Rel Visit Grade/ Clinical Test Cohort Patient Category Name date Name Units LLN ULN Flag Significance Day Result

Chemistry
Hematology
Urine

DATE: HH:MM/DDMMMYYYY

Programming note: Repeat for table 14.3.4.2 Listing of Laboratory Values with CTCAE Grade 3 or Higher (Safety Population)
Programming note: for CTCAE Grade/ Flag, show CTCAE grade if the lab test is graded via CTCAE criteria. If not, indicate H
for above upper limit of normal or L for below lower limit of normal


Table 14.3.4.3

Listing of Liver Function Tests of Potential Concern (Safety Population)

| | | | | | | | | | | | | | Concurrent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | AST, ALT |
| | | | | | | | | | | | | Concurrent | and Total |
| | | | | | | | | | | | | AST, ALT | Bilirubin, |
| | | Test | Sample | Rel | Visit | | | | Result | CTCAE | Clinical | and Total | without ALP |
| Cohort | Patient | Name | date | Day | Name | Result | Units | ULN | xULN | Grade | Significance | Bilirubin | abnormality |

Programming Note: present data supporting table 14.3.7. Only those lab test results should be presented.

Programming Note: result x ULN should be the derived value (result/ULN) rounded to one decimal.

Programming Note: Concurrent columns should indicate which abnormal results qualified for the "concurrent" flags in table 14.3.7.


Table 14.3.5.1a

Summary of Hematology and Coagulation Results and Change from Baseline (Cohort 1, Safety Population)

| | | Coh | nort 1A: | Coh | ort 1B: | Co | hort 1: |
|---|---|---|---|---|---|---|---|
| Parameter | Stati<br>stic | F' | T-2102 | FT-2 | 102 + AZA | C | verall |
| | | (1 | N = ) | (1 | 4 = ) | ( | N = ) |
| | | Valu<br>e | Change<br>from BL | Valu<br>e | Change<br>from BL | Valu<br>e | Change<br>from BL |
| WBC (unit) | | | | | | | |
| C1D1 | | | | | | | |
| | n | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX |
| | SD<br>media | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x |
| | n | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | xx - | | xx - | |
| | max | XX | xx - xx | XX | XX - XX | XX | XX - XX |
| C1D8 | n | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX |
| | SD<br>media | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x |
| | n | XX | XX | XX | XX | XX | XX |
| | min - | XX - | | xx - | | XX - | |
| | max | XX | xx - xx | XX | XX - XX | XX | XX - XX |
| C1D15 | n | XX | XX | XX | xx | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX |
| | SD<br>media | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | n | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | xx - | | xx - | |
| | max | XX | xx - xx | XX | xx - xx | XX | xx - xx |
| C1D22 | n | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX |
| | SD<br>media | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | n | XX | XX | XX | xx | XX | xx |

DATE: HH:MM/DDMMMYYYY

| | min - | xx - | | xx - | | xx - | |
|---|---|---|---|---|---|---|---|
| | max | XX | xx - xx | XX | xx - xx | XX | xx - xx |
| C2D1 | ~ | | | | | | |
| CZDI | n | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX |
| | SD<br>media | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | n | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | xx - | | xx - | |
| | max | XX | xx - xx | XX | xx - xx | XX | xx - xx |
| (etc for all cycle/ days for the parameter with at least 3 | | | | | | | |
| Patients reported in the overall column). | n | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | XX |
| | SD<br>media | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| | n | XX | XX | XX | XX | XX | XX |
| | min - | xx - | | xx - | | xx - | |
| | max | XX | xx - xx | XX | xx - xx | XX | xx - xx |

BL = Baseline

Note: Baseline is defined as the most recent measurement

prior to the first administration of study drug.

Programming note: repeat for Cohorts 2-5

(etc. for all hematology parameters)

Programming note: repeat for Table 14.3.5.2 Chemistry


Table 14.3.6.1a

Hematology and Coagulation Shifts from Baseline to Worst Value on Study, Overall and by Dose Group (Cohort 1, Safety Population)

| Cohort | Baseline<br>Grade | | | Waxat Cxaa | de on Study | | |
|---|---|---|---|---|---|---|---|
| Parameter | Grade | Normal | 1 | 2 | 3 | 4 | 5 |
| rarameter | | NOTILIAL | 1 | 2 | 3 | 4 | J |
| ohort 1A: FT-2102 (N=xx) | | | | | | | |
| WBC | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 1 | | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 2 | | n (%) | n (%) | n (%) | n (%) | n (% |
| | 3 | | n (%) | n (%) | n (%) | n (%) | n (% |
| | 4 | ( - / | n (%) | n (%) | n (%) | n (%) | n (% |
| PDG | M 1 | | . (0) | ~ (0) | - (0) | - (0) | - 40 |
| RBC | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 1 | ( - / | n (%) | n (%) | n (%) | n (%) | n (% |
| | 2 | , , | n (%) | n (%) | n (%) | n (%) | n (% |
| | 3 | ( - / | n (%) | n (응) | n (응) | n (%) | n (% |
| | 4 | n (%) | n (응) | n (%) | n (%) | n (%) | n (% |
| Platelets | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 3 | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 4 | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| (etc. for all hematology pages | arameters) | | | | | | |
| phort 1B: FT-2102+AZA (N=xx) | | | | | | | |
| WBC | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 3 | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| | 4 | n (%) | n (%) | n (%) | n (%) | n (%) | n (% |
| RBC | Normal | n (응) | n (%) | n (%) | n (%) | n (%) | n (% |
| - | 1 | | n (%) | n (%) | n (%) | n (%) | n (% |
| | 2 | | n (%) | n (%) | n (%) | n (%) | n (% |
| | 3 | , , | n (%) | n (%) | n (%) | n (%) | n (% |
| | 4 | ( - / | n (%) | n (%) | n (%) | n (%) | n (% |
| | 4 | 11 (.0) | 11 (.0) | 11 (.0) | 11 (.0) | 11 (.0) | 11 ( |

| Platelets | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
|---|---|---|---|---|---|---|---|
| | 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 2 | 2 n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 3 | 8 n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| (etc.) | 4 | l n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cohort 1: Overall (N=xx) | | | | | | | |
| WBC | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 2 | 2 n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 3 | 8 n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 4 | n (%) | n (%) | n (응) | n (%) | n (%) | n (%) |
| RBC | Normal | n (%) | n (%) | n (응) | n (%) | n (응) | n (%) |
| | 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 2 | 2 n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 3 | 8 n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 4 | l n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Platelets | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 1 | , , | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 2 | ( - / | n (%) | n (%) | n (%) | n (%) | n (%) |
| | 3 | | n (%) | n (%) | n (%) | n (%) | n (%) |
| (etc.) | 4 | l n (%) | n (%) | n (%) | n (%) | n (%) | n (용) |

Programming note: repeat for Cohorts 2-5

Programming note: repeat for Table 14.3.6.2 Chemistry Shifts (Safety Population)

DATE: HH:MM/DDMMMYYYY

Note: Baseline is defined as the most recent measurement prior to the first administration of study drug.

Note: CTCAE v 4.03 is applied to lab values.

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Table 14.3.7a

Summary of Liver Function Tests of Potential Concern (All Patients Receiving Single Agent Therapy, Safety Population)

| | | Cohort 1A:<br>FT-2102 | Cohort 2A:<br>FT-2102 | Cohort 3A:<br>FT-2102 | Cohort 4A:<br>FT-2102 | Cohort 5:<br>FT-2102 | Overall:<br>FT-2102 |
|---|---|---|---|---|---|---|---|
| Parameter | Statistic | (N = ) | (N = ) | (N = ) | (N = ) | (N = ) | (N = ) |
| ALT | | | | | | | |
| ALT >3X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT >5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT >10X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT >20X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST | | | | | | | |
| AST >3X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >10X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >20X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST, ALT | | | | | | | |
| AST or ALT >3X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST or ALT >5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST or ALT >10X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST or ALT >20X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Bilirubin | | | | | | | |
| Total Bilirubin >1.5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Bilirubin >=2X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALP | | | | | | | |
| ALP >2.5X ULN<br>ALP >5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

DATE: HH:MM/DDMMMYYYY

| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|---|---|---|
| Concurrent AST, ALT and Total Bilirubin* | | | | | | | |
| (AST or ALT $>3$ X ULN) and Total Bilirubin $>1.5$ X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| (AST or ALT >3X ULN) and Total<br>Bilirubin >2X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Concurrent AST, ALT and Total Bilirubin, without ALP abnormality** | | | | | | | |
| (AST or ALT >3X ULN) and Total<br>Bilirubin >1.5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| (AST or ALT $>$ 3X ULN) and Total Bilirubin $>$ 2X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT>3x ULN or AST>3x ULN with CONCURRENT report of selected adverse event(s)*** | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

ULN = Upper limit of normal

Note: A Patient may be counted in more than one row.

<sup>\*</sup>Laboratory parameters must be met within +/- 7 days of those parameters to be counted as concurrent.

<sup>\*\*</sup> ALP must be <2x ULN for all tests drawn within +/- 7 days of the concurrent elevated AST/ALT and Bilirubin.

<sup>\*\*\*</sup>Selected adverse events: Nausea, Vomiting, Anorexia, Abdominal pain, Abdominal discomfort, Fatigue, Jaundice, Pruritus, Chromaturia, Faeces discoloured.


Table 14.3.7b

Summary of Liver Function Tests of Potential Concern (Safety Population)

| | | Cohort 1A:<br>FT-2102 | Cohort 1B:<br>FT-2102 + AZA | Cohort 1:<br>Overall |
|---|---|---|---|---|
| Parameter | Statistic | (N = ) | (N = ) | (N = ) |
| ALT | | | | |
| ALT >3X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT >5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT >10X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT >20X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST | | | | |
| AST >3X ULN | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >5X ULN | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >10X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST >20X ULN | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST, ALT | | | | |
| AST or ALT >3X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST or ALT >5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST or ALT >10X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AST or ALT >20X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Bilirubin | | | | |
| Total Bilirubin >1.5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Bilirubin >=2X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALP | | | | |
| ALP >2.5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALP >5X ULN | | | | |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Concurrent AST, ALT and Total Bilirubin* | | | | |
| (AST or ALT $>3$ X ULN) and Total Bilirubin $>1.5$ X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

DATE: HH:MM/DDMMMYYYY

| (AST or ALT $>$ 3X ULN) and Total Bilirubin $>$ 2X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Concurrent AST, ALT and Total Bilirubin, without ALP abnormality** | | | | |
| (AST or ALT $>$ 3X ULN) and Total Bilirubin $>$ 1.5X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| (AST or ALT $>$ 3X ULN) and Total Bilirubin $>$ 2X ULN | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No post-baseline values meet the criteria | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALT>3x ULN or AST>3x ULN with CONCURRENT report of selected adverse event(s)*** | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

ULN = Upper limit of normal

Note: A Patient may be counted in more than one row.

Programming note: repeat for cohorts 3-5.

<sup>\*</sup>Laboratory parameters must be met within +/- 7 days of those parameters to be counted as concurrent.

<sup>\*\*</sup> ALP must be <2x ULN for all tests drawn within +/- 7 days of the concurrent elevated AST/ALT and Bilirubin.

<sup>\*\*\*</sup>Selected adverse events: Nausea, Vomiting, Anorexia, Abdominal pain, Abdominal discomfort, Fatigue, Jaundice, Pruritus, Chromaturia, Faeces discoloured.


Table 14.3.8a

Summary of Vital Signs and Change from Baseline by Time Point, Overall and by Dose Group (Cohort 1, Safety Population)

| | | ( | Cohort 1A: | | | Cohort 1: | |
|---|---|---|---|---|---|---|---|
| Parameter | Statistic | | FT-2102 | | | Overall | |
| | | | (N = ) | | (N = ) | | (N = ) |
| | | Value | Change from BL | Value | Change from BL | Value | Change from BL |
| SBP (unit)<br>C1D1 | | | | | | | |
| | n | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | xx |
| | SD | xx.x | XX.X | XX.X | XX.X | xx.x | xx.x |
| | median | XX | XX | XX | XX | XX | XX |
| | min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| C1D8 | n | XX | XX | xx | XX | XX | XX |
| | mean | xx | XX | XX | XX | XX | xx |
| | SD | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x |
| | median | XX | XX | XX | XX | xx | xx |
| | min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| C1D15 | n | XX | XX | XX | XX | XX | xx |
| 01210 | mean | XX | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| | median | XX | XX | xx | XX | xx | XX |
| | min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| C1D22 | n | vv | vv | vv | vv | xx | XX |
| CIDZZ | mean | XX<br>XX | XX<br>XX | xx | XX<br>XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | median | XX | XX | XX | XX | XX | XX |
| | min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| C2D1 | n | XX | XX | XX | XX | XX | XX |
| | mean | XX | XX | XX | XX | XX | xx |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| | median | XX | XX | XX | XX | XX | xx |
| | min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
(etc for all cycle/ days for the parameter with at least 3 Patients reported in the overall column).

(etc. for all vital signs)

| n | XX | XX | XX | XX | XX | XX |
|-----------|---------|---------|---------|---------|---------|---------|
| mean | XX | XX | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| median | XX | XX | XX | XX | XX | XX |
| min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |

BL = Baseline

Programming note: repeat for Cohorts 2-5

DATE: HH:MM/DDMMMYYYY

Note: Baseline is defined as the most recent measurement prior to the first administration of study drug.


nfidential Page 1 of x

### Table 14.3.9a

## Summary of ECG Results and Change from Baseline (Cohort 1, Safety Population)

| | | | Cohort 1A: | | С | ohort 1B: | ( | Cohort 1: |
|---|---|---|---|---|---|---|---|---|
| Parameter | | | | FT-2102 | FT- | -2102 + AZA | | Overall |
| Visit | Time Point | Statistic | (N = ) | | (N = ) | | | (N = ) |
| QRS (unit)<br>C1D1 | | | Value | Change from BL | Value | Change from BL | Value | Change from BL |
| CIDI | Pre-dose | n | XX | XX | XX | xx | XX | XX |
| | 110 0000 | mean | XX | XX | XX | XX | XX | XX |
| | | SD | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | median | xx | XX | xx | XX | xx | XX |
| | | min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| | 4 hours | n | xx | xx | xx | xx | xx | xx |
| | | mean | xx | XX | XX | XX | XX | XX |
| | | SD | xx.x | XX.X | xx.x | XX.X | XX.X | XX.X |
| | | median | XX | XX | XX | XX | XX | XX |
| | | min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| | 8 hours | n | XX | xx | xx | xx | xx | XX |
| | | mean | XX | XX | XX | XX | XX | XX |
| | | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | median | XX | XX | XX | XX | XX | XX |
| | | min - max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| C1D2 | Pre-dose | n | XX | xx | xx | xx | xx | XX |
| | | mean | XX | XX | XX | XX | XX | XX |
| | | SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | median | XX | XX | XX | XX | XX | XX |
| | | min - max | xx - xx | XX - XX | xx - xx | xx - xx | xx - xx | xx - xx |

(etc for all cycle/ days/ time points for the parameter with at least 3 Patients reported in the overall column).

| XX | XX | XX | XX | XX | XX |
|---|---|---|---|---|---|
| XX | XX | XX | XX | XX | XX |
| xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX | XX | XX | XX | XX | XX |
| xx - xx | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| | xx<br>xx.x<br>xx | xx xx<br>xx.x xx.x<br>xx xx | xx xx xx xx.x xx.x xx.x xx xx xx | XX XX XX XX.X XX.X XX.X XX XX XX | XX XX XX XX XX.X XX.X XX.X XX.X XX XX XX XX |

(etc. for all ECG parameters)

BL = Baseline

Programming note: repeat for Cohorts 2-5

DATE: HH:MM/DDMMMYYYY

Note: Baseline is defined as the most recent measurement prior to the first administration of study drug.


### Table 14.3.10.1a

QTcF Shifts from Baseline (Single Agent Therapy, Safety Population)

| | | Maximum Post-Baseline Value | | | | | |
|---|---|---|---|---|---|---|---|
| | | <=450 msec | >450 to | >480 to | >500 msec | | >60 msec |
| | | | <=480 msec | <=500 msec | | msec Change | Change from |
| Treatment Group | Baseline Value | | | | | from Baseline | Baseline |
| | | n (응) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cohort 1 (N=xx) | <=450 mse | С | | | | | |
| | >450 to <=480 mse | С | | | | | |
| | >480 to <=500 mse | С | | | | | |
| | >500 mse | С | | | | | |
| | Tota | 1 | | | | | |
| Cohort 2 (N=xx) | <=450 mse | С | | | | | |
| | >450 to <=480 mse | С | | | | | |
| | >480 to <=500 mse | С | | | | | |
| | >500 mse | С | | | | | |
| | Tota | 1 | | | | | |
| Cohort 3 (N=xx) | <=450 mse | | | | | | |
| | >450 to <=480 mse | | | | | | |
| | >480 to <=500 mse | С | | | | | |
| | >500 mse | С | | | | | |
| | Tota | 1 | | | | | |
| Cohort 4 (N=xx) | <=450 mse | | | | | | |
| | >450 to <=480 mse | | | | | | |
| | >480 to <=500 mse | С | | | | | |

DATE: HH:MM/DDMMMYYYY

>500 msec

Total

Cohort 5 (N=xx) <=450 msec

>450 to <=480 msec

>480 to <=500 msec

>500 msec

Total

Repeat for:

Table 14.3.10.1b QTcF Shifts from Baseline (Combination Therapy, Safety Population)

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Figure 14.3.10.2a

Maximum Post Baseline QTcF vs Baseline QTcF (Single Agent Therapy, Safety Population)



Repeat for 14.3.10.2b (Combination Therapy, Safety Population)

# Programming notes:

- One axis represents baseline QTcF and the other axis represents maximum post-baseline QTcF. Include unscheduled visits as candidates for maximum.
- Color code the dots by cohort.
- Add reference lines for QTcF of 450, 480, and 500 on both axes.

#### Confidential


Table 14.3.11a
Concomitant Medications (Cohort 1)

| | | Cohort 1A: | Cohort 1B: | Cohort 1: |
|--------------|-----------|------------|---------------|-----------|
| Parameter | Statistic | FT-2102 | FT-2102 + AZA | Overall |
| | | (N = ) | (N = ) | (N = ) |
| Drug class 1 | n (%) | | | |
| ATC text 1 | n (%) | | | |
| ATC text 2 | n (%) | | | |
| ATC text 3 | n (%) | | | |
| etc. | n (%) | | | |
| Drug class 2 | n (%) | | | |
| ATC text 1 | n (%) | | | |
| ATC text 2 | n (%) | | | |
| ATC text 3 | n (%) | | | |
| etc. | n (%) | | | |

Repeat for Cohorts 2-5

DATE: HH:MM/DDMMMYYYY

Note: Patients are counted once per drug class and ATC. Concomitant Medications are coded with the WHO Drug version March 2018.

# 10. DATA LISTING SHELLS


Protocol 2102-ONC-102

Listing 16.2.1.1

Study Completion Status

First Dose Last Dose Reason for Date of Reason for Date of FT-Date of FT-Terminating Terminating Last Last Dose Rel Cohort Patient 2102 2102 Treatment Study Day Contact


DATE: HH:MM/DDMMMYYYY

Listing 16.2.1.2

Pre-Screening Consent

Pre-Screening IDH1 Mutation Consent Date for Date of Tissue Cohort Patient Consent Result Archival Tumor Tissue Collection


DATE: HH:MM/DDMMMYYYY

Listing 16.2.1.3

Enrollment

Study Phase Pharmaco- Consent for C3 Tumor Cohort Patient Screen Failure and Stage Safety Lead In genomics Consent Tissue Sample


DATE: HH:MM/DDMMMYYYY

Listing 16.2.2.1

Inclusion and Exclusion Criteria

Informed Protocol Version Cohort Patient Consent Date Consented Inclusion/ Exclusion Criteria Not Met


DATE: HH:MM/DDMMMYYYY

Listing 16.2.2.2

Protocol Violations

Violation Violation

Cohort Patient Severity Category Violation Description

Major

Minor


DATE: HH:MM/DDMMMYYYY

Listing 16.2.3.1

Analysis Sets

Response
Cohort Patient DLT Evaluable Set Safety Set Evaluable Set PK Set PD Set

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Listing 16.2.4.1

Demographics and Baseline Information

Age at Child Bearing
Cohort Patient Consent Height (cm) Sex at Birth Potential Ethnicity Race


Listing 16.2.4.2

Baseline Disease Data and Cancer Diagnosis

| | | | Initial | | | | Current | | | | _ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Diagnosis | | | TNM | | Recurrence | | | TNM | |
| Cohort | Patient | Diagnosis | Date | Grade | Stage | Stage | Diagnosis | Date | Grade | Stage | Stage | Fibrosis |


Listing 16.2.4.3

IDH1 and Other Mutations

IDH Mutation

Cohort Patient Sample Date Method Site of Tissue Result IDH Mutation Other Mutations


Listing 16.2.4.4

Medical History

Cohort Patient Start Date Verbatim Term SOC PT CTC Grade End Date

DATE: HH:MM/DDMMMYYYY

Note: Medical Histories are coded with the MedDRA version 21.0.


Listing 16.2.4.5

Prior Anti-Cancer Therapies

Therapy Type/ e/ WHO Drug

Therapy Name/ WHO Drug Start Date/
Cohort Patient Regimen WHO Drug Name Class End Date Best Response

DATE: HH:MM/DDMMMYYYY

Note: Prior anti-cancer therapy medications are coded with the WHO Drug version March 2018.

### Programming notes:

• For Best Response, abbreviate responses as: CR, PR, MR, SD, PD, ND, UN


DATE: HH:MM/DDMMMYYYY

Listing 16.2.4.6

Prior Radiotherapy

| Type of | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Cohort | Patient | Radiation | Start Date | End Date | Dose | Unit | Location | Response |


Listing 16.2.4.7

Major Surgical Tumor Resections

Cohort Patient Surgical Procedure Description Location Procedure Date


DATE: HH:MM/DDMMMYYYY

Listing 16.2.4.8

Child Pugh Score

| | | | | | | нератіс | |
|---|---|---|---|---|---|---|---|
| | Assessment | Total | Serum | | | Encepal- | Child Pugh |
| Cohort Patien | t Date | Bilirubin | Albumin | INR | Ascites | opathy | Score |


DATE: HH:MM/DDMMMYYYY

Listing 16.2.4.9

Hepatitis B and C

Cohort Patient Assessment Date Assessment Time Method of Assessment Result Titer Unit Result Titer Unit


DATE: HH:MM/DDMMMYYYY

Listing 16.2.4.10

Archival Tumor Tissue

Was the sample sent to the Cohort Patient Collection Date Sample Type Tissue Site lab?


DATE: HH:MM/DDMMMYYYY

Listing 16.2.5.1

FT-2102 Administration

| | | | | | | Actual | | |
|---|---|---|---|---|---|---|---|---|
| | | Start Date | End Date | Assigned | | Total Daily | Dose | |
| Cohort | Patient | (Rel Day) | (Rel Day) | Dose | Frequency | Dose | Modification | Reason |


DATE: HH:MM/DDMMMYYYY

Listing 16.2.5.2

FT-2102 Drug Accountability

| | | | Disp | ensed | Retu | ırned | Taken per | Pt Diary | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Total<br>Dose | Total Dose<br>Not Taken<br>and Not | |
| | | | 50 mg | 150 mg | 50 mg | 150 mg | 50 mg | 150 mg | Taken | Returned | Percent |
| Cohort | Patient | Cycle | Capsules | Capsules | Capsules | Capsules | Capsules | Capsules | (mg) | (mg) | Compliance |


Listing 16.2.5.3

Azacitidine, Nivolumab, Cisplatin, and Gemcitabine Administration

| | | | | Dosing | | Assigned | | | Volume | | Interruption/ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Cycle/ | Date | Start/ | Dose | Prepared | Volume of | Admin- | Dose | Reason/ Start |
| | | | Time | (Rel | Stop | (Unit)/ | Dose | Prepared | istered | Modification/ | Time/ Stop |
| Cohort | Patient | Drug | Point | Day) | Time | Route | (mg) | Dose (mL) | (mL) | Reason | Time |

Azacitidine Nivolumab Cisplatin Gemcitabine


DATE: HH:MM/DDMMMYYYY

Listing 16.2.5.4

Pharmacokinetic Concentrations

Cohort Patient Visit Sample Date Rel Day Value Laboratory Comments

FORMA Therapeutics 2102-ONC-102 Statistical Analysis Plan 28 June 2019, Version 2.0


DATE: HH:MM/DDMMMYYYY

Listing 16.2.5.5

Pharmacokinetic Parameters

Cohort Patient - Cmax Tmax Thalf AUC


DATE: HH:MM/DDMMMYYYY

Listing 16.2.6.1

Target Lesions (RECIST)

| | | Imaging | | Lesion | Method of | | | Longest |
|---|---|---|---|---|---|---|---|---|
| | | Date (Rel | Lesion | Location/ | Measurement & | Lesion | Assessment | Diameter |
| Cohort Patier | t Visit | Day) | Number | Description | Contrast | State | Result | (mm) |

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Listing 16.2.6.2

Non-Target and New Lesions (RECIST)

| | | | Imaging | Lesion | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Date | Number/ | Lesion | Method of | | | Longest |
| | | | (Rel | New | Location/ | Measurement & | Lesion | Assessment | Diameter/ |
| Cohort | Patient | Visit | Day) | Lesion | Description | Contrast | State | Result | Short Axis |


Protocol 2102-ONC-102

Listing 16.2.6.3

Measurable Lesions (RANO)

| Cohort | Patient | Visit | Imaging<br>Date<br>(Rel<br>Day) | Lesion<br>Number | Lesion<br>Location<br>Category | Location<br>Description | Method of<br>Measurement<br>& MRI<br>Details | Lesion<br>Assessment<br>Result | Longest<br>Diameter<br>(mm) | Perpendicular<br>Measurement<br>(mm) | Lesion<br>Area<br>(mm^2) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Cerebrum | Print<br>Location | | | | | |
| | | | | | Cerebellum | from nodal | | | | | |
| | | | | | Brainstem | location or | | | | | |
| | | | | | Spine | extranodal location | | | | | |
| | | | | | Other | and | | | | | |
| | | | | | | location | | | | | |
| | | | | | | description fields | | | | | |


Listing 16.2.6.4

Non-Measurable and New Lesions (RANO)

| Cohort | Patient | Visit | Imaging<br>Date<br>(Rel<br>Day) | Lesion<br>Number/<br>New<br>Lesion | Lesion<br>Location<br>Category | Location<br>Description | Method of<br>Measurement<br>& MRI<br>Details | Lesion<br>Assessment<br>Result | Longest<br>Diameter<br>(mm) | Perpen-<br>dicular<br>Measurement<br>(mm) | Lesion<br>Area<br>(mm^2) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Cerebrum | Print<br>Location | | | | | |
| | | | | | Cerebellum | from nodal | | | | | |
| | | | | | Brainstem | location or | | | | | |
| | | | | | Spine<br>Other | extranodal<br>location<br>and | | | | | |
| | | | | | | location<br>description<br>fields | | | | | |

DATE: HH:MM/DDMMMYYYY

FORMA Therapeutics Confidential Page 1 of x Protocol 2102-ONC-102

Listing 16.2.6.5

Response Assessment (RECIST)

Non-Assessment Target Target Best Progression Date (Rel Date (Rel Lesion Lesion New Overall Overall Cohort Patient Visit Day) Response Response Lesions Response Response Day)


Listing 16.2.6.6

Response Assessment (RANO)

Non-

| | Assessment | Measurable | Measurable | | | | | Best | Progression |
|---|---|---|---|---|---|---|---|---|---|
| | Date (Rel | Lesion | Lesion | New | Steroid | Clinical | Overall | Overall | Date (Rel |
| Cohort Patient Visit | Day) | Response | Response | Lesions | Status | Status | Response | Response | Day) |

DATE: HH:MM/DDMMMYYYY


Listing 16.2.6.7

Response Assessment (Cheson)

| | | | | Sum of the | | Non- | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Assessment | Product | Measurable | Measurable | | | Best | Progression |
| | | | Date (Rel | Diameters | Lesion | Lesion | New | Overall | Overall | Date (Rel |
| Cohort | Patient | Visit | Day) | (mm^2) | Response | Response | Lesions | Response | Response | Day) |

DATE: HH:MM/DDMMMYYYY


DATE: HH:MM/DDMMMYYYY

Listing 16.2.6.8

Survival Status

| | | Date Last | | Disease Progression | Treated with Anti- | Start Date of New |
|---|---|---|---|---|---|---|
| | | Known Alive | Patient Status at | Not Previously | Cancer Therapy for | Treatment (Rel |
| Cohort | Patient | (Rel Day) | Time of Follow Up | Reported? | Disease? | Day) |


Listing 16.2.6.9

Serum AFP, CA-19-9, and CEA

Date of Serum AFP Laboratory
Cohort Patient Visit Sample Rel Day Value CA19-9 Value CEA Value Comments


Listing 16.2.6.10

EQ-5D-5L Quality of Life Assessment

| | | | | | | | | | rour |
|---|---|---|---|---|---|---|---|---|---|
| | | | Assessment | | Self | Usual | Pain/ | Anxiety/ | Health |
| Cohort | Patient | Visit | Date (Rel Day) | Mobility | Care | Activities | Discomfort | Depression | Today |


DATE: HH:MM/DDMMMYYYY

Listing 16.2.6.11

2-HG MRS Assessments

Assessment

Cohort Patient Visit Date Rel Day 2-HG Value Imaging Reader Comments


Listing 16.2.6.12

Archival Tumor Tissue and Biopsy

Sample Collection Tissue Collection Sample Sent Cohort Patient Visit Date Rel Day Sample Type Site to Lab?


DATE: HH:MM/DDMMMYYYY

Listing 16.2.6.13

Pharmacogenomics Samples

Pharmacogenomics Sample Cohort

Visit Collected? Patient Sample Date Rel Day Sample Time


Listing 16.2.7.1

Adverse Events by Patient and Verbatim Term

| | | | | | | | | | | Action | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | Taken | |
| | | | | | | | | | | with | Other |
| | | Verbatim | Preferred | Start Date | Stop Date | CTCAE | | | Relationship | Study | Action |
| Cohort | Patient | Term | Term | (Rel Day) | (Rel Day) | Grade | SAE | Outcome | to Drug <sup>1</sup> | Drug <sup>2</sup> | Taken |

Programming Note: Sort by cohort, Patient, start date, and preferred term

## 

DATE: HH:MM/DDMMMYYYY

Note: Adverse Events are coded with the MedDRA version 21.0.

Note: The combination drug is Azacitidine in cohort 1b and 3b, Nivolumab in cohort 2b, and Gemcitibine + Cisplatin in cohort 4b.

<sup>1</sup> Relationship to Drug: None, REM = Remote, POS= Possible, PROB= Probable, DEF= Definite and NA= Not Applicable

<sup>&</sup>lt;sup>2</sup> Action Taken with Study Drug: None = Dose Not Changed; INT = Dose Interrupted; RED = Dose Reduced; WD = Drug Withdrawn.


Listing 16.2.7.2

Adverse Events by Patient and MedDRA System Organ Class and Preferred Term

| | | | | | | | | | | Actio | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | n | |
| | | | | | Stop | | | | | Taken | Other |
| | | | | Start | Date | | | | | with | Actio |
| Cohor | Patien | System Organ | Preferred | Date (Rel | (Rel | CTCAE | SA | Outcom | Relationshi | Study | n |
| t | t | Class | Term | Day) | Day) | Grade | E | е | p to Drug <sup>1</sup> | Drug <sup>2</sup> | Taken |

Programming Note: Sort by cohort, Patient, system organ class, preferred term, and start date.

DATE: HH:MM/DDMMMYYYY

Note: Adverse Events are coded with the MedDRA version 21.0.

Note: The combination drug is Azacitidine in cohort 1b and 3b, Nivolumab in cohort 2b, and Gemcitibine + Cisplatin in cohort 4b.

1 Relationship to Drug: None, REM = Remote, POS= Possible, PROB= Probable, DEF= Definite and NA= Not Applicable

<sup>&</sup>lt;sup>2</sup> Action Taken with Study Drug: None = Dose Not Changed; INT = Dose Interrupted; RED = Dose Reduced; WD = Drug Withdrawn.


Listing 16.2.7.3

Adverse Events by MedDRA System Organ Class, Preferred Term, Cohort, and Patient

| | | | | | Stop | | | | | Action | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Date | | | | | Taken with | Other |
| System Organ | | | | Start Date | (Rel | CTCAE | | | Relationship | Study | Action |
| Class | Preferred Term | Cohort | Patient | (Rel Day) | Day) | Grade | SAE | Outcome | to Drug1 | Drug <sup>2</sup> | Taken |

Programming Note: Sort by system organ class, preferred term, cohort, Patient, and start date.

DATE: HH:MM/DDMMMYYYY

Note: Adverse Events are coded with the MedDRA version 21.0.

Note: The combination drug is Azacitidine in cohort 1b and 3b, Nivolumab in cohort 2b, and Gemcitibine + Cisplatin in cohort 4b.

1 Relationship to Drug: None, REM = Remote, POS= Possible, PROB= Probable, DEF= Definite and NA= Not Applicable

<sup>&</sup>lt;sup>2</sup> Action Taken with Study Drug: None = Dose Not Changed; INT = Dose Interrupted; RED = Dose Reduced; WD = Drug Withdrawn.

OMO A D


Listing 16.2.8.1

Laboratory Results: Hematology

| | | | | | | | | | CICAL | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Sample date | Visit | | | | | Grade/ | Clinical |
| Cohort | Patient | Test Name | (Rel Day) | Name | Result | Units | LLN | ULN | Flag | Significance |

Programming note: for CTCAE Grade/ Flag, show CTCAE grade if the lab test is graded via CTCAE 4.03 criteria. If not, indicate H for above upper limit of normal or L for below lower limit of normal

Programming note: repeat for 16.2.8.2, 16.2.8.3, 16.2.8.4, 16.2.8.6

Programming note: tests that should be in 16.2.8.6 include TSH testing, pregnancy, and Hepatitis B and C testing


DATE: HH:MM/DDMMMYYYY

Listing 16.2.8.5

Laboratory Normal Ranges

Laboratory Name Start Date Stop Date Gender Age Category LLN ULN

FORMA Therapeutics


Protocol 2102-ONC-102

Listing 16.2.9.1

Vital Signs

Respiratory Temperature Assessment Date Assessment Weight Pulse Rate SBP DBP (kg) Cohort Patient Visit Time ( C) (beats/min) (breaths/mim) (mmHg) (mmHg) (Rel Day)


Listing 16.2.9.2

Physical Examination

If Abnormal, Was
Overall Abnormality Present at
Cohort Patient Visit Assessment Date Rel Day Assessment Screening


Listing 16.2.9.3

Electrocardiogram Results

Overall Evaluation/ Assessment Date Time Time of Clinical Abnormal, Cohort Patient Visit (Rel Day) Point ECG ECG # PR HR QRS QT QTcF Significance Specify

Start


Protocol 2102-ONC-102 Listing 16.2.9.4

Prior and Concomitant Medications

Date (Rel Day) / Stop WHO Reason for Dose Date Drug Medication/ and (Rel Cohort Patient Medication Class ATC Text Indication Units Frequency Route Day) Prior/ Concomitant

Note: Prior and Concomitant Medications are coded with the WHO Drug version March 2018.


DATE: HH:MM/DDMMMYYYY

Listing 16.2.9.5

Concomitant Procedures

Reason for Cohort Patient Procedure Procedure Location Procedure Date Rel Day

Note: sort by cohort, Patient, and procedure date.


Listing 16.2.9.6

Systemic Steroid Dosing

| | | | | | | | | Start Date<br>(Rel Day)/ |
|---|---|---|---|---|---|---|---|---|
| | | | WHO Drug | | Dose and | | | Stop Date |
| Cohort | Patient | Medication | Class | ATC Text | Units | Frequency | Route | (Rel Day) |


DATE: HH:MM/DDMMMYYYY

Listing 16.2.9.7

ECOG Performance Status

Assessment

Cohort Patient Visit Date Rel Day ECOG Performance Status

## 11. REVISION HISTORY

| Version/ Date | Revisions |
|---|---|
| VEISION/ Date | Revisions |
| 1.0/ 05MAR2019 | First version |
| 2.0/ 28JUN2019 | Update SAP to align with version 3.0 of the protocol. Edit PK analysis details, minor edits/ clarifications to table shells, add QTcF figure, clarify handling of missing date parts, edit criteria for liver |
| | function test summary table. |

## 12. STUDY SCHEMATIC



FORMA Therapeutics 2102-ONC-102 Statistical Analysis Plan 28JUN2019, Version 2.0

Combo A=FT-2102 + 5-azacitidine; Combo B=FT-2102 + PD-1 inhibitor (nivolumab); Combo C=FT-2102 + GemCis; Chondro=chondrosarcoma; DLT=dose limiting toxicity; HBC=hepatobiliary cancer; IHCC=intrahepatic cholangiocarcinoma; mut=mutation; SA=single-agent FT-2102.

Combination therapy in cohorts 1-4 may also be examined in the event that the single agent cohort passes the futility analysis and the enrollment in the single agent cohort is completed **Up to** 6 patients with relapsed or refractory non-CNS solid tumors harboring an IDH1 R132X mutation in exploratory Cohort 5a will be treated with single-agent FT-2102.